# JOHNSON & JOHNSON VISION CARE, INC.

# Clinical Study Protocol

Clinical Characterization of Symptomatic Populations

Protocol CR-5969

Version: 3.0

Date: 03 October 2017

Investigational Products: ACUVUE OASYS®1-Day with HydraLuxe<sup>™</sup> Technology (senofilcon A) is a daily disposable marketed and FDA approved contact lens which will be worn as a daily disposable.

Key Words: Senofilcon A, ACUVUE OASYS® 1-Day with HydraLuxe™ Technology, daily disposable, daily wear, dispensing, symptomatic, characterization, CLDEQ-8, OSDI, Sensitivity Questionnaire (Highly Sensitive Person-HSP Scale), Meibomian Gland, Lipiview, tear film lipid layer thickness, blink patterns, tear film stability, tear film lipid pattern, lid wiper epitheliopathy, corneal staining, conjunctival staining, conjunctival folds, lid margin evaluation, Korb Meibomian Gland Evaluator (MGE)

Statement of Compliance to protocol, GCP and applicable regulatory guidelines: This trial will be conducted in compliance with the protocol, ISO 14155, the International Conference on Harmonization Good Clinical Practice E6 (ICH-GCP), the Declaration of Helsinki, and all applicable regulatory requirements.

#### **Confidentiality Statement:**

This document contains confidential information, which should not be copied, referred to, released or published without written approval from Johnson & Johnson Vision Care, Inc. The information may not be disclosed to others except to the extent necessary to obtain Institutional Review Board/Independent Ethics Committee approval and informed consent, or as required by International, Federal and State Laws, as applicable. Persons to whom this information is disclosed must be informed that this information is privileged and confidential and that it should not be further disclosed without the written permission of Johnson & Johnson Vision Care, Inc. Any supplemental information that may be added to this document is also confidential and proprietary to Johnson & Johnson Vision Care, Inc. and must be kept in confidence in the same manner as the contents of this document.

#### TABLE OF CONTENTS PROTOCOL TITLE, NUMBER, VERSION.....6 SPONSOR NAME AND ADDRESS......6 MEDICAL MONITOR......6 AUTHORIZED SIGNATURES......7 CHANGE HISTORY......8 SYNOPSIS 9 INTRODUCTION AND BACKGROUND ......16 1.1. 1.2. 1.3. 1.4. 1.5. Relevant Literature References and Prior Clinical Data Relevant to Proposed Clinical Study......17 STUDY OBJECTIVES, ENDPOINTS AND HYPOTHESES ......18 2.1. 2.2. 2.3. TARGETED STUDY POPULATION ......20 3.1. 3.2. Inclusion Criteria 20 3.3. 3.4. STUDY DESIGN AND RATIONALE......21 4.1. 4.2. 4.3. Enrollment Target and Study Duration \_\_\_\_\_\_22 TEST ARTICLE ALLOCATION AND MASKING......22 5.1. 5.2. 5.3. Procedures for Maintaining and Breaking the Masking......22

Identity of Test Articles......23

6.1.

6.2.

| 6.3. | Administration of Test Articles | 24 |
|---|---|---|
| 6.4. | Packaging and Labeling | 25 |
| 6.5. | Storage Conditions | 25 |
| 6.6. | Collection and Storage of Samples | 25 |
| 6.7. | Accountability of Test Articles | 25 |
| 7. S | TUDY EVALUATIONS | 26 |
| 7.1. | Time and Event Schedule | 26 |
| 7.2. | Detailed Study Procedures | 29 |
| Pı | re-Visit Screening: | 29 |
| V | ISIT 1: | 30 |
| V | ISIT 2: | 36 |
| V | ISIT 3: | 39 |
| V | ISIT 4: | 42 |
| FI | INAL EVALUATION | 45 |
| 7.3. | Unscheduled Visits | 45 |
| 7.4. | Laboratory Procedures | 46 |
| 8. SI | UBJECTS COMPLETION/WITHDRAWAL | 46 |
| 8.1. | Completion Criteria | 46 |
| 8.2. | Withdrawal/Discontinuation from the Study | 47 |
| 9. PI | RE-STUDY AND CONCOMITANT INTERVENTION/MEDICATION | 47 |
| 10. | DEVIATIONS FROM THE PROTOCOL | 47 |
| 11. | STUDY TERMINATION | 48 |
| 12. | PROCEDURE FOR HANDLING PRODUCT QUALITY COMPLAINTS | 48 |
| 13. | ADVERSE EVENTS | 49 |
| 13.1. | . Definitions and Classifications | 49 |
| 13.2. | . Assessing Adverse Events | 52 |
| 13 | 3.2.1. Causality Assessment | 52 |
| 13 | 3.2.2. Severity Assessment | 52 |
| 13.3. | . Documentation and Follow-Up of Adverse Events | 53 |
| 13.4. | . Reporting Adverse Events | 54 |
| 13 | 3.4.1. Reporting Adverse Events to Sponsor | 54 |
| | 3.4.2. Reporting Adverse Events to the Responsible IEC/IRB and Euthorities | |
| | 3.4.3. Event of Special Interest | |
| 13.5. | . Reporting of Pregnancy | 55 |

| 14. S' | TATISTICAL METHODS | 56 |
|---|---|---|
| 14.1. | General Considerations | 56 |
| 14.2. | Sample Size Justification | 56 |
| 14.3. | Analysis Populations | 57 |
| 14.4. | Level of Statistical Significance | 57 |
| 14.5. | Primary Analysis | 57 |
| 14.6. | Secondary Analysis | 58 |
| 14.7. | Other Exploratory Analyses | 58 |
| 14.8. | Interim Analysis | 58 |
| 14.9. | Procedure for Handling Missing Data and Drop-Outs | 58 |
| 14.10. | Procedure for Reporting Deviations from Statistical Plan | 58 |
| 15. D | ATA HANDLING AND RECORD KEEPING/ARCHIVING | 58 |
| 15.1. | Electronic Case Report Form/Data Collection | 58 |
| 15.2. | Subject Record | 59 |
| 16. D | ATA MANAGEMENT | 59 |
| 16.1. | Access to Source Data/Document | 59 |
| 16.2. | Confidentiality of Information | 59 |
| 16.3. | Data Quality Assurance | 60 |
| 17. M | IONITORING | 60 |
| 18. E | THICAL AND REGULATORY ASPECTS | 60 |
| 18.1. | Study-Specific Design Considerations | 60 |
| 18.2. | Investigator Responsibility | 61 |
| 18.3. | Independent Ethics Committee or Institutional Review Board (IEC/IRB) | 61 |
| 18.4. | Informed Consent | 62 |
| 18.5. | Privacy of Personal Data | 63 |
| 19. S | TUDY RECORD RETENTION | 64 |
| 20. F | INANCIAL CONSIDERATIONS | 65 |
| 21. P | UBLICATION | 65 |
| 22. R | EFERENCES | 65 |
| APPENI | DIX A: PATIENT REPORTED OUTCOMES (STUDY QUESTIONNAIRES) | 67 |
| APPENI | DIX B: PATIENT INSTRUCTION GUIDE | 79 |
| APPENI | DIX C: PACKAGE INSERT (APPROVED PRODUCT) | 101 |
| APPENI | DIX D: LIPVIEW II MANUFACTURER INSTRUCTIONS | 130 |
| APPENI | DIX E: MEIBOSCALE | 178 |

CR-5969 v3.0

| APPENDIX F: EVALUATION OF LID WIPER EPITHELIOPATHY (LWE) |
|---|
| APPENDIX G: LIPCOF GRADING SCALE180 |
| APPENDIX H: MEIBOMIAN GLAND EVALUATOR MANUFACTURER INSTRUCTIONS |
| APPENDIX I: MEIBOMIAN GLAND SECRETION GRADING SCALE |
| APPENDIX J: CLINICAL TECHNICAL PROCEDURES (CTP)183 |
| Pre-Ocular and Pre-Lens Wettability |
| Limbal and Conjunctival (Bulbar) Redness |
| Expanded Sodium Fluorescein Corneal Staining |
| Lens Fitting Characteristics |
| Subject Reported Ocular Symptoms/Problems |
| Front and Back Surface Lens Deposit Grading Procedure |
| Determination of Distance Spherocylindrical Refractions |
| Biomicroscopy Scale |
| Conjunctival Staining |
| Keratometry Procedure |
| Distance and Near Visual Acuity Evaluation |
| Lens Insertion and Removal |
| White Light Lens Surface Wettability |
| APPENDIX K: WORK AID: NON-INVASIVE TEAR BREAK-UP TIME (NIBUT) MEASUREMENT USING THE MEDMONT E300 CORNEAL TOPOGRAPHER 250 |
| PROTOCOL COMPLIANCE INVESTIGATOR(S) SIGNATURE PAGE255 |
| TABLE OF CONTENTS Figure 1: Study Flowchart |
| TABLE OF CONTENTS |
| Table 1: Test Articles23 |
| Table 2a: Ancillary Supplies- Instrumentation Equipment |
| Table 2b: Ancillary Supplies, Solution-Rinsing/Storage |
| Table 2c: Ancillary Supplies, Solution- Artificial Tears/ Rewetting Drops |
| Table 3: Time and Events |

#### PROTOCOL TITLE, NUMBER, VERSION

Title: Clinical Characterization of Symptomatic Populations

Protocol Number: CR-5969

Version: 3.0

Date: 03 October 2017

#### **SPONSOR NAME AND ADDRESS**

Johnson & Johnson Vision Care, Inc. (JJVC) 7500 Centurion Parkway Jacksonville, FL 32256

#### MEDICAL MONITOR

Name: Elizabeth Dow, OD, FAAO Title: Principal Research Optometrist

Address: 7500 Centurion Parkway, Suite 100; Jacksonville, FL 32256

Email: edow1@its.jnj.com

CR-5969 v3.0

The Medical Monitor must be notified by the clinical institution/site by e-mail, fax, or telephone within 24 hours of learning of a Serious Adverse Event. The Medical Monitor may be contacted during business hours for adverse event questions. General study related questions should be directed towards your assigned clinical research associate.

The Medical Monitoring Plan is maintained as a separate document and included in the Trial Master File.

#### **AUTHORIZED SIGNATURES**

The signature below constitutes the approval of this protocol and the attachments, and provides the necessary assurances that this trial will be conducted according to all stipulations of the protocol, including all statements regarding confidentiality, and according to local legal and regulatory requirements and applicable U.S. federal regulations,<sup>4</sup> ICH guidelines,<sup>2</sup> ISO 14155,<sup>1</sup> and the Declaration of Helsinki.<sup>3</sup>

| Author | See Electronic Signature Report | |
|---------------------|------------------------------------------|-----------|
| | Elizabeth Dow, OD, FAAO | DATE |
| | Principal Research Optometrist | |
| Clinical Operations | | |
| Manager | See Electronic Signature Report | DAME |
| | Clinical Operations Manager | DATE |
| | Chinical Operations Manager | |
| Biostatistician | See Electronic Signature Report | |
| | | DATE |
| | Biostatistician Manager | |
| D : 14 | G 70 | |
| Data Management | See Electronic Signature Report | To A CYNY |
| | Clinical Project Manager- Data & Systems | DATE |
| | Chinical Project Manager- Data & Systems | |
| Reviewer | Cas Floatuania Cignatura Danaut | |
| Reviewei | See Electronic Signature Report | DATE |
| | Project Lead | DATE |
| | 110Jeor Deud | |
| Fellow Reviewer | See Electronic Signature Report | |
| | | DATE |
| | Clinical Research Fellow | |
| Approver | See Electronic Signature Report | |
| | Dringing Daggarah Ontonotrict | DATE |
| | Principal Research Optometrist | |
| | See Electronic Signature Report | |
| Approver | | DATE |
| | R&D Director- Drug & Combination | |
| | Products | |

### **CHANGE HISTORY**

| Version | Originator | Description of Change(s) and Section | Date |
|---|---|---|---|
| A CESTOII | Originator | Number(s) Affected | <b>-</b> 3.00 |
| 1.0 | Flizabeth Dow | | 27 JUL 2017 |
| 2.0 | Elizabeth Dow | <ul> <li>Original Protocol</li> <li>Specified Clinical Study Sites</li> <li>Specified enrollment details</li> <li>Specified Meibomian gland expressibility procedure</li> <li>Updated artificial tear/rewetting drops</li> <li>Updated rinsing/storage solutions</li> <li>Updated tear film stability method &amp; endpoint - Medmont</li> <li>Specified Tearscope use - lipid pattern</li> <li>Removed masking of test articles</li> <li>Updated signers</li> <li>Corrected clinical site name</li> <li>Corrected Expanded Corneal Staining step wording</li> <li>Removed preserved solution from ancillary supplies</li> <li>Replaced study lens storage with discard</li> </ul> | 15 SEP 2017 |
| 3.0 | Elizabeth Dow | <ul> <li>Typo corrections including Asymptomatic/symptomatic distribution</li> <li>T&amp;E Table: Tearscope</li> <li>Removal of infectious and immunosuppressive exclusion criteria</li> <li>Provided allowance for LogMAR in addition to Snellen acuity</li> <li>Unscheduled visit amendment</li> <li>Objective amendment</li> <li>Meibomian Gland Imaging study step moved to follow tear assessments</li> </ul> | 03 OCT 2017 |

### **SYNOPSIS**

| Protocol Title | Clinical Characterization of Symptomatic Populations |
|---|---|
| Sponsor | JJVC, 7500 Centurion Parkway, Jacksonville, FL 32256 |
| Clinical Phase | Development phase, phase 0 |
| Trial Registration | This study will be registered on ClinicalTrials.gov. |
| Test Article(s) | Investigational Products: ACUVUE OASYS® 1-Day with |
| | HydraLuxe <sup>TM</sup> Technology - Senofilcon A (Daily disposable) |
| | Control Products: none |
| Wear and Replacement | Wear Schedule: Daily Disposable |
| Schedules | Replacement Schedule: Daily Disposable |
| Objectives | There are two primary objectives of this study: |
| 5 3, 5 5 5 7, 5 5 | 1. To explore the difference in characteristics between |
| | symptomatic and asymptomatic subjects with and without contact lenses utilizing the following metrics: Meibomian gland imaging, meibomian gland expressibility, lid margin evaluation, lid wiper epitheliopathy, and conjunctival folds. 2. Assess any change in clinical metrics throughout 4-weeks of ACUVUE OASYS® 1-Day with HydraLuxe <sup>TM</sup> Technology wear |
| Study Endpoints | Primary endpoints: |
| Study Enapoints | Meibomian gland imaging, meibomian gland expressibility, lid |
| | margin evaluation, lid wiper epitheliopathy, and conjunctival folds. |
| | Secondary endpoints: Conjunctival redness, conjunctival staining tear film lipid layer thickness, tear film stability, tear film lipid pattern. |
| | Other observations: |
| | 1. Blink patterns |
| | 2. Lens fit characteristics. This will be recorded by the |
| | investigator using |
| | 3. Lens surface characteristics. This will be recorded by the |
| | investigator using |
| | 4. Additional physiology characteristics. This will be recorded |
| | by the investigator using |
| | 5. Snellen or LogMAR Visual Acuity |
| | 6. Average daily and comfortable wear time |
| | 7. Reasons for discontinuation |
| | 8. Adverse events |
| | 9. Lens Damage |
| | 10. Subject reported ocular symptoms |
| | 11. CLUE Vision |
| | 12. Frequency of artificial tear/rewetting drop use |

| | 13. Questionnaires (CLUE comfort, MRD, OSDI, Bare Eye, Sensitivity) |
|---|---|
| Study Design | This is an unmasked, non-randomized, single arm, stratified, dispensing investigation of symptomatic and asymptomatic subject populations. Subjects will be assigned to a single study lens type to be worn bilaterally for approximately 4 weeks followed by no contact lens wear for 1 week. This study will be conducted at up to three clinical study sites, including VRC, Jacksonville FL and Centre for Contact Lens Research, University of Waterloo, Ontario. |
| | There will be a total of 4 visits. The time of day of each study visit shall occur within +/- 2 hours of the time of Visit 1. |
| | Pre-Screen Communication (via phone or email): CLDEQ-8 |
| | Visit 1 (habitual lenses on eye ≥6 hrs): Baseline and eligibility: Physiology, Questionnaires (CLDEQ-8, Sensitivity, CLUE, and MRD), CL history. Fitting lens: Fit/dispense ACUVUE OASYS® 1-Day with HydraLuxe™ Technology × 2 weeks |
| | Visit 2 (ACUVUE OASYS® 1-Day with HydraLuxe <sup>TM</sup> Technology on eye ≥6 hrs): Physiology, Questionnaires (CLDEQ-8, CLUE, and MRD) Dispense ACUVUE OASYS® 1-Day with HydraLuxe <sup>TM</sup> Technology for an additional 2 weeks |
| | Visit 3 (ACUVUE OASYS® 1-Day with HydraLuxe <sup>™</sup> Technology on eye ≥6 hrs): Physiology, Questionnaires (CLDEQ-8, CLUE, and MRD) |
| | BARE EYE WASHOUT: Discontinue lens wear for 7±1 days |
| | Visit 4 (Bare eye): Physiology, Questionnaires (Bare Eye, OSDI, and MRD) |
| | See the flow chart at the end of the synopsis table for the schematic of the study visits and procedures of main observations (Figure 1). |
| Sample Size | Approximately 200 potential subjects will be pre-screened, with a target of completing 75 subjects: 45 symptomatic and 30 asymptomatic |
| Study Duration | The study will last approximately 5 months and include a 3-month enrollment period. |

| Anticipated Study | Subjects, ages 18-55 that are current spherical soft contact lens |
|---|---|
| Population | wearers are to complete this clinical study. |
| | Across sites approximately 200 potential subjects will be pre- |
| | screened, with a target of completing 45 in the symptomatic group |
| | (approximately 10 at VRC) and 30 in the asymptomatic group |
| | (approximately 10 at VRC). |
| | Symptomatology will be confirmed by a baseline CLDEQ-8 |
| | questionnaire (habitual lenses): |
| | Symptomatic: (CLDEQ- 8 score of 15 or greater) |
| El Tito Cit | Asymptomatic: (CLDEQ- 8 score of 7 or lower) |
| Eligibility Criteria | Potential subjects must satisfy all of the following criteria to be |
| | enrolled in the study: |
| | 1. The subject must read, understand, and sign the |
| | STATEMENT OF INFORMED CONSENT and receive a |
| | fully executed copy of the form |
| | 2. Appear able and willing to adhere to the instructions set forth |
| | in this clinical protocol |
| | 3. Between 18 and 55 (inclusive) years of age at the time of |
| | screening |
| | 4. Be a current soft contact lens wearer in both eyes with a |
| · | minimum of 3 days/week wear time over the last 1 month by |
| | self-report 5. Hove a baseline CLDEO 8 seems of eithers |
| | 5. Have a baseline CLDEQ-8 score of either: a) 7 or lower |
| | b) 15 or greater |
| | 6. Subjects must possess a functional / usable pair of spectacles |
| | and bring them to the visit (only if applicable to the |
| | investigators discretion). |
| | 7. Subjects must pass a pre-screening questionnaire |
| | 8. Subjects must be willing to discontinue all contact lens wear |
| | for approximately 1 week |
| | 9. Subjects must present to Visit 1 with their habitual lens on |
| | eye for at least 6 hours |
| | Inclusion Criteria after Baseline |
| | 1. The subject's vertex corrected spherical distance refraction |
| | must be in the range (+/-0.250 D) of -1.00 D to -6.50 D |
| | (inclusive) in each eye |
| | 2. The subject's vertex corrected refractive cylinder must be |
| | equal or less than -1.00 diopters in each eye |
| | 3. Have spherical best corrected visual acuity of 20/30 (0.20 |
| | LogMAR) or better in each eye |
| | • |

Potential subjects who meet any of the following criteria will be excluded from participating in the study:

- 1. Currently pregnant or lactating, by self-report
- 2. Any ocular or systemic allergies, disease or use of medication which may interfere with contact lens wear (at the discretion of the investigator).
- 3. Any active ocular abnormalities/conditions that may interfere with contact lens wear (at the discretion of the investigator).
- 4. Any corneal distortion resulting from previous hard or rigid gas permeable contact lens wear
- 5. Habitual contact lens wear modality as extended wear (≥1 night per month of extended wear)
- 6. Habitual contact lens is rigid gas permeable, toric, monovision or multi-focal
- 7. Any previous, or planned (during the course of the study) ocular surgery (e.g., radial keratotomy, PRK, LASIK, etc.)
- 8. Participation in any contact lens or lens care product clinical trial within 2 weeks prior to study enrollment.
- 9. Employee or employee's immediate family member of clinical site (e.g., Investigator, Coordinator, Technician)
- 10. Current habitual use of Restasis, Xiidra, ocular steroids, or any medication (Rx or over the counter (OTC)) that may interfere with contact lens wear (at the discretion of the investigator)

#### Exclusion Criteria after Baseline

- 11. Any ocular allergies, infections or other ocular abnormalities that are known to interfere with contact lens wear and/or participation in the study. This may include, but not be limited to entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, or corneal distortion
- 12. Any Grade 3 or greater biomicroscopy findings (this includes, corneal edema, corneal staining, corneal vascularization, conjunctival injection, tarsal abnormalities, bulbar injection) on the FDA classification scale (CTP-2018)

# Disallowed Medications/Interventions

Restasis, Xiidra, ocular steroids, or any medication (Rx or OTC) that may interfere with contact lens wear at the discretion of the investigator

| Measurements and | Objective clinical metrics: |
|---|---|
| Procedures | Physiology: Meibomian gland imaging, Meibomian gland expressibility, tear film lipid layer thickness, blink patterns, tear film stability, tear film lipid pattern, lid wiper epitheliopathy, conjunctival staining, conjunctival folds, lid margin evaluation Biomicroscopy Conjunctival Redness Expanded Corneal Staining Visual Acuity |
| | Subjective symptomatology: Questionnaires: CLDEQ-8, CLUE, MRD, Bare Eye, OSDI, and Sensitivity |
| Microbiology or Other | None |
| Laboratory Testing | |
| Study Termination | The occurrence of one or more Unanticipated Adverse Device Effect (UADE), or any SAE where relationship to study agent cannot be ruled out, will result in stopping further dispensing investigational product. |
| Ancillary Supplies/ | Lipiview |
| Study-Specific Materials | Korb Meibomian Gland Evaluator (MGE) |
| | Refresh ® Classic Lubricant Eye Drops Preservative Free and/or |
| | Refresh ® Lubricating Eye Drops Preservative Free |
| Principal Investigator(s) and Study | Study Sites: This study will be conducted at up to three clinical study sites, including VRC, Jacksonville FL and Centre for Contact Lens |
| Institution(s)/Site(s) | Research, University of Waterloo, Ontario. |
| | A full list of Principal Investigators, clinical sites, and institutions is kept separately from the Study Protocol and is included in the study Trial Master File. |

Figure 1: Study Flowchart



#### COMMONLY USED ABBREVIATIONS AND DEFINITIONS OF TERMS

ADD Plus Power Required for Near Use

ADE Adverse Device Effect

AE Adverse Event/Adverse Experience
BCVA Best Corrected Visual Acuity

BSCVA Best Spectacle Corrected Visual Acuity

CFR Code of Federal Regulations

CLDEQ-8 Contact Lens Dry Eye Questionnaire-8

CLUE Contact Lens User Experience

COAS Complete Ophthalmic Analysis System

COM Clinical Operations Manager CRA Clinical Research Associate

CRF Case Report Form

CRO Contract Research Organization

CT Center Thickness

CTP Clinical Technical Procedure

D Diopter

DEQ-5 Dry Eye Questionnaire- 5
DMC Data Monitoring Committee
eCRF Electronic Case Report Form
EDC Electronic Data Capture

ETDRS Early Treatment Diabetic Retinopathy Study

FDA Food and Drug Administration

GCP Good Clinical Practice

HIPAA Health Insurance Portability and Accountability Act

IB Investigator's Brochure ICF Informed Consent Form

ICH International Conference on Harmonization

IDE Investigational Device Exemption
IEC Independent Ethics Committee
IRB Institutional Review Board

ISO International Organization for Standardization

ITT Intent-to-Treat

JJVC Johnson & Johnson Vision Care, Inc.

LC Limbus Center

LIPCOF Lid Parallel Conjunctival Folds

LogMAR Logarithm of Minimal Angle of Resolution MedDRA<sup>©</sup> Medical Dictionary for Regulatory Activities

MOP Manual of Procedures
NIH National Institutes of Health

OD Right Eve

OHRP Office for Human Research Protections
OHSR Office for Human Subjects Research

OS Left Eye

OSDI Ocular Surface Disease Index

OU Both Eyes

PD **Protocol Deviation** Protected Health Information PHI PΙ Principal Investigator Patient Instruction Guide PIG **Product Quality Complaint POC** Patient Reported Outcome **PRO Quality Assurance QA** OC **Quality Control** SAE Serious Adverse Event/Serious Adverse Experience SAP Statistical Analysis Plan Statistical Analysis System SAS Standard Deviation SD SOP Standard Operating Procedure Unanticipated Adverse Device Effect **UADE** Unanticipated Serious Adverse Device Effect USADE VA Visual Acuity

#### 1. INTRODUCTION AND BACKGROUND

When exploring differences in characteristics between existing symptomatic and asymptomatic contact lens wearers, controlled clinical studies provide information on objective and subjective endpoints. Stratifying subjects into symptomatic and asymptomatic populations and measuring physiology and symptomatology aims to guide learning into the contact lens wearing experience. Past publications have found correlations between ocular symptoms and meibomian gland and lid margin endpoints.<sup>5-8</sup> The primary purpose of this clinical study is to evaluate objective endpoints and see if these measures have potential to differentiate symptomatic and asymptomatic contact lens wearers.<sup>9,10</sup>

#### 1.1. Name and Descriptions of Investigational Products

This study will use a single contact lens type: ACUVUE OASYS® 1-Day with HydraLuxe™ Technology is made of senofilcon A material, an FDA approved product. Further details about the test articles are found in Section 6 of this protocol.

#### 1.2. Intended Use of Investigational Products

The intended use of the investigative product is to compensate for myopia and hyperopia. During the study, each test article will be worn bilaterally in daily disposable modality for approximately 4 weeks.

#### 1.3. Summary of Findings from Nonclinical Studies

Not Applicable - Marketed product only

#### 1.4. Summary of Known Risks and Benefits to Human Subjects

The following risks/adverse events can be associated with wearing soft contact lenses in general:

- The eyes may burn, sting and/or itch.
- There may be a feeling of something in the eye (foreign body, scratched area).
- There may be the potential for some temporary impairment due to peripheral infiltrates, peripheral corneal ulcers and corneal erosion.
- There may be the potential for other physiological observations, such as local or generalized edema, corneal neovascularization, corneal staining, injection, tarsal abnormalities, iritis and conjunctivitis, some of which are clinically acceptable in low amounts.
- There may be excessive watering, unusual eye secretions, or redness of the eye.
- Poor visual acuity, blurred vision, rainbows or halos around objects, photophobia, or dry eyes may also occur if the lenses are worn continuously or for too long a time.

There is no direct benefit to the subject for participating in the study, although they will be able to try out marketed contact lenses. The information from this study aims to guide learning into the contact lens wearing experience of existing symptomatic and asymptomatic patients.

For the most comprehensive clinical information regarding ACUVUE OASYS® 1-Day with HydraLuxe<sup>TM</sup> Technology (senofilcon A) contact lenses, refer to the latest version of the package insert.

# 1.5. Relevant Literature References and Prior Clinical Data Relevant to Proposed Clinical Study

Many publications correlating objective ocular measures to symptoms exist. For this clinical study, we will mainly focus on the primary endpoints of lid wiper epitheliopathy, meibomian gland imaging, meibomian gland expressibility, lid margin evaluation, and conjunctival folds in subjects grouped by CLDEQ-8 scores.

The CLDEQ-8 is a validated outcome measure for soft contact lenses wearers. It has been highly correlated with habitual baseline status and change in overall opinion when subjects are refit with contact lenses. A CLDEQ-8 score of  $\geq$ 12 is proposed to identify contact lens wearers who could benefit from clinical management of their CL- related symptoms. A three-point change in CLDEQ-8 scores has also been shown to be clinically important. For this particular study, to ensure that we are recruiting symptomatic subjects we will have a CLDEQ cut off of  $\geq$ 15.

During this study, subjects will respond to subjective questionnaires investigating their symptomology both with contact lens wear (Visits 1, 2 & 3) and without (bare eye/spectacle wear) (Visit 4). Symptomology surveys associated with contact lens wear in this study include: CLDEQ-8, CLUE, and MRD. Symptomology surveys associated with bare eye/spectacle wear include: OSDI, MRD, and Bare Eye Questionnaire.



The Bare Eye Questionnaire is a non-validated questionnaire prepared specifically for this study and based on the questions of the DEQ-5<sup>15</sup>. The DEQ-5 questionnaire asks subjects to report their symptomology over the past month. To create the Bare Eye Questionnaire, each DEQ-5 question has been changed from "in the past month" to "since your last visit" to accommodate the 1 week bare eye period in this study. It will be scored in the same manner as the DEQ-5. Though this approach produces a non-validated questionnaire, it allows for similar questions to be asked throughout all study visits. Additionally, artificial tear/rewetting drop use and frequency will be asked verbally at all study visits.

The International Workshop on Meibomian Gland Dysfunction states that Meibomian Gland Dysfunction may well be the leading cause of dry eye disease throughout the world.<sup>5</sup> Through meibomian gland imaging, prior publications have investigated the number of functioning meibomian glands and found correlations to dryness symptoms.<sup>6,7</sup> Studies have also shown that the lid margins signs (rounding, notching, or vascularity of lid margins, hyperkeratinization, plugging of orifices, main duct dropout, and conjunctival congestion) all had a positive correlation with ocular symptoms.<sup>8</sup>

According to publications by Korb et al, lid wiper epitheliopathy is found significantly more often in symptomatic subjects than asymptomatic subjects.<sup>11</sup> Other publications have also found correlations between lid wiper epitheliopathy as well as conjunctival folds, specifically nasally located ones, and dry eye symptoms.<sup>12,13</sup>

For the most comprehensive clinical information regarding ACUVUE OASYS® 1-Day with HydraLuxe<sup>TM</sup> Technology (senofilcon A) contact lenses, refer to the latest version of the package insert (APPENDIX C: PACKAGE INSERT (APPROVED PRODUCT).

#### 2. STUDY OBJECTIVES, ENDPOINTS AND HYPOTHESES

#### 2.1. Objectives

**Primary Objectives:** 

There are two primary objectives of this study:

- 1. To explore the difference in characteristics between symptomatic and asymptomatic subjects with and without contact lenses utilizing the following metrics: Meibomian gland imaging, meibomian gland expressibility, lid margin evaluation, lid wiper epitheliopathy, and conjunctival folds.
- 2. Assess any change in clinical metrics throughout 4-weeks of ACUVUE OASYS® 1-Day with HydraLuxe™ Technology wear

#### Secondary Objective:

1) To explore the difference in characteristics between symptomatic and asymptomatic subjects in their habitual lenses utilizing the following metrics: corneal staining, conjunctival staining, conjunctival redness, team film lipid layer thickness, tear film stability, tear film lipid pattern

#### **Exploratory Objectives:**

Other observations will include additional parameters (slit lamp findings, entrance/exit visual acuity) and questionnaires (CLUE comfort, OSDI<sup>14</sup> Bare Eye<sup>15</sup>, Sensitivity<sup>16</sup>, and MRD).

#### 2.2. Endpoints

#### **Primary Endpoints:**

Meibomian gland imaging, meibomian gland expressibility, lid margin evaluation, Lid wiper epitheliopathy, and conjunctival folds.

Secondary Endpoints: conjunctival redness, conjunctival staining, corneal staining, tear film lipid layer thickness, tear film stability, tear film lipid pattern.

#### Other observations:

- 1. Blink patterns
- 2. Lens fit characteristics. This will be recorded by the investigator using
- 3. Lens surface characteristics. This will be recorded by the investigator using
- 4. Additional physiology characteristics. This will be recorded by the investigator using
- 5. Snellen or LogMAR Visual Acuity
- 6. Average daily and comfortable wear time
- 7. Reasons for discontinuation
- 8. Adverse events
- 9. Lens Damage
- 10. Subject reported ocular symptoms
- 11. CLUE Vision
- 12. Frequency of artificial/rewetting drop tear use
- 13. Questionnaires (CLUE comfort, MRD, OSDI Bare Eye, Sensitivity)

#### 2.3. Hypotheses

#### **Primary Hypothesis**

Due to the exploratory nature of this study no explicit hypothesis testing will be conducted. Instead tables or figures will accompany each objective for evaluation.

#### Secondary Hypothesis

Not applicable.

#### Other Hypothesis

Not applicable.

#### 3. TARGETED STUDY POPULATION

#### 3.1. General Characteristics

Subjects, ages 18-55 that are current spherical soft contact lens wearers are to complete this clinical study.

Across sites approximately 200 potential subjects will be pre-screened, with a target of completing 45 in the symptomatic group (approximately 10 at VRC) and 30 in the asymptomatic group (approximately 10 at VRC).

Symptomatology will be confirmed by a baseline CLDEQ-8 questionnaire (habitual lenses):

Symptomatic: (CLDEQ- 8 score of 15 or greater)

Asymptomatic: (CLDEQ- 8 score of 7 or lower)

#### 3.2. Inclusion Criteria

Potential subjects must satisfy all of the following criteria to be enrolled in the study:

- 1. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form
- 2. Appear able and willing to adhere to the instructions set forth in this clinical protocol
- 3. Between 18 and 55 (inclusive) years of age at the time of screening
- 4. Be a current soft contact lens wearer in both eyes with a minimum of 3 days/week wear time over the last 1 month by self-report
- 5. Have a baseline CLDEQ-8 score of either:
  - a) 7 or lower
  - b) 15 or greater
- 6. Subjects must possess a functional / usable pair of spectacles and bring them to the visit (only if applicable to the investigators discretion).
- 7. Subjects must pass a pre-screening questionnaire
- 8. Subjects must be willing to discontinue all contact lens wear for approximately 1 week
- 9. Subjects must present to visit 1 with their habitual lenses on eye for at least 6 hours

#### Inclusion Criteria after Baseline

- 10. The subject's vertex corrected spherical distance refraction must be in the range (+/-0.250 D) of -1.00 D to -6.50 D (inclusive) in each eye
- 11. The subject's vertex corrected refractive cylinder must be equal or less than -1.00 diopters in each eye
- 12. Have spherical best corrected visual acuity of 20/30 (0.20 LogMAR) or better in each eye

#### 3.3. Exclusion Criteria

Potential subjects who meet any of the following criteria will be excluded from participating in the study:

- 1. Currently pregnant or lactating, by self-report
- 2. Any ocular or systemic allergies, disease or use of medication which may interfere with contact lens wear (at the discretion of the investigator).
- 3. Any active ocular abnormalities/conditions that may interfere with contact lens wear (at the discretion of the investigator).

- 4. Any corneal distortion resulting from previous hard or rigid gas permeable contact lens wear
- 5. Habitual contact lens wear modality as extended wear (≥1 night per month of extended wear)
- 6. Habitual contact lens is rigid gas permeable, toric, monovision or multi-focal
- 7. Any previous, or planned (during the course of the study) ocular surgery (e.g., radial keratotomy, PRK, LASIK, etc.)
- 8. Participation in any contact lens or lens care product clinical trial within 2 weeks prior to study enrollment.
- 9. Employee or employee's immediate family member of clinical site (e.g., Investigator, Coordinator, Technician)
- 10. Current habitual use of Restasis, Xiidra, ocular steroids, or any medication (RX or OTC) that may interfere with contact lens wear (at the discretion of the investigator)

#### **Exclusion Criteria after Baseline**

- 11. Any ocular allergies, infections or other ocular abnormalities that are known to interfere with contact lens wear and/or participation in the study. This may include, but not be limited to entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, or corneal distortion
- 12. Any Grade 3 or greater biomicroscopy findings (this includes, corneal edema, corneal staining, corneal vascularization, conjunctival injection, tarsal abnormalities, bulbar injection) on the FDA classification scale

#### 3.4. Enrollment Strategy

Study subjects will be recruited from the Institution/clinical site's subject database and/or utilizing Independent Ethics Committee (IEC) or Institutional Review Board (IRB) approved materials. Subjects who have reported states of symptomatology and asymptomatology in previous contact lens clinical studies or surveys will initially be targeted for enrollment to improve enrollment efficiency. The clinical site will administer a pre-screening on potential subjects before they attend the initial study visit utilizing IEC/IRB approved recruitment materials. The pre-screening is not required if the subject has a CLDEQ-8 score on file with the clinical site for his/her current habitual contact lenses.

#### 4. STUDY DESIGN AND RATIONALE

#### 4.1. Description of Study Design

This is an unmasked, non-randomized, single arm, stratified, dispensing investigation of symptomatic and asymptomatic subject populations. Subjects will be assigned to a single study lens type to be worn bilaterally for approximately 4 weeks followed by no contact lens wear for approximately 1 week.

This study will be conducted at up to three clinical study sites, including VRC, Jacksonville FL and Centre for Contact Lens Research, University of Waterloo, Ontario. The time of day of each study visit shall occur within +/-2 hours of the time of the first visit.


#### 4.2. Study Design Rationale

The study has incorporated some features of the precursor study, stratified design is undertaken to explore the difference in characteristics between symptomatic and asymptomatic subjects while wearing habitual lenses, in addition to change that occurs when refit with ACUVUE OASYS® 1-Day with HydraLuxe<sup>TM</sup> Technology (senofilcon A).

#### 4.3. Enrollment Target and Study Duration

Subjects, ages 18-55 that are current spherical soft contact lens wearers are to complete this clinical study.

Across sites approximately 200 potential subjects will be pre-screened, with a target of completing 45 in the symptomatic group (approximately 10 at VRC) and 30 in the asymptomatic group (approximately 10 at VRC).

Symptomatology will be confirmed by a baseline CLDEQ-8 questionnaire (habitual lenses):

Symptomatic: (CLDEQ- 8 score of 15 or greater)

Asymptomatic: (CLDEQ- 8 score of 7 or lower)

The study will last approximately 5 months and include a 3-month enrollment period.

This study will be conducted at up to three clinical study sites, including VRC, Jacksonville FL and Centre for Contact Lens Research, University of Waterloo, Ontario.

Once the informed consent has been signed the subject will be considered enrolled.

#### 5. TEST ARTICLE ALLOCATION AND MASKING

#### 5.1. Test Article Allocation

The lenses will be worn in a bilateral fashion. Randomization is not applicable in this study due to the use of a single test article type.

The test article assignment of subjects must be performed at the Initial Visit. The following must have occurred prior to test article assignment:

- · Informed consent has been obtained
- Subject meets all the applicable inclusion/exclusion criteria
- Subject history and baseline information has been collected

#### 5.2. Masking

Not applicable. There will be no masking in this open labeled study.

### 5.3. Procedures for Maintaining and Breaking the Masking

Not applicable. There will be no masking in this open labeled study.

#### 6. STUDY INTERVENTION

### 6.1. Identity of Test Articles

The following contact lenses will be used in this study:

Table 1: Test Articles

| | Test 1 |
|---|---|
| Name | ACUVUE OASYS®1-Day with |
| | HydraLuxe™ Technology |
| Manufacturer | JJVC |
| Compass Protocol(s) and/or Lot Number or | 17CP1260 |
| Other Identifier* | |
| Lens Material | Senofilcon A |
| Nominal Base Curve @ 22°C | 8.5 |
| Nominal Diameter @ 22°C | 14.3 |
| Nominal Distance Powers (D) | -1.00 to -6.00 (0.25 steps), -6.50 |
| Nominal Cylinder Powers (D) and Axes | NA |
| Nominal ADD Powers (D) | NA |
| Center Thickness (Optional) | 0.085 |
| Oxygen Permeability (Dk) | 103.0 |
| Wear Schedule in Current Study | Daily Disposable |
| Replacement Frequency | Daily |
| Packaging Form (vial, blister, etc.) | Blister |
| Other distinguishing items (e.g., dye, | JJVC marketed and FDA approved |
| packaging solution, optical design, etc.) | production lenses |

Each subject assigned test article will wear lenses approximately 4 weeks and wear approximately 50-66 contact lenses.

# 6.2. Ancillary Supplies/Products

Table 2a: Ancillary Supplies-Instrumentation Equipment

| Instrumentation Equipment | | |
|---|---|---|
| Name | LipiView | Korb Meibomian Gland<br>Evaluator (MGE) |
| Manufacturer | TearScience | TearScience |
| Diagnostic test | Meibomian Gland Imaging Lipid Layer Thickness Blink Characteristics | Meibomian Gland<br>Expressibility |


Table 2b: Ancillary Supplies, Solution-Rinsing/Storage

| | Solution: Rinsing/Storage |
|-----------------------------------------|---------------------------|
| Solution Name/Description | Lacripure |
| Manufacturer | Menicon |
| Preservative | None |
| Other distinguishing items | NA |
| (dye, packaging, approval status, etc.) | |

Table 2c: Ancillary Supplies, Solution- Artificial Tears/ Rewetting Drops

The following solutions may be used equivalently in this study, as available in country of clinical study site:

| chincal study site. | | |
|---|---|---|
| | Solution: Artificial Tears/ Rewe | tting Drops |
| Salution Name/Description | Refresh ® Classic Lubricant | Refresh ® Lubricating Eye |
| Solution Name/Description | Eye Drops Preservative Free | Drops Preservative Free |
| Manufacturer | Allergan | Allergan |
| Preservative | None | None |
| Active Ingredients | Polyvinyl Alcohol 1.4%<br>Povidone 0.6% | Contains per mL: Polyvinyl alcohol 14 mg Povidone 6 mg |
| Other distinguishing items (dye, packaging, approval status, etc.) | Refresh Classic Lubricant Eye Drops 8. Sinche Use Conteners COTT OF DATE OF THE PROPERTY. | MILD DRYEYE Proceedings Fig. Refresh Lubricating Eye Drops For use with all confact lenses is of cond hard. |

#### 6.3. Administration of Test Articles

Test articles will be dispensed to subject meeting all eligibility requirements, including any dispensing requirements set forth in this clinical protocol. Subjects will be dispensed an adequate supply of test articles to complete the study. The lenses will be dispensed with right and left eye designation. Lost or damaged test articles may be replaced at the discretion of the Investigator and/or the Sponsor.

#### 6.4. Packaging and Labeling

The test articles will be packaged in blisters as the primary packaging. The test articles will be in cartons sealed with a tamper evident seal, commercial cartons, or in plastic bags as the secondary packaging form. The sample study labels are shown below:



#### 6.5. Storage Conditions

Test articles will be maintained at ambient temperatures at the clinical site. Test articles must be kept under secure conditions.

#### 6.6. Collection and Storage of Samples

When possible, any lens or test article associated with an Adverse Events and/or a Product Quality Complaint must be retained and stored in a glass vial with moderate solution pending directions from the sponsor for potential return to JJVC.

#### 6.7. Accountability of Test Articles

JJVC will provide the Investigator with sufficient quantities of study articles and supplies to complete the investigation. The Investigator is asked to retain all lens shipment documentation for the test article accountability records.

Test article must be kept in a locked storage cabinet, accessible only to those assigned by the Investigator for dispensing. The Investigator may delegate this activity to authorized study site personnel listed on the Site Delegation Log. All test articles must be accounted. This includes:

- 1. What was dispensed for the subject for trial fitting, to wear out of the office, or issued for the subject to replace appropriately between visits
- 2. What was returned to the Investigator unused
- 3. The number and reason for unplanned replacements

The Investigator will collect all unused test articles from the subjects at the end of the subject's participation. Subject returned unused test articles must be separated from the clinical study inventory of un-dispensed test articles, and must be labeled with the subject number and date of return. Following final reconciliation of test articles by the monitor, the Investigator or monitor will package and return all unused test articles to JJVC.



If there is a discrepancy between the shipment documents and the contents, contact the study monitor <u>immediately.</u>

Reference : Site Instructions for Test Article Receipt and Test Article Accountability for additional information.

#### 7. STUDY EVALUATIONS

#### 7.1. Time and Event Schedule

Table 5: Time and Events

| Event | Pre-Visit<br>Communication<br>(if applicable) | Visit<br>1 | Visit 2<br>(14±2<br>days<br>following<br>V1) | Visit 3<br>(14±2<br>days<br>following<br>V2) | BARE EYE<br>WASHOUT<br>(7±1 days) | Visit 4<br>(7±1 days<br>following<br>V3) |
|---|---|---|---|---|---|---|
| Subject<br>Identification | X | | | | | |
| Privacy Notice | X | | | | | |
| Study Informed<br>Consent | | X | | | | |
| Adverse Events Concomitant Review and Medical History review | | | X | Х | | Х |
| Demographics | | X | | | | |
| Medical History<br>& Concomitant<br>Medications | | Х | | | | |
| Habitual Contact<br>Lens Info | | Х | | | | |
| CL wear time | | X | X | X | | |
| Compliance | | X | X | X | | X |
| CLDEQ-8<br>Questionnaire | X | X | X | X | | |
| Sensitivity<br>Questionnaire | | Х | | | | |
| Eligibility after screening | | X | | | | |
| Subject<br>Classification | | X | | | | |

| Event | Pre-Visit<br>Communication<br>(if applicable) | Visit<br>1 | Visit 2<br>(14±2<br>days<br>following<br>V1) | Visit 3<br>(14±2<br>days<br>following<br>V2) | BARE EYE<br>WASHOUT<br>(7±1 days) | Visit 4<br>(7±1 days<br>following<br>V3) |
|---|---|---|---|---|---|---|
| Subject Reported<br>Ocular<br>Symptoms | | Х | Х | X | | Х |
| CLUE and MRD questionnaire | | X | X | X | | |
| Bare Eye<br>questionnaire | | | | | | Х |
| OSDI<br>questionnaire | | | | | | X |
| MRD<br>questionnaire | | | | | | X |
| Artificial Tear/Rewetting Drop Use Question | | X | Х | X | | X |
| Entrance Visual Acuity | | X | Х | X | | X |
| Tear film lipid<br>layer thickness | | Х | X | X | | X |
| Blink patterns | | X | X | X | | X |
| Meibomian<br>Gland Imaging | | X | | X | | X |
| Tear film<br>stability by<br>Medmont | | X | Х | X | | Х |
| Tear film lipid<br>pattern<br>(Tearscope) | | X | X | X | | X |
| Limbal &<br>Conjunctival<br>(Bulbar) Redness | | Х | X | Х | | X |
| Lens Wettability<br>Characteristics | | Х | X | Х | | · |
| Lens Surface<br>Deposits | | X | X | X | | |
| Subjective Lens<br>Fit Assessment | | X | Х | X | | |
| Lens Removal | | X | X | X | | *************************************** |
| Keratometry | | X | | | | |

| Event | Pre-Visit<br>Communication<br>(if applicable) | Visit<br>1 | Visit 2<br>(14±2<br>days<br>following<br>V1) | Visit 3<br>(14±2<br>days<br>following<br>V2) | BARE EYE<br>WASHOUT<br>(7±1 days) | Visit 4<br>(7±1 days<br>following<br>V3) |
|---|---|---|---|---|---|---|
| Subjective<br>Sphero-<br>cylindrical<br>Refraction | | X | | | | X |
| Subjective Best<br>Sphere<br>Refraction | | X | | | | |
| Lid wiper epitheliopathy | | X | X | X | | Х |
| Biomicroscopy | | X | X | X | | X |
| Expanded Sodium Fluorescein Corneal Staining | | X | Х | X | | Х |
| Lid margin<br>evaluation | | X | | X | | X |
| Conjunctival staining | | Х | X | X | | X |
| Conjunctival folds | | X | X | X | | X |
| Meibomian<br>gland<br>expressibility | | Х | | X | | X |
| Eye Rinse | | X | X | X | | X |
| Eligibility after<br>Baseline | | X | | | | |
| Lens Assignment | | X | | | | |
| Lens Insertion | | X | X | | | |
| Lens Settling | | X | | | | |
| Exit Visual Acuity | | X | X | X | | |
| Subjective Best<br>Sphere Over<br>Refraction | | X | | | | |
| Lens Power<br>Modification | | Х | | | | |
| Continuance | | X | X | X | | |
| Dispense<br>Instructions | | X | X | | | |

| Event | Pre-Visit<br>Communication<br>(if applicable) | Visit<br>1 | Visit 2<br>(14±2<br>days<br>following<br>V1) | Visit 3<br>(14±2<br>days<br>following<br>V2) | BARE EYE<br>WASHOUT<br>(7±1 days) | Visit 4<br>(7±1 days<br>following<br>V3) |
|---|---|---|---|---|---|---|
| Subject Instruction to discontinue contact lens wear | | | | X | | |
| Final Exam Form and Investigator Signature | | | | | | X |
| Study<br>Completion | | | | | | X |

# 7.2. Detailed Study Procedures

Pre-Visit Screening: If applicable (via phone or email)

| | | PRE- VISIT COMMUNICATION |
|---|---|---|
| Step | Procedure | Details |
| 1. | Preliminary Subject Identification | The clinical study site will search through their subject database to find potential subjects who may be eligible to participate. Subjects may be contacted by telephone or sent an electronic survey via email. |
| 2. | Subject's Privacy<br>Notice and<br>Disclosure | The clinical study site must provide notice to subjects regarding the collection and disclosure of personal information. Each subject must provide verbal consent by phone to allow the collection and disclosure of the personal information collected in the screening questionnaire. The verbal consent will be documented in the Screening Questionnaire. |
| 3. | CLDEQ-8<br>Questionnaire | Subject will be contacted by the clinical study site to complete a CLDEQ-8 questionnaire (which will be provided separately) over the phone or via email to determine preliminary eligibility. |

The subjects must present to Visit 1 wearing their habitual contact lenses for a minimum of 6 hours. Subjects will be asked to bring their habitual contact lens blisters and/or boxes with them to the visit.

| | | Visit 1: Screening |
|---|---|---|
| Step | Procedure | Details |
| 1.1 | Statement of Informed Consent | Each subject must read, understand, and sign the Statement of Informed Consent before being enrolled into the study. The Principal Investigator or his/her designee conducting the informed consent discussion must also sign the consent form. Note: The subject must be provided a signed |
| 1.2 | Demographics | copy of this document. Record the subject's date of birth, gender, race and ethnicity. |
| 1.3 | Medical History and<br>Concomitant<br>Medications | Questions regarding the subjects' medical history and concomitant medications. |
| 1.4 | Habitual Contact<br>Lenses | Questions regarding the subject's habitual contact lens type, parameters, wear schedule (frequency), replacement schedule, and care system (if any). |
| 1.5 | Current contact lens wear times | Record the mode of their current contact lens wear, as well as their habitual wear time (WT) and comfortable wear time (CWT). |
| 1.6 | Compliance | Confirm the subject's minimum wear time |
| 1.7 | CLDEQ-8<br>Questionnaire | The subject will respond to the CLDEQ-8 Questionnaire (Appendix A) |
| 1.8 | Artificial Tear/Rewetting Drop Use | The subject will be asked about their artificial tear/rewetting drop use. |
| 1.9 | Sensitivity Questionnaire | Subjects will respond to a Sensitivity Questionnaire (Appendix A) |
| 1.10 | Eligibility after<br>Screening | All responses to Screening Inclusion Criteria questions must be answered "yes" and all responses to Exclusion Criteria must be answered "no" for the subject to be considered eligible. |
| 1.11 | Subject<br>Classification | Symptomatic if (s)he: • Has a CLEDQ-8 score of 15 or greater. Asymptomatic if (s)he: • Has a CLEDQ-8 score of 7 or less |

| NOTE: Subjects who do not qualify as |
|----------------------------------------------------|
| symptomatic or asymptomatic will continue to |
| the final evaluation and be exited from the study. |

| | , | Visit 1: Baseline | |
|---|---|---|---|
| Step | Procedure | Details | |
| 1.12 | Subject Reported | Subjects will respond to a verbal open-ended | |
| | Ocular Symptoms | symptoms questionnaire. | |
| 1.13 | CLUE and MRD | The subject will respond to the CLUE and MRD | |
| | questionnaire | Baseline Questionnaire (Appendix A) | |
| 1.14 | Entrance Visual | Record the distance visual acuity (OD, OS) to | |
| | Acuity | the nearest letter with their habitual contact lens | |
| | | correction in place. Subjects must read the | |
| | | smallest line until at least 50% of the letters are | |
| 1 15 | 70 1 (71 | read incorrectly. | |
| 1.15 | Pre-lens tear film | Record the Pre-lens tear film lipid layer | Measure per |
| | lipid layer thickness | thickness, OD & OS | Lipiview II |
| | , | | manufacturer instruction |
| | · | | (Appendix D) |
| 1.16 | Blink Patterns | Record the Blink Patterns, OD & OS | Measure per |
| **** | | record the Blink I determs, OB & OB | Lipiview II |
| | | | manufacturer |
| | | | instruction |
| | | | (Appendix D) |
| 1.17 | Habitual Pre-lens | Record the Pre-lens tear film stability (NIBUT), | NIBUT |
| | tear film stability | OD & OS | Medmont |
| | (Medmont) | | Work Aid |
| 4.40 | | | (Appendix K) |
| 1.18 | Habitual Pre-lens | Record the Pre-lens tear film lipid pattern, OD | |
| | tear film lipid pattern | & OS | |
| 1.19 | (Tearscope) Habitual Lens | Limbal & Conjunctival (Bulbar) Redness (0.5 | |
| 1.19 | Related Limbal & | scale units) findings will be assessed using a | |
| | Conjunctival | more detailed scale for internal purposes only. | |
| | (Bulbar) Redness | more detailed sould for internal purposes only. | |
| 1.20 | Habitual Lens | Record the white light lens wettability of both | |
| | Wettability | lenses. | |
| | Characteristics | | |
| 1.21 | Habitual Lens | Record any front and back surface lens deposits. | |
| | Surface Deposits | | |
| 1.22 | Habitual Lens | Evaluate overall lens fit acceptance (acceptable | |
| | Subjective Lens Fit | or unacceptable) based on centration, movement | |
| | Assessment | and other fitting characteristics. | |

| | 1 | | |
|---|---|---|---|
| | | An unacceptable fit is deemed by one of the | |
| | | following criteria: | |
| | | <ul> <li>limbal exposure at primary gaze or with extreme eye movement;</li> </ul> | |
| | | edge lift; | |
| | | excessive movement in primary and up | |
| | | gaze; or | |
| | | • insufficient movement in all three of the | |
| | | following conditions: primary gaze, up | |
| | | gaze, and Josephson push up. | |
| 1.23 | Remove Habitual | The subject's habitual lenses will be removed | |
| | Contact Lenses | and discarded or stored as appropriate. | |
| 1.24 | Keratometry | Record the keratometry readings OD and OS in | |
| | | diopters. This can come from any appropriate | |
| | | instrument. | |
| 1.25 | Subjective Sphero- | Complete subjective spherocylindrical | |
| | cylindrical | refraction and record the resultant distance | |
| | Refraction | visual acuity (OD, OS) to the nearest letter. | |
| 1.26 | Subjective Best | Perform subjective best sphere refraction with a | |
| | Sphere Refraction | phoropter and record the best corrected distance | |
| 1.07 | <b>*</b> * | visual acuity (OD, OS) to the nearest letter. | E14'6 |
| 1.27 | Lid wiper | Record the lid wiper epitheliopathy (upper & | Evaluation of<br>LWE |
| | epitheliopathy | lower), OD & OS | (Appendix F) |
| | | | (Appendix 1) |
| 1.28 | Biomicroscopy | FDA Slit Lamp Classification Scale will be | |
| | | used to grade the findings and determine | |
| | | eligibility. | |
| | | If any of the security laws for divine and are do 2 are | |
| | | If any of these slit lamp findings are grade 3 or higher, the subject may not continue at this | |
| | | time, but may return up to one additional time to | |
| · | | determine eligibility. If discontinued a final | |
| | | examination must be completed. | |
| 1.29 | Expanded Sodium | Corneal Staining Assessment (1.0 scale units) | *************************************** |
| | Fluorescein Corneal | will be assessed using a more detailed scale for | <del></del> |
| | Staining | internal purposes only. | |
| 1.30 | Conjunctival staining | Record the conjunctival staining by sodium | |
| | | fluorescein only, OD & OS | |
| 1.31 | Conjunctival folds | Record the Conjunctival folds, OD & OS | LIPCOF |
| | | | Grading Scale |
| 1.00 | + 1 1 | D 14 C1 C1 1 11/2 1 | (Appendix G) |
| 1.32 | Lid margin | Record the presence of the following additional | |
| | Evaluation | biomicroscopy findings (upper & lower), OD & | |
| | | OS: | |

| | | <ul> <li>(no/normal or yes/abnormal):</li> <li>a) Irregularity: notching of margin</li> <li>b) Vascularity of lid margin: telangiectasia</li> <li>c) Meibomian gland pouting, plugging, or capping</li> <li>d) Lid/lash margin debris findings such as cylindrical dandruff or collarettes</li> </ul> | |
|---|---|---|---|
| 1.33 | Meibomian Gland<br>Expressibility<br>(Lower lid, 3<br>regions) | Record the Meibomian Gland Expressibility, OD & OS via Meibomian Gland Secretion Grading Scale (Appendix I) | Procedure per<br>Meibomian<br>Gland<br>Evaluator<br>manufacturer<br>instructions.<br>(Appendix H) |
| 1.34 | Eye Rinse | The study investigator or technician will rinse the subject's eyes thoroughly with a study provided solution. | |
| 1.35 | Meibomian Gland<br>Imaging (lower only) | Record the grading of the lower Meibomian gland images via the Meiboscale (Appendix E), OD & OS | Measure per<br>Lipiview II<br>manufacturer<br>instruction<br>(Appendix D) |
| 1.36 | Eligibility after<br>Baseline | All responses to Inclusion Criteria questions must be answered "yes" and all responses to Exclusion Criteria questions must be answered "no" for the subject to be considered eligible. | |

| | Visit 1: Treatment 1 Lens Fitting | |
|---|---|---|
| Step | Procedure | Details |
| 1.37 | Lens | All subjects will be assigned the study lens. |
| | Assignment | Select the closest available contact lens power |
| | | (+/-0.25D) based on the vertex corrected subjective |
| | | best sphere refraction. |
| 1.38 | Lens Insertion | The subject inserts the study lenses. |
| | | Check for lens damage under the slit lamp before |
| | | proceeding with lens settling. |
| | | Replace damaged lenses if applicable. |
| 1.39 | Lens Settling | Allow the study lenses to settle for a minimum of 5 |
| | | minutes. |
| 1.40 | Visual Acuity | Record the distance visual acuity with the contact |
| | | lenses (OD, OS) to the nearest letter. Subjects must |
| | | read the smallest line until at least 50% of the letters |
| | | are read incorrectly. |

| 1.41 | Subjective Best<br>Sphere Over<br>Refraction | Perform a spherical over-refraction OD and OS using any acceptable means (i.e., phoropter, trial lenses, flipper bars) in normal room illumination and record the resultant distance visual acuity OD and OS. $A \le +/-0.25$ D spherical over-refraction must be achieved to continue. |
|---|---|---|
| 1.42 | Lens Power<br>Modification (if<br>applicable) | Adjust the lens power if the subject's best sphere over-refraction is outside of plano or +/-0.25D. For each power modification, remove the lens, assign the new lens power, and repeat steps (1.37-1.42). Record the resultant distance visual acuity OD and OS. Up to <b>two</b> power modifications are allowed. |
| 1.43 | Subject<br>Reported<br>Ocular<br>Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire. |
| 1.44 | Study Lens Subjective Lens Fit Assessment | Evaluate overall lens fit acceptance (acceptable or unacceptable) based on centration, movement and other fitting characteristics. An unacceptable fit is deemed by one of the following criteria: Imbal exposure at primary gaze or with extreme eye movement; edge lift; excessive movement in primary and up gaze; or insufficient movement in all three of the following conditions: primary gaze, up gaze, and Josephson push up. |
| 1.45 | Study Lens<br>Wettability<br>Characteristics | Record the white light lens wettability of both lenses. |
| 1.46 | Study Lens Surface Deposits | Record any front and back surface lens deposits. |
| 1.47 | Continuance | For the subject to continue in the study, they must meet all three of the following criteria: • Visual acuity in test lenses is 20/30 (0.20 LogMAR) or better OD and OS • The lens fit is acceptable OD and OS |

| | | 1 70.1 7 |
|---|---|---|
| | | Investigator approval. If the Investigator |
| | | does not approve the dispensing of the study |
| | | lens, then the study is terminated for that |
| | | subject. |
| 1.48 | Dispense | The lenses will be dispensed for a 14±2 day wearing period. |
| | | Dispense enough lenses to last the subject to their scheduled follow-up visit. Do not dispense extras*. |
| | | The lenses will be dispensed with right and left eye designation. |
| | | The lenses will be worn as daily disposable only. |
| | | Study approved rewetting drops are permitted if needed. Dispense enough artificial |
| | | tears/rewetting drops to last the subject to their scheduled follow-up visit. Instruct the subject to track the approximate frequency of rewetting drop use. |
| | | Subjects may use reading glasses over contact lenses as needed |
| | | <ul> <li>A patient instruction guide will be provided.</li> <li>Subjects will be scheduled for Visit 2 in approximately 14 days, within +/-2 hours of the time of Visit 1, ensuring that they wear the study lens at least 6 hours/day each day.</li> </ul> |
| | | * Note: In the event a lens is lost or damaged, the subject will return to the clinical site for |
| | | replacement. As much as reasonably possible, a |
| | | damaged lens and packaging should be returned to |
| | | the clinical site (wet, if possible) and then returned to |
| | | the Sponsor. If lens damage is present, complete the |
| | | Product Quality Complaint Form, if applicable. The |
| | | lens will be stored in labeled vial with study |
| | | provided solution, and clearly differentiated from the |
| | | other worn lenses that will be shipped back to the |
| | | Sponsor. |



# VISIT 2: 2-week (±2) day after Visit 1 (Duration ~ 1.5 hour)

The time of day of each study visit shall occur within +/-2 hours of the time of the first visit

# Subjects will present with study lenses on eye following at least 6 hours of wear

| | Visit 2: Treatment 1 Follow-Up 1 | | | | | | |
|---|---|---|---|--|--|--|--|
| Step | Procedure | Details | | | | | |
| 2.1. | Adverse Events | Review the subject's adverse events and | | | | | |
| | Concomitant | concomitant medications and record any changes | | | | | |
| | Review and | from the previous study visit. | | | | | |
| | Medical History | Record any adverse events or medical history | | | | | |
| | review | changes from the previous study visit. | | | | | |
| 2.2. | Contact Lens | Record the present wearing time and comfortable | | | | | |
| | Wearing Time | wearing time. | | | | | |
| 2.3. | Compliance | Confirm compliance with the prescribed wear schedule. | | | | | |
| 2.4. | CLDEQ-8 | The subject will respond to the Contact Lens Dry | | | | | |
| | Questionnaire | Eye Questionnaire (Appendix A) | <u> </u> | | | | |
| 2.5. | Subject Reported | Subjects will respond to a verbal open-ended | | | | | |
| | Ocular Symptoms | symptoms questionnaire. | | | | | |
| 2.6. | CLUE and MRD | The subject will respond to the PRO Follow-Up | | | | | |
| | Questionnaire | Questionnaire (Appendix A) | | | | | |
| 2.7. | Artificial | The subject will be asked about their artificial | | | | | |
| | Tear/Rewetting | tear/rewetting drop use. | | | | | |
| | Drop Use | | - | | | | |
| 2.8. | Entrance Visual | Record the distance visual acuity with the contact | | | | | |
| | Acuity | lenses (OD, OS) to the nearest letter. Subjects must | | | | | |
| | | read the smallest line until at least 50% of the | | | | | |
| - | 7.1 | letters are read incorrectly. | | | | | |
| 2.9. | Pre-lens tear film | Record the Pre-lens tear film lipid layer thickness, | Measure per | | | | |
| | lipid layer | OD & OS | Lipiview II | | | | |
| | thickness | | manufacturer | | | | |
| | | | instruction | | | | |
| 0.10 | D1: 1 D // | D 14 DU 1 D OD 0 OG | (Appendix D) | | | | |
| 2.10. | Blink Patterns | Record the Blink Patterns, with Lipiview OD & OS | Measure per | | | | |
| | | | Lipiview II | | | | |
| | | | manufacturer | | | | |
| | | | instruction | | | | |
| 2 11 | Dua 1 C1 | December Due Language Class at a Little (AUDLIE) | (Appendix D) | | | | |
| 2.11. | | Record the Pre-lens tear film stability (NIBUT), | NIBUT<br>Modmont | | | | |
| | stability | OD & OS | Medmont | | | | |
| | (Medmont) | | Work Aid | | | | |
| | | | (Appendix K) | | | | |
| | T | | <u></u> |
|---|---|---|---|
| 2.12. | Pre-lens tear film lipid pattern (Tearscope) | Record the Pre-lens tear film lipid pattern, OD & OS | |
| 2.13. | | Limbal & Conjunctival (Bulbar) Redness (0.5 scale units) findings will be assessed using a more detailed scale for internal purposes only. | |
| 2.14. | Study Lens<br>Wettability<br>Characteristics | Record the white light lens wettability of both lenses. | |
| 2.15. | Study Lens Surface Deposits | Record any front and back surface lens deposits. | |
| 2.16. | Subjective Study Lens Fit Assessment | Evaluate overall lens fit acceptance (acceptable or unacceptable) based on centration, movement and other fitting characteristics. | |
| | | An unacceptable fit is deemed by one of the following criteria: | |
| | | <ul> <li>limbal exposure at primary gaze or with extreme eye movement;</li> <li>edge lift;</li> </ul> | |
| | | excessive movement in primary and up gaze; or | |
| | | <ul> <li>insufficient movement in all three of the<br/>following conditions: primary gaze, up<br/>gaze, and Josephson push up.</li> </ul> | |
| | | <u>Note:</u> if lens fit is unacceptable subject will be discontinued from the study. | |
| 2.17. | Lens Removal and Discard | The lenses will be removed and discarded for ocular physiological examination. | |
| 2.18. | Lid wiper epitheliopathy | Record the lid wiper epitheliopathy (upper/lower), OD & OS | Evaluation of LWE (Appendix F) |
| 2.19. | Biomicroscopy | FDA Slit Lamp Classification Scale will be used to grade the findings and determine eligibility. | |
| | | Adverse events shall be documented and followed for significant slit lamp findings. | |
| 2.20. | Expanded Sodium Fluorescein Corneal Staining | Corneal Staining Assessment (1.0 scale units) will be assessed using a more detailed scale for internal purposes only. | |
| 2.21. | Conjunctival staining | Record the conjunctival staining by sodium fluorescein only, OD & OS | |

| 2.22. | Conjunctival folds | Record the Conjunctival folds, OD & OS | LIPCOF Grading Scale (Appendix G) |
|---|---|---|---|
| 2.23. | Eye Rinse | The study investigator or technician will rinse the subject's eyes thoroughly with a study provided solution. | |
| 2.24. | Spectacle wear or Lens Insertion | The subject may wear spectacles or insert a new pair of study lenses, as desired. | |
| 2.25. | Exit Visual<br>Acuity | Record the distance visual acuity (OD, OS) to the nearest letter and correction used. Subjects must read the smallest line until at least 50% of the letters are read incorrectly. | |
| 2.26. | Continuance | For the subject to continue in the study, they must meet all three of the following criteria: • Entrance visual acuity in the test lenses is 20/30 (0.20 LogMAR) or better OD and OS • The lens fit is acceptable OD and OS • Investigator approval. | |
| 2.27. | Dispense | <ul> <li>The lenses will be dispensed for an additional 14±2 days wearing period. During this time, they are instructed to wear the lenses every day and at least 6 hours per day that they are worn.</li> <li>Dispense enough lenses to last the subject to their scheduled follow-up visit. Do not dispense extras*.</li> <li>The lenses will be dispensed with right and left eye designation.</li> <li>The lenses will be worn as daily disposable only.</li> <li>Rewetting drops are permitted if needed. Dispense enough artificial tears/rewetting drops to last the subject to their scheduled follow-up visit, if needed. Instruct the subject to track the approximate frequency of rewetting drop use.</li> <li>* Note: In the event a lens is lost or damaged, the</li> </ul> | |
| | | subject will return to the clinical site for replacement. As much as reasonably possible, a damaged lens and packaging should be returned to the clinical site (wet, if possible) and then returned to the Sponsor. If lens damage is present, complete the Product Quality Complaint Form. The lens will be stored in labeled vial with study provided solution, and clearly differentiated from the other | |

| worn lenses that will be shipped back to the |
|----------------------------------------------|
| Sponsor. |

# VISIT 3: 2-week (±2) day after Visit 2 (Duration ~ 1.5 hour)

The time of day of each study visit shall occur within +/-2 hours of the time of the first visit

# Subjects will present with study lenses on eye following at least 6 hours of wear

| | Visit 3: Treatment 1 Follow-Up 2 | | |
|---|---|---|---|
| Step | Procedure | Details | |
| 3.1. | Adverse | Review the subject's adverse events and concomitant | |
| | Events | medications and record any changes from the | |
| | Concomitant | previous study visit. | |
| | Review and | Record any adverse events or medical history | |
| | Medical | changes from the previous study visit. | |
| | History review | | |
| 3.2. | Contact Lens | Record the present wearing time and comfortable | |
| | Wearing Time | wearing time. | |
| 3.3. | Compliance | Confirm compliance with the prescribed wear | |
| | | schedule. | |
| 3.4. | Return any | Subjects will return any unused study lenses | |
| | unused study | | |
| | lenses | | |
| 3.5. | CLDEQ-8 | The subject will respond to the Contact Lens Dry | : |
| <u>.</u> | Questionnaire | Eye Questionnaire (Appendix A) | |
| 3.6. | Subject | Subjects will respond to a verbal open-ended | |
| | Reported | symptoms questionnaire. | |
| | Ocular | | |
| | Symptoms | | |
| 3.7. | CLUE and | The subject will respond to the CLUE and MRD | |
| | MRD | Questionnaire (Appendix A) | |
| | Questionnaire | | |
| 3.8. | Artificial | The subject will be asked about their artificial | |
| | Tear/Rewettin | tear/rewetting drop use | |
| 2.0 | g Drop Use | | |
| 3.9. | Entrance | Record the distance visual acuity with the contact | |
| | Visual Acuity | lenses (OD, OS) to the nearest letter. Subjects must | |
| | | read the smallest line until at least 50% of the letters | |
| 2.10 | B 1 | are read incorrectly. | |
| 3.10. | Pre-lens tear | Record the Pre-lens tear film lipid layer thickness, | Measure per |
| | film lipid layer | OD & OS | Lipiview II |
| | thickness | | manufacturer |
| | | | instruction |
| | | | (Appendix D) |

| 3.11. | Blink Patterns | Record the Blink Patterns, with Lipiview OD & OS | Measure per<br>Lipiview II<br>manufacturer<br>instruction<br>(Appendix D) |
|---|---|---|---|
| 3.12. | Pre-lens tear<br>film stability<br>(Medmont) | Record the Pre-lens tear film stability (NIBUT), OD & OS | NIBUT<br>Medmont<br>Work Aid<br>(Appendix K) |
| 3.13. | Pre-lens tear<br>film lipid<br>pattern<br>(Tearscope) | Record the Pre-lens tear film lipid pattern, OD & OS | |
| 3.14. | Study Lens Limbal & Conjunctival (Bulbar) Redness | Limbal & Conjunctival (Bulbar) Redness (0.5 scale units) findings will be assessed using a more detailed scale for internal purposes only. | |
| 3.15. | Study Lens Wettability Characteristics | Record the white light lens wettability of both lenses. | |
| 3.16. | Study Lens Surface Deposits | Record any front and back surface lens deposits. | |
| 3.17. | Subjective<br>Study Lens Fit<br>Assessment | Evaluate overall lens fit acceptance (acceptable or unacceptable) based on centration, movement and other fitting characteristics. | |
| | | An unacceptable fit is deemed by one of the following criteria: • limbal exposure at primary gaze or with extreme eye movement; • edge lift; | |
| | | <ul> <li>excessive movement in primary and up gaze; or</li> <li>insufficient movement in all three of the</li> </ul> | |
| | | following conditions: primary gaze, up gaze, and Josephson push up. | |
| | | Note: if lens fit is unacceptable subject will be discontinued from the study. | |
| 3.18. | Lens Removal | The lenses will be removed and discarded. | |
| 3.19. | Lid wiper epitheliopathy | Record the lid wiper epitheliopathy (upper/lower), OD & OS | Evaluation of LWE (Appendix F) |

| 3.20. | Biomicroscopy | FDA Slit Lamp Classification Scale will be used to grade the findings and determine eligibility. Adverse events shall be documented and followed | |
|---|---|---|---|
| | | for significant slit lamp findings. | |
| 3.21. | Expanded Sodium Fluorescein Corneal Staining | Corneal Staining Assessment (1.0 scale units) will be assessed using a more detailed scale for internal purposes only. | |
| 3.22. | Conjunctival staining | Record the conjunctival staining by sodium fluorescein only, OD & OS | |
| 3.23. | Conjunctival folds | Record the Conjunctival folds, OD & OS | LIPCOF Grading Scale (Appendix G) |
| 3.24. | Lid margin<br>Evaluation | Record the presence of the following additional biomicroscopy findings (upper & lower), OD & OS: (no/normal or yes/abnormal): a. Irregularity: notching of margin b. Vascularity of lid margin: telangiectasia c. Meibomian gland pouting, plugging, or capping d. Lid/lash margin debris findings such as cylindrical dandruff or collarettes | |
| 3.25. | Meibomian<br>Gland<br>Expressibility<br>(3 regions) | Record the Meibomian Gland Expressibility, OD & OS via Meibomian Gland Secretion Grading Scale (Appendix I) | Procedure per<br>Meibomian<br>Gland<br>Evaluator<br>manufacture<br>instructions.<br>(Appendix H) |
| 3.26. | Eye Rinse | The study investigator or technician will rinse the subject's eyes thoroughly with a study provided solution. | |
| 3.27. | Meibomian<br>Gland Imaging<br>(lower only) | Record the grading of the Meibomian gland images, OD & OS | Measure per<br>Lipiview II<br>manufacturer<br>instruction<br>(Appendix D) |
| 3.28. | Exit Visual<br>Acuity | Record the distance visual acuity (OD, OS) to the nearest letter and correction used (spectacles as appropriate). Subjects must read the smallest line until at least 50% of the letters are read incorrectly. | |

| 3.29. | Continuance | For the subject to continue in the study, they must meet the following criteria: | |
|---|---|---|---|
| | | <ul> <li>Subject must agree to discontinue all contact<br/>lens wear for 7±1 days.</li> </ul> | |
| | | Investigator approval. | 1 |
| 3.30. | Subject | Contact lens wear will be discontinued for 7±1 days. | |
| | Instruction | Rewetting drops are permitted if needed. Dispense enough artificial tears/rewetting drops to last the subject to their scheduled follow-up visit, if needed. Instruct the subject to track the approximate frequency of rewetting drop use. | |

# BARE EYE WASH OUT: 1 WEEK (7±1 Days)

VISIT 4: 7±1 Days after V3. (Visit Duration ~ 2 hour)

The time of day of each study visit shall occur within +/-2 hours of the time of the first visit.

# Subjects may present wearing spectacles, as appropriate after at least 6 waking hours.

| *********** | Visit 4: Bare eye follow-up | | |
|---|---|---|---|
| Step | Procedure | Details | |
| 4.1. | Adverse | Review the subject's adverse events and concomitant | |
| | Events | medications and record any changes from the | |
| | Concomitant | previous study visit. | |
| | Review and | Record any adverse events or medical history | |
| | Medical | changes from the previous study visit. | |
| | History review | | |
| 4.2. | Compliance | Confirm that subjects have not worn contact lens | |
| | | since the last visit. | |
| | | If the subject is non-compliant, complete the Final | |
| | | Evaluation. | - <u>-</u> |
| 4.3. | Subject | Subjects will respond to a verbal open-ended | |
| | Reported | symptoms questionnaire. | |
| | Ocular | | |
| | Symptoms | | |
| 4.4. | Bare Eye | The subject will respond to the Bare Eye | |
| | Questionnaire | Questionnaire (Appendix A) | |
| 4.5. | OSDI | The subject will respond to the OSDI Questionnaire | |
| | Questionnaire | (Appendix A) | |
| 4.6. | MRD | The subject will respond to the MRD Questionnaire | |
| | Questionnaire | (Appendix A) | |

| 4.7. | Artificial | The subject will be asked about artificial | |
|---|---|---|---|
| | Tear/Rewettin<br>g Drop Use | tear/rewetting drop use. | |
| 4.8. | Entrance<br>Visual Acuity | Record the distance visual acuity with the contact lenses (OD, OS) to the nearest letter. Subjects must read the smallest line until at least 50% of the letters are read incorrectly. | |
| 4.9. | Bare Eye tear<br>film lipid layer<br>thickness | Record the Bare Eye tear film lipid layer thickness, OD & OS | Measure per<br>Lipiview II<br>manufacturer<br>instruction<br>(Appendix D) |
| 4.10. | Blink Patterns | Record the Blink Patterns, OD & OS | Measure per<br>Lipiview II<br>manufacturer<br>instruction<br>(Appendix D) |
| 4.11. | Bare Eye tear film stability (Medmont) | Record the Bare Eye tear film stability (NIBUT), OD & OS | NIBUT<br>Medmont<br>Work Aid<br>(Appendix K) |
| 4.12. | Bare Eye tear film lipid pattern (Tearscope) | Record the Pre-lens tear film lipid pattern, OD & OS | |
| 4.13. | Limbal &<br>Conjunctival<br>(Bulbar)<br>Redness | Limbal & Conjunctival (Bulbar) Redness (0.5 scale units) findings will be assessed using a more detailed scale for internal purposes only. | |
| 4.14. | Lid wiper epitheliopathy | Record the lid wiper epitheliopathy (upper/lower), OD & OS | Evaluation of LWE (Appendix F) |
| 4.15. | Biomicroscopy | FDA Slit Lamp Classification Scale will be used to grade the findings and determine eligibility. Adverse events shall be documented and followed for significant slit lamp findings. | |
| 4.16. | Expanded Sodium Fluorescein Corneal Staining | Corneal Staining Assessment (1.0 scale units) will be assessed using a more detailed scale for internal purposes only. | |
| 4.17. | Conjunctival staining | Record the conjunctival staining by sodium fluorescein only, OD & OS | |

| 4.18. | Conjunctival | Record the Conjunctival folds, OD & OS | LIPCOF |
|---|---|---|---|
| 4.10. | Conjunctival | Record the Conjunctival folds, OD & OS | |
| | folds | | Grading Scale |
| | | | (Appendix G) |
| 4.19. | Lid margin | Record the presence of the following additional | |
| | Evaluation | biomicroscopy findings (upper & lower), OD & OS: | |
| | | (no/normal or yes/abnormal): | |
| | | a. Irregularity: notching of margin | |
| | | b. Vascularity of lid margin: telangiectasia | |
| | | c. Meibomian gland pouting, plugging, or | |
| | | capping | |
| | | d. Lid/lash margin debris findings such as | |
| | | cylindrical dandruff or collarettes | |
| 4.20. | Meibomian | Record the Meibomian Gland Expressibility, OD & | Procedure per |
| 7.20. | Gland | OS via Meibomian Gland Secretion Grading Scale | Meibomian |
| | Expressibility | (Appendix I) | Gland |
| | | (Appendix I) | Evaluator |
| | (3 regions) | | manufacturer |
| | | | instructions. |
| | | we shallow. | (Appendix H) |
| 4.21. | Eye Rinse | The study investigator or technician will rinse the | |
| | | subject's eyes thoroughly with a study provided | |
| | | solution. | |
| 4.22. | Meibomian | Record the grading of the Meibomian gland images, | Measure per |
| | Gland Imaging | OD & OS | Lipiview II |
| | (lower only) | | manufacturer |
| | <b>`</b> | | instruction |
| | | | (Appendix D) |

#### FINAL EVALUATION

The final evaluation will ordinarily take place immediately following the last scheduled follow-up visit per the study protocol. It may also take place at any point the subject discontinues the study or is terminated from the study. If the subject is a screen-failure and a refraction and /or biomicroscopy procedure has just been performed, you may intentionally blank out these forms at the final evaluation in EDC

| Final Evaluation | | |
|---|---|---|
| Step | Procedure | Details |
| F.1 | Final Exam<br>Form | Indicate if the subject completed the study successfully. If subject discontinued from the study indicate the reason. |
| F.2 | Subjective<br>spherocylindrical<br>Refraction | Perform bare-eye subjective spherocylindrical refraction with a phoropter and record the best corrected <u>distance</u> visual acuity to the nearest letter (OD, OS, OU). |
| F.3 | Exit Slit Lamp<br>Biomicroscopy | FDA Slit Lamp Classification Scale will be used to grade the findings. If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops may be instilled. |

#### 7.3. Unscheduled Visits

If, during the investigation, a subject requires an unscheduled visit to the clinical site, the following information will be collected as applicable:

- Chief complaint prompting the visit. If the reason is an adverse event, the applicable eCRF for the adverse event must be completed and subject record completed as appropriate
- Date and time of the visit and all procedures completed at the unscheduled visit
- Review of adverse event and concomitant medications
- Documentation of any test article dispensed or collected from the subject, if applicable
- Slit lamp findings (using the Slit Lamp Classification Scale)

If the Investigator withdraws a subject from the study, the final study visit case report forms must be completed indicating the reason(s) why the subject was withdrawn. The subject record must be completed documenting the date and primary reason for withdrawal and the study CRA notified.

Any ocular and non-ocular Adverse Events that are ongoing at the time of the study visit will be followed by the Investigator, within licensure, until they have resolved, returned to pretreatment status, stabilized, or been satisfactorily explained. If further treatment i.e., beyond licensure is required, the subject will be referred to the appropriate health care provider.

The following information will be collected during an unscheduled visit.

| Step | Procedure | Details | |
|---|---|---|---|
| U.1 | Chief Complaints | Record the subject's chief complaints for | |
| | | reasons for the unscheduled visit | |
| U.2 | Change of | Questions regarding the change of subjects' | |
| | Medical History | medical history and concomitant medications. | : |
| | and Concomitant | | |
| | Medications | | |
| U.3 | Entrance VA | Record the entrance distance visual acuity (OD, | |
| | 0.11 | OS) to the nearest letter. | |
| U.4 | Subjective Sphero- | Perform bare-eye subjective spherocylindrical | |
| | cylindrical | refraction with a phoropter (adopt the | |
| | Refraction | maximum plus to maximum visual acuity | |
| | | (MPMVA) approach and use the duo-chrome | |
| | | test for binocular balancing) and record the best | |
| | | corrected distance visual acuity to the nearest | |
| U.5 | Clit I ama | letter (OD, OS, OU). FDA Slit Lamp Classification Scale will be | |
| 0.5 | Slit Lamp<br>Biomicroscopy | used to grade the findings. If no slit lamp | |
| | Diomicroscopy | finding is noted on the EDC form it is | |
| | | considered as a zero "0" grade for all | |
| | | observations listed. | |
| | | After the slit lamp examination, at the | |
| | | discretion of the Investigator, rinse the | |
| | | subject's eyes thoroughly with study provided | |
| | | solution. | |
| U.6 | Dispensing | Dispense replacement lens(es) and/or artificial | |
| | | tears/rewetting drops as needed | |
| U.7 | Exit Visual Acuity | Record the subject's exit distance visual acuity | 55001409810514 |
| | _ | (OD, OS and OU) to the nearest letter with the | |
| | | subjects wearing the study provided contact | |
| | | lenses or spectacle glasses (as applicable). | |

# 7.4. Laboratory Procedures

Not Applicable.

## 8. SUBJECTS COMPLETION/WITHDRAWAL

## 8.1. Completion Criteria

Subjects are considered to have completed the study if they:

- Provided informed consent;
- Are eligible;
- Completed all assigned study visits.

• Have not withdrawn/discontinued from the study for any reason described in Section 8.2

## 8.2. Withdrawal/Discontinuation from the Study

A subject will be withdrawn from the study for any of the following reasons:

- Subject death during the study period
- Subject withdrawal of consent
- Subject not compliant to protocol
- Subject lost to follow-up
- Subject no longer meets eligibility criteria (e.g. the subject becomes pregnant)
- Subject develops significant or serious adverse events causing discontinuation of study lens wear
- Subjects who have experienced a Corneal Infiltrative Event (CIE)
- Investigator's clinical judgment regarding the subject safety reasons (that it is in the best interest of the subject to stop treatment)

For discontinued subjects, the Investigator will make every effort to obtain:

- Complete the current visit (scheduled or unscheduled)
- Complete the Final Evaluation, indicating the reason that the subject was discontinued from the study
- Record the spherocylindrical refraction with best corrected distance visual acuity (when applicable)
- Collect used test article(s) (worn or brought to the visit) from the subject and discard them, unless otherwise stated in Section 7.2
- Collect all unused test article(s) from the subject

An additional subject may be enrolled if a subject discontinues from the study prematurely.

In cases where a subject is lost to follow-up, every possible effort must be made to contact the subject and determine the reason for discontinuation/withdrawal. The measures taken to follow up must be documented including two written attempts and a certified letter (or equivalent) as the final attempt.

#### 9. PRE-STUDY AND CONCOMITANT INTERVENTION/MEDICATION

Concomitant medications will be documented during screening and updated during the study. Disallowed medications for this study include: Restasis, Xiidra, ocular steroids, or any medication (RX or OTC) that may interfere with contact lens wear (at the discretion of the investigator).

Concomitant therapies that are disallowed include: Not applicable.

## 10. DEVIATIONS FROM THE PROTOCOL

Investigator will notify study sponsor upon identification of a protocol deviation. Major protocol deviations must be reported to the sponsor within 24 hours after discovery of the

protocol deviation. The Investigator will report deviations per IRB/IEC requirements. All deviations will be tracked and corrective actions implemented as appropriate.

If it becomes necessary for the Investigator to implement a deviation in order to eliminate an immediate hazard to the trial subject, the Investigator may implement the deviation immediately without notification to the sponsor. Within 24 hours after the implemented deviation, the Investigator must notify and provide the rationale to the Sponsor and, as required, the IEC/IRB.

#### 11. STUDY TERMINATION

The occurrence of one or more Unanticipated Serious Adverse Device Effect (USADE), or any SAE where the relationship to study agent cannot be ruled out, may result in stopping further dispensing of test article.

The Sponsor will determine when a study will be stopped. The Principal Investigator always has the discretion to initiate stopping the study based on patient safety or if information indicates the study's results are compromised.

JJVC reserves the right to terminate the study at any time for any reason. Additionally, the IEC/IRB reserves the right to terminate the study if an unreasonable risk is determined. The study can be terminated by the Principal Investigator at the individual clinical site due to specific clinical observations, if in their opinion, after a discussion with JJVC, it is determined that it would be unwise to continue at the clinical site.

JJVC (and the IEC/IRB and DMC, if applicable) will evaluate all adverse events. If it is determined that an adverse event presents an unreasonable risk, the investigation, or that part of the investigation presenting the risk, will be terminated, as soon as possible.

Should the study be terminated (either prematurely or as scheduled), the Investigator will notify the IEC/IRB and Regulatory Authority as required by local regulatory requirements.

## 12. PROCEDURE FOR HANDLING PRODUCT QUALITY COMPLAINTS

A Product Quality Complaint (PQC) refers to any written, electronic, or oral communication that alleges deficiencies related to the identity, quality, durability, reliability, safety, effectiveness or performance of test articles after they have been released for clinical trial use.

Potential complaints may come from a variety of sources including but not limited to subjects, clinical research associates (CRA), clinical operations managers (COM), medical monitors, and site personnel, etc. The following are not considered product quality complaints:

- Subject satisfaction inquiries reported via "Subjective Questionnaires" and "Patient Reported Outcomes (PRO)"
- Clinical test articles that are stored improperly or damaged after receipt at the investigational site
- Lens replacements that occur due to drops/fall-outs



• Damage deemed by clinicians or clinical staff to be caused by handling by the user, and not indicative of a quality deficiency (i.e. tears, rips, etc.), only in situations where there is no deficiency alleged by the subject

Within 24 hours of site personnel becoming aware that a PQC has occurred, the PQC must be recorded in the EDC system, which will trigger an automatic email notification to the appropriate COM/CRA and Clinical QA representative. In cases where the EDC system in use is not configured to send automatic notifications or when an EDC system is not used, the COM/CRA is responsible for notifying Clinical QA upon discovery that a PQC has occurred.

Upon receipt of the EDC notification, the COM/CRA will contact the study site to collect additional information which will include:

- Date the complaint was received/recorded in the EDC System (Date of Sponsor Awareness)
- Who received the complaint
- Study number
- Clinical site information (contact name, site ID, telephone number)
- Lot number(s)
- Unique Subject Identifier(s)
- Indication of who first observed complaint (site personnel or subject)
- OD/OS indication, along with whether or not the lens was inserted
- Any related AE number if applicable
- Detailed complaint description (scheduled/unscheduled visit, wear time, symptoms, resolution of symptoms, etc.)
- Eye Care Provider objective (slit lamp) findings if applicable
- Confirmation of product availability for return (and tracking information, if available), or rationale if product is not available for return (Refer to for test article return instructions)

Once a complaint is received, it will be assessed by the COM, CRA, or trained site personnel to determine if it is an Adverse Event/Serious Adverse Event (AE/SAE). If the complaint results in an AE/SAE, the COM/CRA, or trained site personnel will follow Section 13 of this protocol. If the AE/SAE was potentially the result of a product quality related deficiency, these procedures also applies and will be executed in parallel.

In some cases, a PQC form may be generated in EDC by the site in error. In this event, the PQC forms will be marked "Intentionally Left Blank" or "ILB". Justification for ILB must be documented.

## 13. ADVERSE EVENTS

#### 13.1. Definitions and Classifications

**Adverse Event (AE)** – An AE is "any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the investigational medical device.

*Note 1* to entry: This definition includes events related to the investigational medical device or the comparator.

Note 2 to entry: This definition includes events related to the procedures involved.

*Note 3* to entry: For users or other persons, this definition is restricted to events related to investigational medical devices."

An AE includes any condition (including a pre-existing condition) that:

- 1. Was not present prior to the study, but appeared or reappeared following initiation of the study
- 2. Was present prior to the study, but worsened during the study. This would include any condition resulting from concomitant illnesses, reactions to concomitant medications, or progression of disease states
- 3. Pregnancy must be documented as an adverse event and must be reported to the clinical monitor and to the Sponsor immediately upon learning of the event

## Serious Adverse Event (SAE) – An SAE is any untoward medical occurrence that:

- Results in death
- Is life threatening
- Requires in-patient hospitalization or prolongation of existing hospitalization
- Results in persistent or significant disability/incapacity (e.g., a sight threatening event, a significant persistent or permanent change, impairment, damage, or disruption to the subject's body)
- Is a congenital anomaly/birth defect, or
- Requires intervention to prevent permanent damage (the use of the test article resulting in a condition which requires medical or surgical intervention to preclude permanent impairment of the body structure or a body function). Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered an SAE when, based upon appropriate medical judgment, they may jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the outcomes listed in the above definition

Diagnoses and conditions that are considered Ocular Serious Adverse Events include, but not limited to:

- Microbial Keratitis (MK)
- Iritis (including cells in the anterior chamber)
- Permanent decrease in best spectacle corrected visual acuity equivalent to 2 acuity lines or greater
- Central Corneal Opacity
- Central Corneal Neovascularization
- Uveitis
- Endophthalmitis
- Hypopyon
- Hyphemia
- Penetration of Bowman's Membrane
- Persistent Epithelial Defect

• Limbal cell Damage leading to Conjunctivalization

Significant Adverse Events – Those events that are usually symptomatic and warrant discontinuation (temporary or permanent) of the test article (excluding Serious Adverse Events).

Diagnoses and conditions that are considered Ocular Significant Adverse Events include, but not limited to the following:

- Contact Lens Induced Peripheral Ulcer (CLPU)
- Significant Infiltrative Events (SIE)
- Superior Epithelial Arcuate Lesions (SEALs)
- Any Temporary Loss of >2 Lines of BSCVA
- Other grade 3 or higher corneal findings, such as abrasions or edema
- Non-contact lens related corneal events e.g. Epidemic Keratoconjunctivitis (EKC)
- Asymptomatic Corneal Scar
- Any corneal event which necessitates temporary lens discontinuation > 2 weeks

**Non-Significant Adverse Events** – Those conditions that are usually asymptomatic and usually do not warrant discontinuation (temporary or permanent) of the test article. However, the Investigator may choose to treat as a precautionary measure.

Diagnoses and conditions that are considered Ocular Non-Significant Adverse Events include, but not limited to the following:

- Non-significant Infiltrative Event (NSIE)
- Contact Lens Papillary Conjunctivitis (CLPC)
- Superficial Punctate Keratitis (SPK)
- Conjunctivitis: Bacterial, Viral, Allergic
- Blepharitis
- Meibomianitis
- Contact Dermatitis
- Localized Allergic Reactions
- Any corneal event not explicitly defined as serious or significant adverse event, which necessitates temporary lens discontinuation <2 weeks

**Adverse Device Effect (ADE)** – An ADE is an "adverse event related to the use of an investigational medical device.

*Note 1* to entry: This definition includes adverse events resulting from insufficient or inadequate instructions for use, deployment, implantation, installation, or operation, or any malfunction of the investigational medical device.

*Note 2* to entry: This definition includes any event resulting from use error or from intentional misuse of the investigational medical device."

Unanticipated Adverse Device Effect (UADE) – Any serious adverse effect on health or safety or any life-threatening problem or death caused by, or associated with, the test article, if that effect, problem, or death was not previously identified in nature, severity, or degree of

incidence in the investigational plan, Investigator's Brochure or protocol, or any other unanticipated serious problem associated with the test article that relates to the rights, safety and welfare of subjects.

## 13.2. Assessing Adverse Events

In conjunction with the medical monitor, the Investigator will evaluate adverse events to ensure the events are categorized correctly. Elements of categorization will include:

- Seriousness/Classifications (see definition in Section 13.1)
- Causality or Relatedness i.e. the relationship between the test article, study treatment or study procedures and the adverse event (not related; unlikely related; possibly related; related see definition in Section 13.2.1)
- Adverse Event Severity Adverse event severity is used to assess the degree of
  intensity of the adverse event (mild; moderate; severe for all events see definition in
  Section 0)
- Outcome not recovered or not resolved; recovering or resolving; recovered or resolved with sequelae; recovered or resolved; death related to adverse event; unknown
- Actions Taken none; temporarily discontinued; permanently discontinued; other action taken

## 13.2.1. Causality Assessment

Causality Assessment – A determination of the relationship between an adverse event and the test article. The test article relationship for each adverse event should be determined by the investigator using these explanations:

- Not Related- An adverse event that is not related to the use of the test article, study treatment or study procedures
- Unlikely Related An adverse event for which an alternative explanation is more likely, e.g. concomitant treatment, concomitant disease(s), or the relationship of time suggests that a causal relationship is not likely
- Possibly Related An adverse event that might be due to the use of the test article, or to the study treatment or study procedures. An alternative explanation, e.g. concomitant treatment, concomitant disease(s), is inconclusive. The relationship in time is reasonable. Therefore, the causal relationship cannot be excluded
- Related An adverse event that is listed as a possible adverse effect (device) or adverse reaction (drug) and cannot be reasonably explained by an alternative explanation, e.g. concomitant treatment of concomitant disease(s). The relationship in time is very suggestive, e.g. it is confirmed by de-challenge and re-challenge

#### 13.2.2. Severity Assessment

Severity Assessment – A qualitative assessment of the degree of intensity of an adverse event as determined by the Investigator or reported to him/her by the subject. The assessment of severity is made irrespective of test article, study treatment or study procedure relationship or seriousness of the event and should be evaluated according to the following scale:

• Mild – Event is noticeable to the subject, but is easily tolerated and does not interfere with the subject's daily activities

- Moderate Event is bothersome, possible requiring additional therapy, and may interfere with the subject's daily activities
- Severe Event is intolerable, necessitates additional therapy or alteration of therapy and interferes with the subject's daily activities

## 13.3. Documentation and Follow-Up of Adverse Events

The recording and documenting of adverse events (ocular and non-ocular) begins when the subjects are exposed to the test article, study treatment or study procedure. Adverse events reported before the use of test article, start of study treatment, or study procedures will be recorded as medical history. However, if the condition deteriorates at any time during the study it will be recorded and reported as an AE. Untoward medical events reported after the subject's exit from the study will be recorded as adverse events at the discretion of the Investigator.

Upon finding an adverse event, the Principal Investigator will document the condition in the subject record and in the eCRFs. He/she will complete the Adverse Event /eCRF.

Complete descriptions of all adverse events must be available in the subject record. All Adverse Events including local and systemic reactions not meeting the criteria for "serious adverse events" shall be captured on the appropriate case report form or electronic data system. All adverse events occurring while the subject is enrolled in the study must be documented appropriately regardless of relationship.

It is the Investigator's responsibility to maintain documentation of each reported adverse event. All adverse events will be followed in accordance with applicable licensing requirements. Such documentation will include the following:

- Adverse event (diagnosis not symptom)
- Drawings or photographs (where appropriate) that detail the finding (e.g., size, location, and depth, etc.)
- Date the clinical site was notified
- Date and time of onset
- Date and time of resolution
- Adverse event classification, severity, and relationship to test articles, as applicable
- Treatment regimen instituted, including concomitant medications prescribed, in accordance with applicable licensing requirements
- Any referral to another health care provider if needed
- Outcome, ocular damage (if any)
- Likely etiology
- Best corrected visual acuity at the discovery of the event and upon conclusion of the event

In addition, if an infiltrate(s) is present, he/she will complete the Corneal Infiltrate Assessment eCRF. Where necessary, a culture of the corneal lesion will be collected to determine if the infection is microbial in nature. If cultures are collected, the date of culture collection and laboratory utilized will be recorded.

Changes in the severity of an AE shall be documented to allow an assessment of the duration of the event at each level of intensity to be performed. Adverse events characterized as intermittent require documentation of the onset and duration of each episode. Changes in the assessment of relationship to the Test Article shall also be clearly documented.

Subjects who present with an adverse event shall be followed by the Investigator, within licensure, until all signs and symptoms have returned to pre-treatment status, stabilized, or been satisfactorily resolved. If further treatment beyond licensure is required, the patient will be referred to the appropriate health care provider. The Investigator will use his/her clinical judgment as to whether or not a subject reporting with an adverse event will continue in the study. If a subject is discontinued from the study, it will be the responsibility of the Investigator to record the reason for discontinuation. The Investigator will also document the adverse event appropriately and complete the Adverse Event eCRF. Any subjects with ongoing adverse events related to the test article, study treatment or study procedures, as of the final study visit date, should be followed to resolution of the adverse event or until referral to an appropriate health care provider, as recommended by the Investigator. Non-ocular adverse events that are not related to the test article, study treatment, or study procedures may be recorded as "ongoing" without further follow-up.

#### 13.4. Reporting Adverse Events

The Investigator will notify the Sponsor of an adverse event by e-mail, facsimile, or telephone as soon as possible and no later than 24 hours from discovery for any serious/significant adverse events, and 2 days from discovery for any non-significant adverse event. In addition, a written report will be submitted by the Principal Investigator to the IEC/IRB according to their requirements (Section 13.4.2). The report will comment whether or not the adverse event was considered to be related to the test article, study treatment or study procedures.

## 13.4.1. Reporting Adverse Events to Sponsor

#### Serious/Significant Adverse Events

The Investigator will inform the sponsor of all serious/significant adverse events occurring during the study period as soon as possible by e-mail, fax, or telephone, but no later than 24 hours following discovery of the event. The Investigator is obligated to pursue and obtain information requested by the Sponsor in addition to that information reported on the eCRF. All subjects experiencing a serious/significant adverse event must be followed up and all outcomes must be reported.

When medically necessary, the Investigator may break the randomization code to determine the identity of the treatment that the subject received. The Sponsor and study monitor should be notified prior to unmasking the test articles.

In the event of a serious/significant adverse event, the Investigator must:

- Notify the Sponsor immediately
- Obtain and maintain in the subject's records all pertinent medical information and medical judgment for colleagues who assisted in the treatment and follow-up of the subject

- Provide the Sponsor with a complete case history which includes a statement as to whether the event was or was not related to the use of the test article
- Notify the IEC/IRB as required by the IEC/IRB reporting procedure according to national regulations

## **Unanticipated (Serious) Adverse Device Effect (UADE)**

In the event of an Unanticipated (Serious) Adverse Device Effect (UADE), the Investigator will submit a report of the UADE to the Sponsor and IEC/IRB as soon as possible, but no later than 24 hours after the Investigator first learns of the effect. This report is in addition to the immediate notification mentioned above.

The Sponsor must conduct an evaluation of the UADE and must report the results of the evaluation to FDA, the IEC/IRB and participating Investigators within 10 working days after the Sponsor first receives notification of the effect.

#### **Non-Serious Adverse Events**

All non-serious adverse events, including non-serious adverse device effects, will be reported to the sponsor by the Investigator no later than 2 days from discovery.

## 13.4.2. Reporting Adverse Events to the Responsible IEC/IRB and Health Authorities

Adverse events that meet the IEC/IRB requirements for reporting must be reported within the IEC/IRB's written guidelines. Each clinical site will refer to and follow any guidelines set forth by their Approving IEC/IRB. Each clinical site will refer to and follow any guidelines set forth by their local governing Health Authorities.

The Sponsor will report applicable Adverse Events to the local health authorities according the written guidelines, including reporting timelines.

#### 13.4.3. Event of Special Interest

None

## 13.5. Reporting of Pregnancy

Subjects reporting pregnancy (by self-report) during the course of the study will be discontinued after the event is recorded as an Adverse Event. Once discontinued, pregnant participants and their fetuses will not be monitored for study related purposes. At the Investigator's discretion, the study participant may be followed by the Investigator through delivery. However, this data will not be collected as part of the clinical study database. Pregnant participants are not discontinued from contact lens or solution related studies for safety concerns, but due to general concerns relating to pregnancy and contact lens use. Specifically, pregnant women are discontinued due to fluctuations in refractive error and/or visual acuity that occur secondary to systemic hormonal changes, and not due to unforeseen health risks to the mother or fetus.

#### 14. STATISTICAL METHODS

#### 14.1. General Considerations

Statistical Analysis will be undertaken by the sponsor or under the authority of the sponsor. A general description of the statistical methods to be implemented in this clinical trial is outlined below.

All data summaries and statistical analyses will be performed using the SAS software Version 9.4 or higher (SAS Institute, Cary, NC). Throughout the analysis of data, the results for each subject/eye will be used when available for summarization and statistical analysis. Unscheduled visits will be summarized separately and will be excluded from the statistical analysis.

Summary tables (descriptive statistics and/or frequency tables) will be provided for all baseline variables, efficacy variables and safety variables as appropriate. Continuous variables will be summarized with descriptive statistics (n, mean, standard deviation (SD), median, minimum and maximum). Frequency count and percentage of subjects or eyes within each category will be provided for categorical data.

Safety variables will be summarized on the safety population whereas efficacy variables will be summarized on the analysis population.

## 14.2. Sample Size Justification

Approximately 75 subjects are targeted to complete the study. Most of the primary endpoints in the current study have sparse historical data. A similar study however, did evaluate lid wiper epitheliopathy between asymptomatic and symptomatic CLDEQ-8 subjects. Because one objective of the current study is to determine which metrics are best at discriminating CLDEQ-8 symptomatology, a sample size calculation was conducted to determine the minimum number of subjects needed for each group in order to detect a significant difference in lid wiper epitheliopathy (asymptomatic vs symptomatic).

Using data from the dependent variable used this for this sample size calculation was defined in the following manner:

- a) Subjects were categorized into asymptomatic (CLDEQ-8 total score ≤10) or symptomatic (CLDEQ-8 total score ≥20).
- b) For each subject, the final lid wiper epitheliopathy grade was determined by taking the mean grade across four sectors: horizontal upper lid, horizontal lower lid, sagittal upper lid, and sagittal lower lid. For example, if a subject had grades of 1.0, 0.5, 1.0, and 0.0, respectively, then his final grade would be 0.625.
- c) A binary variable was created: 1 = final lid wiper epitheliopathy grade worsened from baseline to 14-hour follow-up and 0 = final lid wiper epitheliopathy grade equaled or improved from baseline to 14-hour follow-up.

Interim analyses for found that approximately 50% of asymptomatic subjects had a worse lid wiper epitheliopathy final grade from baseline to 14-hour follow-up, whereas 80% of symptomatic subjects had a worse lid wiper epitheliopathy final grade. Using these

proportions, an alpha level = .05, and power = .80, a Fisher's Exact Conditional Test for Two Independent Proportions revealed that 37 subjects per group would be needed to detect a significant difference in the proportion of worsening. This amounts to a total of 74 subjects, which closely matches the study goal of targeting 75 subjects to complete the study.

Ideally subjects would be recruited on a 1:1 ratio but in this study, a greater proportion of symptomatic subjects are being recruited, anticipating greater interpatient variability in the symptomatic population.

Because lid wiper epitheliopathy is only one of the exploratory metrics to be examined, the total sample size is not dependent on merely this one endpoint. Hence, an approximation of 30 asymptomatic and 45 symptomatic subjects will be sufficient for the current study's objectives.

## 14.3. Analysis Populations

All subjects who were administered any test article excluding subjects who drop out prior to administering any test article. At least one observation should be recorded.

#### **Safety Population:**

All subjects who were administered any test article excluding subjects who drop out prior to administering any test article. At least one observation should be recorded.

## **Per-Protocol Population:**

All subjects who have successfully completed all visits and did not substantially deviate from the protocol as determined by the trial cohort review committee prior to database hard lock (Per-Protocol Population). Justification of excluding subjects with protocol deviations in the per-protocol population set will be documented in a memo to file.

#### 14.4. Level of Statistical Significance

All planned analysis for this study will be conducted with an overall type I error rate of 5%. No adjustment for multiple comparisons will be conducted unless specified otherwise.

#### 14.5. Primary Analysis

Descriptive tables or figures will be provided for all objective clinical metrics.

In addition, a logistic regression model will be analyzed using CLDEQ-8 group (asymptomatic vs symptomatic) as a dependent variable and all primary and secondary endpoints as fixed effects. These endpoints will be transformed into z scores so that they can all be compared on a similar scale. Endpoints will be ranked on which showed the best potential to differentiate asymptomatic and symptomatic subjects. This will be determined by plotting each regression coefficient with 95% confidence intervals as a function of CLDEQ-8 group.

## Primary safety analysis:

The maximum grades of any biomicroscopy finding will be reported descriptively with clinically significant grades being assessed at Grade 3 or higher.



#### 14.6. Secondary Analysis

Not applicable

## 14.7. Other Exploratory Analyses

Descriptive tables or figures will be provided for all subjective symptomatology.

Other efficacy analysis: Not applicable

Other safety analysis: Not applicable

## 14.8. Interim Analysis

Not Applicable

## 14.9. Procedure for Handling Missing Data and Drop-Outs

Missing or spurious values will not be imputed. The count of missing values will be included in the summary tables and listings.

Subject dropout is expected to be one of the main reasons of missing data in this clinical trial. Past clinical trials don't provide the evidence that subject dropout is systematic or not-at-random. To evaluate the impact of missing data, sensitivity analysis will be conducted using multiple imputation methods if the proportion of subject dropout is greater than the 15%.

## 14.10. Procedure for Reporting Deviations from Statistical Plan

The analysis will be conducted according to that specified in above sections. There are no known reasons for which it is planned to deviate from these analysis methods. If for any reason a change is made, the change will be documented in the study report along with a justification for the change.

#### 15. DATA HANDLING AND RECORD KEEPING/ARCHIVING

#### 15.1. Electronic Case Report Form/Data Collection

The data for this study will be captured on electronic case report forms (eCRFs) using an EDC system BioClinica. An authorized data originator will enter study data into the eCRFs using the EDC system.

The clinical data will be recorded on dedicated eCRFs specifically designed to match the study procedures for each visit. Once completed, the eCRFs will be reviewed for accuracy and completeness and signed by the Investigator.

The sponsor or sponsor's representatives will be authorized to gain access to the subject recordation for the purposes of monitoring and auditing the study.

Edit checks, electronic queries, and audit trails are built into the system to ensure accurate and complete data collection. Data will be transmitted from the clinical site to a secure central database as forms are completed or updated, ensuring information accuracy, security, and confidentiality. After the final database lock, the Investigator will be provided with Individual

Patient Profiles (IPP) including the full audit trail on electronic media in PDF format for all of the study data. The IPP must be retained in the study files as a certified copy of the source data for the study.

The content and structure of the eCRFs are compliant with ISO14155:2011. 1

## 15.2. Subject Record

At a minimum, subject record should be available for the following:

- subject identification
- eligibility
- study identification
- study discussion
- provision of and date of informed consent
- visit dates
- results of safety and efficacy parameters as required by the protocol
- a record of all adverse events
- follow-up of adverse events
- medical history and concomitant medication
- test article receipt/dispensing/return records
- date of study completion
- reason for early discontinuation of test article or withdrawal from the study, if applicable

The subject record is the eCRF or an external record. The author of an entry in the subject record must be identifiable. The first point of entry is considered to be the source record.

Adverse event notes must be reviewed and initialed by the Investigator.

#### 16. DATA MANAGEMENT

#### 16.1. Access to Source Data/Document

The Investigator/Institution will permit trial-related monitoring, audits, IEC/IRB review and regulatory inspection(s) by providing direct access to source data/documents. Should the clinical site be contacted for an audit by an IEC/IRB or regulatory authority, JJVC must be contacted and notified in writing within 24 hours.

#### 16.2. Confidentiality of Information

Information concerning the investigational product and patent application processes, scientific data or other pertinent information is confidential and remains the property of JJVC. The Investigator may use this information for the purposes of the study only. It is understood by the Investigator that JJVC will use information developed in this clinical study in connection with the development of the investigational product and therefore may disclose it as required to other clinical investigators and to regulatory agencies. In order to allow the use of the information derived from this clinical study, the Investigator understands that he/she

has an obligation to provide complete test results and all data developed during this study to the Sponsor.

## 16.3. Data Quality Assurance

Steps will be taken to ensure the accuracy and reliability of data, include the selection of qualified investigators and appropriate clinical sites and review of protocol procedures with the Principal Investigator. The Principal Investigator, in turn, must ensure that all Sub-Investigators and clinical site personnel are familiar with the protocol and all study-specific procedures and have appropriate knowledge of the study article.

Training on case report form completion will be provided to clinical site personnel before the start of the study. The Sponsor will review case report forms for accuracy and completeness remotely during the conduct of the study, during monitoring visits, and after transmission to data management. Any data discrepancies will be resolved with the Investigator or designee, as appropriate.

Quality Assurance representatives from JJVC may visit clinical sites to review data produced during the study and to access compliance with applicable regulations pertaining to the conduct of clinical trials. The clinical sites will provide direct access to study-related source data/documents and reports for the purpose of monitoring and auditing by JJVC and for inspection by local and regulatory authorities.

#### 17. MONITORING

The study monitors will maintain close contact with the Principal Investigator and the Investigator's designated clinical site personnel. The monitor's responsibilities will include:

- Ensuring that the investigation is being conducted according to the protocol, any subsequent amendments, and regulatory requirements are maintained
- Ensuring the rights and wellbeing of subjects are protected
- Ensuring adequate resources, including facilities, laboratories, equipment, and qualified clinical site personnel
- Ensuring that protocol deviations are documented with corrective action plans, as applicable
- Ensuring that the clinical site has sufficient test article and supplies
- Clarifying questions regarding the study
- Resolving study issues or problems that may arise
- Reviewing of study records and source documentation verification in accordance with the monitoring plan

#### 18. ETHICAL AND REGULATORY ASPECTS

## 18.1. Study-Specific Design Considerations

Potential subjects will be fully informed of the risks and requirements of the study and, during the study, subjects will be given any new information that may affect their decision to continue



participation. Subjects will be told that their consent to participate in the study is voluntary and may be withdrawn at any time with no reason given and without penalty or loss of benefits to which they would otherwise be entitled. Only subjects who are fully able to understand the risks, benefits, and potential adverse events of the study, and provide their consent voluntarily will be enrolled.

## 18.2. Investigator Responsibility

The Principal Investigator is responsible for ensuring that the clinical study is performed in accordance with the signed agreement, the investigational plan, Section 4 of the ICH E6 guidelines on Good Clinical Practice (GCP),<sup>2</sup> and applicable regulatory requirements. GCP is an international ethical and scientific quality standard for designing, conducting, recording, and reporting studies that involve the participation of human subjects. Compliance with this standard provides public assurance that the rights, safety, and well-being of study subjects are protected, consistent with the principles of the Declaration of Helsinki 64<sup>th</sup> WMA General Assembly 2013<sup>3</sup> and that the clinical study data are credible. The Investigator must maintain clinical study files in accordance with Section 8 of the ICH E6 guidelines on Good Clinical Practice (GCP),<sup>2</sup> and applicable regulatory requirements.

## 18.3. Independent Ethics Committee or Institutional Review Board (IEC/IRB)

Before the start of the study, the Investigator (or Sponsor when applicable) will provide the IEC/IRB with current and complete copies of the following documents (where applicable):

- Final protocol and, if applicable, amendments
- Sponsor-approved informed consent form (and any other written materials to be provided to the subjects)
- Investigator's Brochure (or equivalent information) and amendments
- Sponsor-approved subject recruitment materials
- Information on compensation for study-related injuries or payment to subjects for participation in the study
- Investigator's curriculum vitae, clinical licenses, or equivalent information (unless not required, as documented by IEC/IRB)
- Information regarding funding, name of the Sponsor, institutional affiliations, other potential conflicts of interest, and incentives for subjects
- Any other documents that the IEC/IRB requests to fulfill its obligation

This study will be undertaken only after IEC/IRB has given full approval of the final protocol, amendments (if any), the informed consent form, applicable recruiting materials, and subject compensation programs, and the Sponsor has received a copy of this approval. This approval letter must be dated and must clearly identify the documents being approved.

During the study the Investigator (or Sponsor when applicable) will send the following documents to the IEC/IRB for their review and approval, where appropriate:

- Protocol amendments
- Revision(s) to informed consent form and any other written materials to be provided to subjects
- If applicable, new or revised subject recruitment materials approved by the Sponsor

- Revisions to compensation for study-related injuries or payment to subjects for participation in the study
- Investigator's Brochure amendments or new edition(s)
- Summaries of the status of the study (at least annually or at intervals stipulated in guidelines of the IEC/IRB)
- Reports of adverse events that are serious, unanticipated, and associated with the test articles, according to the IRB's requirements
- New information that may adversely affect the safety of the subjects or the conduct of the study
- Major protocol deviations as required by the IEC/IRB
- Report of deaths of subjects under the Investigator's care
- Notification if a new Investigator is responsible for the study at the clinical site
- Any other requirements of the IEC/IRB

For protocol amendments that increase subject risk, the amendment and applicable informed consent form revisions must be submitted promptly to the IEC/IRB for review and approval before implementation of the change(s).

At least once a year, the IEC/IRB will review and reapprove this clinical study. This request should be documented in writing.

At the end of the study, the Investigator (or Sponsor where required) will notify the IEC/IRB about the study completion. Documentation of this notification must be retained at the clinical site and a copy provided to the CRO or Sponsor as applicable.

#### 18.4. Informed Consent

Each subject must give written consent according to local requirements after the nature of the study has been fully explained. The consent form must be signed before performance of any study-related activity. The consent form that is used must be approved by both the Sponsor and by the reviewing IEC/IRB. The informed consent is in accordance with principles that originated in the Declaration of Helsinki,<sup>3</sup> current ICH<sup>2</sup> and ISO 14155<sup>1</sup> guidelines, applicable regulatory requirements, and Sponsor Policy.

Before entry into the study, the Investigator or an authorized member of the clinical site personnel must explain to potential subject the aims, methods, reasonably anticipated benefits, and potential hazards of the study, and any discomfort it may entail. Subjects will be informed that their participation is voluntary and that they may withdraw consent to participate at any time.

The subject will be given sufficient time to read the informed consent form and the opportunity to ask questions. After this explanation and before entry into the study, consent should be appropriately recorded by means of the subject's dated signature. After having obtained the consent, a copy of the informed consent form must be given to the subject.

Each subject for this study will complete an assent and a parent or legal guardian must give written informed consent according to local requirements after the nature of the study has



been fully explained. The assent and consent forms must be signed before performance of any study-related activity. The assent and consent forms that are used must be approved by both the Sponsor and by the reviewing IEC/IRB. The assent and informed consent forms should be in accordance with principles that originated in the Declaration of Helsinki, current ICH and GCP guidelines, applicable regulatory requirements, and Sponsor policy. Before entry into the study or pre-screening, the Investigator or an authorized member of the clinical site personnel must explain to the potential subject and parent and/or legal guardian the aims, methods, reasonably anticipated benefits, and potential hazards of the study or pre-screening, and any discomfort it may entail. Subjects and parent and/or legal guardian will be informed that their participation is voluntary and that they may withdraw consent to participate at any time. They will be informed that choosing not to participate will not affect the care the subject Finally, they will be told that the Investigator will maintain a subject will receive. identification register for the purposes of long-term follow-up if needed and that their records may be accessed by health authorities and authorized Sponsor personnel without violating the confidentiality of the subject, to the extent permitted by the applicable law(s) or regulations. By signing the assent and informed consent form, the subject is authorizing such access and agrees to be contacted after study completion by health authorities and authorized Sponsor personnel for the purpose of obtaining consent for additional safety evaluations if needed.

## 18.5. Privacy of Personal Data

The collection, processing and disclosure of personal data and medical information related to the Study Subject, and personal data related to Principal Investigator and any clinical site personnel (e.g., name, clinic address and phone number, curriculum vitae) is subject to compliance with the Data Protection Act of 1998 and other applicable personal data protection and security laws and regulations. Appropriate measures will be employed to safeguard these data, to maintain the confidentiality of the person's related health and medical information, to properly inform the concerned persons about the collection and processing of their personal data, to grant them reasonable access to their personal data and to prevent access by unauthorized persons.

All information obtained during the course of the investigation will be regarded as confidential. All personal data gathered in this trial will be treated in strictest confidence by Investigators, monitors, Sponsor's personnel and IEC/IRB. No data will be disclosed to any third party without the express permission of the subject concerned, with the exception of Sponsor personnel (monitor, auditor), IEC/IRB and regulatory organizations in the context of their investigation related activities that, as part of the investigation will have access to the CRFs and subject records.

The collection and processing of personal data from subjects enrolled in this study will be limited to those data that are necessary to investigate the efficacy, safety, quality, and utility of the investigational product(s) used in this study.

These data must be collected and processed with adequate precautions to ensure confidentiality and compliance with applicable data privacy protection laws and regulations. The Sponsor ensures that the personal data will be:

- processed fairly and lawfully
- collected for specified, explicit, and legitimate purposes and not further processed in a way incompatible with these purposes
- adequate, relevant, and not excessive in relation to said purposes
- accurate and, where necessary, kept current

Explicit consent for the processing of personal data will be obtained from the participating subject before collection of data. Such consent should also address the transfer of the data to other entities and to other countries.

The subject has the right to request through the Investigator access to his personal data and the right to request rectification of any data that are not correct or complete. Reasonable steps should be taken to respond to such a request, taking into consideration the nature of the request, the conditions of the study, and the applicable laws and regulations.

Appropriate technical and organizational measures to protect the personal data against unauthorized disclosures or access, accidental or unlawful destruction, or accidental loss or alteration must be put in place. Sponsor personnel whose responsibilities require access to personal data agree to keep the identity of study subjects confidential.

#### 19. STUDY RECORD RETENTION

In compliance with the ICH/GCP guidelines,<sup>2</sup> the Investigator/Institution will maintain all CRFs and all subject records that support the data collected from each subject, as well as all study documents as specified in ICH/GCP<sup>2</sup> and all study documents as specified by the applicable regulatory requirement(s). The Investigator/Institution will take measures to prevent accidental or premature destruction of these documents.

Essential documents must be retained until at least two (2) years after the last approval of a marketing application in an ICH region and until there are no pending or contemplated marketing applications in an ICH region or until at least two (2) years have elapsed since the formal discontinuation of clinical development of the investigational product. These documents will be retained for a longer period if required by the applicable regulatory requirements or instructed by the Sponsor. It is the responsibility of the Sponsor to inform the Investigator/Institution as to when these documents no longer need to be retained.

If the responsible Investigator retires, relocates, or for other reasons withdraws from the responsibility of keeping the study records, custody must be transferred to a person who will accept the responsibility. The Sponsor must be notified in writing of the name and address of the new custodian. Under no circumstance shall the Investigator relocate or dispose of any study documents before having obtained written approval from the Sponsor.

If it becomes necessary for the Sponsor or the appropriate regulatory authority to review any documentation relating to this study, the Investigator must permit access to such reports. If the Investigator has a question regarding retention of study records, he/she should contact JJVC.



#### 20. FINANCIAL CONSIDERATIONS

Remuneration for study services and expenses will be set forth in detail in the Clinical Research Agreement. The Research Agreement will be signed by the Principal Investigator and a JJVC management representative prior to study initiation.

JJVC reserves the right to withhold remuneration for costs associated with protocol violations such as:

- Continuing an ineligible subject in the study
- Scheduling a study visit outside the subject's acceptable visit range

JJVC reserves the right to withhold final remuneration until all study related activities have been completed, such as:

- Query resolution
- Case Report Form signature
- Completion of any follow-up action items

#### 21. PUBLICATION

This study will be registered on ClinicalTrials.gov.

#### 22. REFERENCES

See Investigator Brochure for additional references and prior data.

- 1. ISO 14155:2011: Clinical Investigation of Medical Devices for Human Subjects Good Clinical Practice. Available at: https://www.iso.org/standard/45557.html
- 2. International Conference on Harmonization Good Clinical Practice E6 (ICH-GCP). Available at: <a href="http://www.ich.org/products/guidelines/efficacy/article/efficacy-guidelines.html">http://www.ich.org/products/guidelines/efficacy/article/efficacy-guidelines.html</a>
- 3. Declaration of Helsinki Ethical principles for Medical Research Involving Human Subjects. Available at: <a href="https://www.wma.net/policies-post/wma-declaration-of-helsinki-ethical-principles-for-medical-research-involving-human-subjects/">https://www.wma.net/policies-post/wma-declaration-of-helsinki-ethical-principles-for-medical-research-involving-human-subjects/</a>
- 4. United States (US) Code of Federal Regulations (CFR). Available at: <a href="https://www.gpo.gov/fdsys/browse/collectionCfr.action?collectionCode=CFR">https://www.gpo.gov/fdsys/browse/collectionCfr.action?collectionCode=CFR</a>
- 5. Nichols KK, Foulks GN, Bron AJ, et al. The International Workshop of meibomian Gland Dysfunction: Executive Summary. *Invest Ophthalmol Vis Sci.* 2011;52:1922-1929.
- 6. Srinivasan S, Menzies K, Sorbara L, Jones L. Infrared imaging of meibomian gland structure using a novel keratography. *Optom Vis Sci.* 2012;89:788-794.
- 7. Korb DR, Blackie CA. Meibomian gland diagnostic expressibility: correlation with dry eye symptoms and gland location. *Cornea*. 27:1142-1147.
- 8. Song H, Zhang M, Hu X, Li K, Jiang X, Liu Y, Lv H, Li X. Correlation Analysis of Ocular Symptoms and Signs in Patients with Dry Eye. *Journal of Ophthalmology*. 2017, Article ID 1247138. (lid eval)
- 9. Chalmers R, Begley CG, Moody K, Hickson-Curran SB. Contact Lens Dry Eye Questionnaire-8 (CLDEQ-8) and option of contact lens performance. *Optom Vis Sci.* 2010;10:1435-1442.

- 10. Chalmers R, Keay L, Hickson-Curran SB, Gleason WJ. Cutoff score and responsiveness of the 8-item Contact Lens Dry Eye Questionnaire (CLDEQ-8) in a Large daily disposable contact lens registry. *Contact Lens & Anterior Eye*. 2016;39: 342-352
- 11. Korb DR, Herman, JP, Greiner JV, Scaffidi RC, Finnemore VM, Exford JM, Blackie CA, Douglass T. Lid Wiper Epitheliopathy and Dry Eye Symptoms. *Eye and Contact Lens*. 2005;31:2-8.
- 12. Chhadva, P. et al. The Impact of Conjunctivochalasis on Dry Eye Symptoms and Signs. *Investigative Ophthalmology & Visual Science*. 2015;56.5:2867–2871.
- 13. Pult H, Purslow C, Murphy PJ. The relationship between clinical signs and dry eye symptoms. *Eye.* 2011;25:505-510.
- 14. Schiffman RM, Christianson MD, Jacobsen G, Hirsch JD, Reis BL. Reliability and validity of the Ocular Surface Disease Index. *Arch Ophthalmol.* 2000;118:615-621.
- 15. Chalmers RL, Begley CG, Caffery B. Validation of the 5-Item Dry Eye Questionnaire (DEQ-5): Discrimination across self-assessed severity and aqueous tear deficient dry eye diagnoses. *Cont Lens Anterior Eye.* 2010;33:55-60.
- 16. Aron EN, Aron A. Sensory-processing sensitivity and its relation to introversion and emotionality. *Journal of Personality and Social Psychology*, 1997;73:345-368.

17.

# APPENDIX A: PATIENT REPORTED OUTCOMES (STUDY QUESTIONNAIRES)
























## APPENDIX B: PATIENT INSTRUCTION GUIDE





ACUVUE OASYS® Brand Contact Lenses 1-Day with HydraLuxe™ Technology

ACUVUE OASYS<sup>®</sup> Brand Contact Lenses 1-Day with HydraLuxe™ Technology for Astigmatism

senofilcon A Soft (hydrophilic) Contact Lenses Visibility Tinted with UV Blocker for Daily Disposable Wear

# PATIENT INSTRUCTION GUIDE



CAUTION: U.S. Federal law restricts this device to sale by or on the order of a licensed practitioner.

# TABLE OF CONTENTS

| INTRODUCTION | 3 |
|------------------------------------------------------|----|
| SYMBOLS KEY | 4 |
| GLOSSARY OF COMMONLY USED TERMS | 5 |
| WEARING RESTRICTIONS & INDICATIONS | 5 |
| WHEN LENSES SHOULD NOT BE WORN (CONTRAINDICATIONS) | 6 |
| WARNINGS | 7 |
| PRECAUTIONS | 8 |
| ADVERSE REACTIONS (POSSIBLE PROBLEMS AND WHAT TO DO) | 9 |
| LENS HANDLING AND INSERTION | 10 |
| Step 1: Getting Started | 10 |
| Step 2: Opening the Packaging | 10 |
| Step 3: Placing the Lens on the Eye | 11 |
| Step 4: Checking Your Lenses | 12 |
| Step 5: Centering the Lens | 13 |
| LENS WEARING | 14 |
| REMOVING YOUR LENSES | 15 |
| EMERGENCIES | 16 |
| INSTRUCTIONS FOR THE PRESBYOPIC PATIENT (MONOVISION) | 16 |
| WEARING AND APPOINTMENT SCHEDULE | 18 |
| PATIENT / EYE CARE PROFESSIONAL INFORMATION | 19 |
| NOTES | 20 |

#### INTRODUCTION

#### About This Booklet:

The information and instructions contained in this booklet apply to the following brands:

- ACUVUE OASYS<sup>®</sup> Brand Contact Lenses 1-Day with HydraLuxe<sup>™</sup> Technology
- ACUVUE OASYS<sup>®</sup> Brand Contact Lenses 1-Day with HydraLuxe™ Technology for Astigmatism

For your eye health, it is important that your contact lenses be worn only as prescribed by your Eye Care Professional. Your Eye Care Professional should be kept fully aware of your medical history and will develop a total program of care based on your specific needs. He or she will review with you all instructions for lens handling and care, including how to safely and easily open the packaging. You will also be taught how to properly apply and remove lenses. This booklet will reinforce those instructions.

#### If you have any questions, always ask your Eye Care Professional.

A "Glossary of Commonly Used Terms" is included for your reference. This contains definitions of medical and technical terminology used in this booklet. In addition, a "Symbols Key" provides an explanation of symbols that may appear on the lens packaging.

Special sections are included in the back of this booklet to record your specific prescribed wearing information as well as to record the contact information for your Eye Care Professional.

#### About Your Lenses and Contact Lens Wear:

Your contact lenses are made from a water loving (hydrophilic) material that has the ability to absorb water, making the lenses soft and flexible. The lenses are tinted to improve visibility for handling and also contain an ultraviolet (UV) radiation absorbing ingredient to block UV radiation.

These lenses are intended for the correction of nearsightedness (myopia) and farsightedness (hyperopia). They are also available for people who may have other conditions, such as astigmatism.

When prescribed for daily disposable wear, lenses should be discarded upon removal; therefore, no cleaning or disinfection is required. You should always have spare lenses or glasses available.

By replacing your contact lenses on a regular basis, lens deposits, which can affect vision and cause irritation and discomfort to the eye, have little chance to build up over time as with conventional lens wear. When you discard the lens, you dispose of potential deposit build-up problems.

# SYMBOLS KEY

# The following symbols may appear on the label or carton:

| Symbol | Definition |
|---|---|
| Ţ <u>i</u> | Consult Instructions for Use |
| <b>W</b> | Manufactured by or in |
| سا | Date of Manufacture |
| $\mathbf{Z}$ | Use By Date (expiration date) |
| LOT | Batch Code |
| STERILE | Sterile Using Steam or Dry Heat |
| 2 | Single Use |
| DIA | Diameter |
| ВС | Base Curve |
| D | Diopter (lens power) |
| CYL | Cylinder |
| AXIS | Axis |
| <b>C€</b><br>0086 | Quality System Certification Symbol |
| W<br>UV Blocking | UV Blocking |
| 0 | Fee Paid for Waste Management |
| <b>R</b> Only | CAUTION: U.S. Federal law restricts this device to sale by or on the order of a licensed practitioner |
| <b>□ ♥</b> | Lens Orientation Correct |
| ¥ × | Lens Orientation Incorrect (Lens Inside Out) |

#### **GLOSSARY OF COMMONLY USED TERMS**

| Term | <b>Definition</b> |
|---|---|
| Astigmatism | A condition where the cornea is not equally curved in all parts of its surface. It is somewhat oval in shape, causing the visual image to be out of focus (blurred). |
| Conjunctivitis | Inflammation of the conjunctiva |
| Cornea | Clear front part of the eye |
| Corneal Ulcer | A sore or lesion on the cornea |
| Inflammation | Swelling, redness, and pain |

# **WEARING RESTRICTIONS & INDICATIONS**

The ACUVUE OASYS<sup>®</sup> Brand Contact Lenses 1-Day with HydraLuxe™ Technology are indicated for daily disposable wear for the correction of nearsightedness (myopia) and farsightedness (hyperopia) in people with non-diseased eyes who may have 1.00D or less of astigmatism.

The ACUVUE OASYS<sup>®</sup> Brand Contact Lenses 1-Day with HydraLuxe™ Technology for Astigmatism are indicated for daily disposable wear for the correction of nearsightedness (myopia) and farsightedness (hyperopia) in people with non-diseased eyes who may have 0.50D to 3.00D of astigmatism.

These lenses contain a UV Blocker to help protect against transmission of harmful UV radiation to the cornea and into the eye.

WARNING: UV ABSORBING CONTACT LENSES are NOT substitutes for protective UV absorbing eyewear such as UV absorbing goggles or sunglasses because they do not completely cover the eye and surrounding area. You should continue to use UV absorbing eyewear as directed.

NOTE: Long-term exposure to UV radiation is one of the risk factors associated with cataracts. Exposure is based on a number of factors such as environmental conditions (altitude, geography, cloud cover) and personal factors (extent and nature of outdoor activities). UV Blocking contact lenses help provide protection against harmful UV radiation. However, clinical studies have not been done to demonstrate that wearing UV Blocking contact lenses reduces the risk of developing cataracts or other eye disorders. Consult your Eye Care Professional for more information.

Your Eye Care Professional will determine your wearing schedule (how long you should wear your lenses each day). When prescribed for daily disposable wear, lenses should be discarded upon removal.

# WHEN LENSES SHOULD NOT BE WORN (CONTRAINDICATIONS)

There are certain health conditions with which contact lenses should not be worn. You should alert your Eye Care Professional to any of the conditions listed below. Only your Eye Care Professional can determine if contact lens wear is right for you.

- Inflammation or infection in or around the eye or eyelids
- Any eye disease, injury, or abnormality that affects the cornea, conjunctiva, or eyelids
- Any previously diagnosed condition that makes contact lens wear uncomfortable
- Severe dry eye
- Reduced corneal sensitivity
- Any systemic disease that may affect the eye or may be made worse by wearing contact lenses
- Allergic reactions on the surface of the eye or surrounding tissues that may be induced or made worse by wearing contact lenses
- Irritation of the eye caused by allergic reactions to ingredients in contact lens solutions (i.e., rewetting drops). These solutions may contain chemicals or preservatives (such as mercury, Thimerosal, etc.) to which some people may develop an allergic response
- Any active eye infection
- If eyes become red or irritated



### WARNINGS

#### What You Should Know About Contact Lens Wear:

# EYE PROBLEMS, INCLUDING CORNEAL ULCERS, CAN DEVELOP RAPIDLY AND LEAD TO LOSS OF VISION. IF YOU EXPERIENCE:

- Eye Discomfort,
- Excessive Tearing,
- Vision Changes,
- Loss of Vision,
- Eye Redness, or
- Other Eye Problems,

# YOU SHOULD IMMEDIATELY REMOVE THE LENSES, AND PROMPTLY CONTACT YOUR EYE CARE PROFESSIONAL.

- When prescribed by your Eye Care Professional for daily disposable wear (i.e., your Eye Care Professional instructs you to remove and discard your lenses at the end of each day), you should not wear your lenses while sleeping. Clinical studies have shown that the risk of serious eye problems is increased when lenses are worn overnight.<sup>1</sup>
- Studies have shown that contact lens wearers who smoke have a higher rate of eye problems than nonsmokers.
- Problems with contact lenses or lens care products could result in serious injury to the eye.
- Proper use and care of your contact lenses and lens care products are essential for the safe use of these products.
- The overall risk of serious eye problems may be reduced by carefully following directions for lens care.

# Specific Instructions for Use and Warnings:

#### Water Activity

#### Instruction for Use

Do not expose your contact lenses to water while you are wearing them.

#### **WARNING:**

Water can harbor microorganisms that can lead to severe infection, vision loss, or blindness. If your lenses have been submersed in water when participating in water sports or swimming in pools, hot tubs, lakes, or oceans, you should discard them and replace them with a new pair. Ask your Eye Care Professional for recommendations about wearing your lenses during any activity involving water.

<sup>&</sup>lt;sup>1</sup>New England Journal of Medicine, September 21, 1989; 321 (12), pp. 773-783

# **PRECAUTIONS**

For your eye health, it is important to carefully follow the handling, insertion, removal, and wearing instructions in this booklet, as well as those prescribed by your Eye Care Professional (see "Lens Handling & Insertion" and "Lens Wearing" sections).

#### General Precautions:

- If you wear your contact lenses to correct presbyopia using monovision, you
  may not be able to get the best corrected visual acuity for either far or near
  vision. Visual needs are different for different people, so your Eye Care
  Professional should work with you when selecting the most appropriate type of
  lens for you.
- Always contact your Eye Care Professional before using any medicine in your eyes.
- Be aware that certain medications, such as antihistamines, decongestants, diuretics, muscle relaxants, tranquilizers, and those for motion sickness may cause dryness of the eye, increased lens awareness (feeling of the lens in the eye), or blurred vision. Always inform your Eye Care Professional if you experience any problems with your lenses while taking such medications. Depending on your symptoms, your Eye Care Professional may recommend rewetting drops that are available for use with soft contact lenses or may recommend that you stop wearing contact lenses while you are using these medications.
- Be aware that if you use oral contraceptives (birth control pills), you could develop changes in vision or comfort when wearing contact lenses.
- As with any contact lens, follow-up visits are necessary to assure the continuing health of your eyes. Ask your Eye Care Professional about the recommended follow-up schedule.

# Who Should Know That You are Wearing Contact Lenses:

- Inform all of your doctors (Health Care Professionals) about being a contact lens wearer.
- Always inform your employer of being a contact lens wearer. Some jobs may require use of eye protection equipment or may require that you not wear contact lenses.



# ADVERSE REACTIONS (POSSIBLE PROBLEMS AND WHAT TO DO)

#### Possible Problems

Be aware that problems can occur while wearing contact lenses and may or may not be associated with the following symptoms:

- Burning, stinging, and/or itchy eyes
- Reduced lens comfort
- Feeling of something in your eye (foreign body, scratched area)
- Swelling or inflammation in or around the eyes
- Eye redness
- Eyelid problems
- Watery eyes
- Unusual eye secretions
- Poor vision
- Blurred vision
- Rainbows or halos around objects
- Sensitivity to light (photophobia)
- Dry eyes

When any of the above symptoms occur, a serious eye condition may be present. You should **immediately be seen by your Eye Care Professional** so that the problem can be identified and treated, if necessary, in order to avoid serious eye damage.

# Recognizing Problems and What To Do

You should conduct a simple 3-part self-examination at least once a day. Ask yourself:

- How do the lenses feel on my eyes?
- How do my eyes look?
- Have I noticed a change in my vision?

If you notice any problems, you should IMMEDIATELY REMOVE YOUR LENS. If the problem or discomfort stops, discard the lens and place a new fresh lens on the eye.

If after inserting the new lens, the problem continues, IMMEDIATELY REMOVE THE LENS AND CONTACT YOUR EYE CARE PROFESSIONAL.

Do NOT use a new lens as self-treatment for the problem.

### LENS HANDLING AND INSERTION

For your eye health, it is important to carefully follow the handling, insertion, removal, and wearing instructions in this booklet, as well as those prescribed by your Eye Care Professional. If you will not or cannot always follow the recommended care procedures, you should not attempt to wear contact lenses.

When you first get your lenses, be sure that you are able to put the lenses on and remove them (or have someone else available who can remove the lenses for you) before leaving your Eye Care Professional's office.

#### Step 1: Getting Started

It is essential that you learn and use good hygiene in the care and handling of your new lenses.

Cleanliness is the first and most important aspect of proper contact lens care. In particular, your hands should be clean, dry, and free of any soaps, lotions, or creams before you handle your lenses.

#### Before you start:

- Always wash your hands thoroughly with a mild soap, rinse completely, and dry with a lint-free towel before touching your lenses.
  - DO NOT touch your contact lenses with your fingers or hands if they are not completely clean, because tiny lens scratches may occur, causing unclear vision and/or injury to your eye.
- You should avoid the use of soaps containing cold cream, lotion, or oily cosmetics before handling your lenses. These substances may come into contact with the lenses and interfere with successful wearing.
  - DO NOT get cosmetics, lotions, soaps, creams, deodorants, or sprays in your eyes or on your lenses. It is best to put on your lenses before putting on makeup. Water-based cosmetics are less likely to damage lenses than oil-based products.

Start off correctly by getting into the habit of always using proper hygiene so that they become automatic.

# Step 2: Opening the Packaging

#### Multi-Pack

Each multi-pack contains individually packaged lenses. Each lens comes in its own lens package designed specifically to keep it sterile. You may choose to keep your lenses inside the multi-pack for storage until you are ready to use them.

#### Lens Package

To open an individual lens package, follow these simple steps:

#### DO NOT use if the sterile blister package is opened or damaged.

- 1. Shake the lens package and check to see that the lens is floating in the solution.
- 2. Peel back the foil closure to reveal the lens. By stabilizing the lens package on the table-top, you will minimize the possibility of a sudden splash.
- 3. Place a finger on the lens and slide the lens up the side of the bowl of the lens package until it is free of the container.

NEVER use tweezers or other tools to remove your lenses from the lens container unless specifically indicated for that use.

Occasionally, a lens may stick to the inside surface of the foil when opened, or to the plastic package itself. This will not affect the sterility of the lens. It is still perfectly safe to use. Carefully remove and inspect the lens following the handling instructions.

#### **Lens Handling Tips**

• Handle your lenses with your fingertips, and be careful to avoid contact with fingernails. It is helpful to keep your fingernails short and smooth.

DO NOT touch the lens with your fingernails.

- Develop the habit of always working with the same lens first to avoid mix-ups.
- After you have removed the lens from the packaging, examine it to be sure that
  it is moist, clean, and free of any nicks or tears. If the lens appears damaged,
  DO NOT use it. Use the next lens in the multi-pack.

ALWAYS handle lenses carefully and avoid dropping them.

# Step 3: Placing the Lens on the Eye

Remember, always start with the same eye.

Once you have opened the lens package, removed, and examined the lens, follow these steps to insert the lens onto your eye:

- 1. BE SURE THE LENS IS NOT INSIDE-OUT by following either of the following procedures:
  - Place the lens on the tip of your index finger and check its profile. The lens should assume a natural, curved, bowl-like shape. If the lens edges tend to point outward, the lens is inside out. Another method is to gently squeeze the lens between the thumb and forefinger. The edges should turn inward. If the lens is inside out, the edges will turn slightly outward.

**OR** 

- Place the lens on the tip of your index finger and, looking up at the lens, locate the numbers 1-2-3. 1-2-3 indicates correct orientation while a reverse of 1-2-3 indicates the lens is inside out. If the lens is inside out (reverse 1-2-3), invert the lens and locate the numbers again to confirm correct lens orientation. Note that the 1-2-3 marking is not present on ACUVUE OASYS® Brand Contact Lenses 1-Day for Astigmatism.
- 2. With the lens on your index finger, use your other hand to hold your upper eyelid so you won't blink.
- 3. Pull down your lower eyelid with the other fingers of your "inserting" hand.
- 4. Look up at the ceiling and gently place the lens on the lower part of your eye.
- 5. Slowly release your eyelid and close your eye for a moment.
- 6. Blink several times to center the lens.
- 7. Use the same technique when inserting the lens for your other eye.

There are other methods of lens placement. If the above method is difficult for you, ask your Eye Care Professional for an alternate method.

### Step 4: Checking Your Lenses

After you have successfully inserted your lenses, you should ask yourself:

- Do I see well?
- How do the lenses feel on my eyes?
- How do my eyes look?

If after placement of the lens, your vision is blurred, check for the following:

- The lens is not centered on the eye (see "Step 5: Centering the Lens", next in this booklet).
- If the lens is centered, remove the lens (see "Removing Your Lenses") and check for the following:
  - Cosmetics or oils on the lens. Dispose of the lens and insert a new fresh lens.
  - The lens is on the wrong eye.
  - The lens is inside out (it would also not be as comfortable as normal). See
     "Step 3: Placing the Lens on the Eye".

If you find that your vision is still blurred after checking the above possibilities, remove both lenses and consult your Eye Care Professional.

**Note:** If a lens is noticeably uncomfortable upon insertion or becomes less comfortable than when it was first inserted, remove the lens immediately and contact your Eye Care Professional. If your examination of your eyes and the lenses shows any other problems,



# IMMEDIATELY REMOVE YOUR LENSES AND CONTACT YOUR EYE CARE PROFESSIONAL

#### Step 5: Centering the Lens

A lens, which is on the cornea (center of your eye), will very rarely move onto the white part of the eye during wear. However, this can occur if insertion and removal procedures are not performed properly. To center a lens, follow either of these procedures:

• Close your eyelids and gently massage the lens into place through the closed lids.

#### **OR**

• Gently move the off-centered lens onto the cornea (center of your eye) while the eye is opened using finger pressure on the edge of the upper lid or lower lid.

# **LENS WEARING**

#### While wearing your lenses, remember the following important precautions:

#### Hazardous Conditions

- If you use aerosol (spray) products, such as hair spray, while wearing lenses, keep your eyes closed until the spray has settled.
- Avoid all harmful or irritating vapors and fumes while wearing lenses.

#### Water Activity

• Do not expose your contact lenses to water while you are wearing them.

#### Lubricating/Rewetting Solutions

- Your Eye Care Professional may recommend a lubricating/rewetting solution for your use. These solutions can be used to wet (lubricate) your lenses while you are wearing them.
- **Do not** use saliva or anything other than the recommended solutions for lubricating or rewetting your lenses. Do not put lenses in your mouth.
- Never rinse your lenses in water from the tap. There are two reasons for this:
  - 1. Tap water contains many impurities that can contaminate or damage your lenses and may lead to eye infection or injury.
  - 2. You might lose your lens down the drain.

# Sticking (Non-Moving) Lens

- For your eye health, it is important the lens moves freely on your eye.
- If the lens sticks (stops moving) on your eye, apply a few drops of the recommended rewetting solution. Wait until the lens begins to move freely on the eye before removing it. If non-movement of the lens continues, you should immediately consult your Eye Care Professional.

# Sharing Lenses

Never allow anyone else to wear your lenses. They have been prescribed to fit
your eyes and to correct your vision to the degree necessary. Sharing lenses
greatly increases the chance of eye infections.

# Adhering to the Prescribed Wearing & Replacement Schedules

- Never wear your lenses beyond the amount of time recommended by your Eye Care Professional.
- Always throw away worn lenses as prescribed by your Eye Care Professional.

## **REMOVING YOUR LENSES**

**CAUTION:** Always be sure the lens is on the cornea (center of your eye) before attempting to remove it. Determine this by covering the other eye. If vision is blurred, the lens is either on the white part of the eye or it is not on the eye at all. To locate the lens, inspect the upper area of the eye by looking down into a mirror while pulling the upper lid up. Then inspect the lower area by pulling the lower lid down.

#### Always remove the same lens first.

- 1. Wash, rinse, and dry your hands thoroughly.
- 2. There are two recommended methods of lens removal: the Pinch Method, and the Forefinger and Thumb Method. You should follow the method that is recommended by your Eye Care Professional.

#### Pinch Method:

- **Step 1.** Look up, slide the lens to the lower part of the eye using the forefinger.
- **Step 2.** Gently pinch the lens between the thumb and forefinger.
- Step 3. Remove the lens.

#### Forefinger and Thumb Method:

- **Step 1.** Place your hand or a towel under your eye to catch the lens.
- **Step 2.** Place your forefinger on the center of the upper lid and your thumb on the center of the lower lid.
- **Step 3.** Press in and force a blink. The lens should fall onto your hand or the towel.

**Note:** The lens may come out, but remain on the eyelid, finger, or thumb.

3. Remove the other lens by following the same procedure.

Remember, there is no cleaning or disinfection needed with your contact lenses when they are prescribed for daily disposable wear. Always dispose of lenses when they are removed and have replacement lenses or glasses available.

**Note:** If these methods of removing your lenses are difficult for you, ask your Eye Care Professional for an alternate method.

#### **EMERGENCIES**

If chemicals of any kind (household products, gardening solutions, laboratory chemicals, etc.) are splashed into your eyes: FLUSH EYES IMMEDIATELY WITH TAP WATER AND IMMEDIATELY CONTACT YOUR EYE CARE PROFESSIONAL OR VISIT A HOSPITAL EMERGENCY ROOM RIGHT AWAY.

# INSTRUCTIONS FOR THE PRESBYOPIC PATIENT (MONOVISION)

### About Presbyopia and Monovision Correction

- Presbyopia is a condition in which the natural lenses in the eyes lose some of their elasticity. This occurs normally with aging as the lenses lose some of their ability to change focus for different distances (loss of reading vision).
- Monovision is a method of correction for presbyopia using contact lenses in which one eye is corrected for distance vision and the other is corrected for near vision.

# Getting Used to Monovision Correction (Adaptation)

- Be aware that, as with any type of lens correction, there are advantages and compromises to monovision contact lens correction. The benefit of clear near vision when looking straight-ahead and upward that you get with your contact lenses for monovision may be accompanied by a vision compromise that may reduce the sharpness of your vision and depth perception for distance and near tasks. Some people have experienced difficulty adapting to this. You may experience symptoms, such as mild blurred vision and variable vision during this adaptation period. These symptoms may last for a brief period or for several weeks as you are getting used to the lenses. The longer these symptoms last, the poorer your chances may be for successful adaptation.
- You should avoid visually demanding situations during the initial adaptation period. It is recommended that you first wear these contact lenses in familiar situations that are not visually demanding. For example, it might be better to be a passenger rather than a driver of a car during the first days of lens wear. Also, it is recommended that you only drive with monovision correction if you pass your state driver's license requirements with monovision correction.
- It is important that you follow your Eye Care Professional's suggestions for getting
  used to monovision contact lens correction. You should discuss any concerns that
  you may have during and after the adaptation period.

#### Additional Correction Needs

- Some patients with monovision correction will need to wear their glasses over their contact lenses to provide the clearest vision for critical tasks. You should discuss this with your Eye Care Professional.
- Some patients will never be fully comfortable functioning under low levels of lighting, such as driving at night. If this happens, you may want to discuss with your Eye Care Professional having additional contact lenses prescribed so that both eyes are

16

- corrected for distance when sharp distance binocular vision is required from both eyes together.
- If you require very sharp near vision during prolonged close work, you may want to have additional contact lenses prescribed so that both eyes are corrected for near when sharp near vision is required from both eyes together.

The decision to be fit with monovision correction is most appropriately left to your Eye Care Professional, in conjunction with you, after carefully considering and discussing your needs.

17

# WEARING AND APPOINTMENT SCHEDULE

# **Prescribed Wearing Schedule**

| Day V | Vearing Time (Hours) |
|---------------|-------------------------------------------------------------|
| 1 | |
| 2 | |
| 3 | |
| 4 | |
| 5 | |
| 6 | |
| 7 | |
| 8 | |
| 9 | |
| 10 | |
| 11 | |
| 12 | |
| 13 | |
| 14 | |
| Appoin | tment Schedule |
| Your ap | pointments are on: |
| Minimu | m number of hours lenses to be worn at time of appointment: |
| Month: | Year: |
| <del></del> - | _ |
| Time: | Day: |



# PATIENT / EYE CARE PROFESSIONAL INFORMATION

| Next Appo | intment: | | | | |
|---|---|---|---|---|---|
| Date: | | | | | |
| Doctor: | | | | | |
| Address: | | | | | |
| Phone: | | | | | |
| | | | | , | · |
| Day | Date | Hours Worn | Day | Date | Hours Worn |
| 1 | | | 8 | | |
| 2 | | | 9 | | |
| 3 | | | 10 | | |
| 4 | | | 11 | | |
| 5 | ************************************** | | 12 | | |
| 6 | | | 13 | · | ···· |
| 7 | | | 14 | | |

IMPORTANT: If you experience any difficulty wearing your lenses or you do not understand the instructions given you, DO NOT WAIT for your next appointment.

CONTACT YOUR EYE CARE PROFESSIONAL IMMEDIATELY.

19

| NOTES |
|-------|
| • |



Johnson & Johnson Vision Care, Inc. 7500 Centurion Parkway Jacksonville, FL 32256 USA Tel: 1-800-843-2020

www.acuvue.com

©Johnson & Johnson Vision Care Companies 2016
In Canada: Johnson & Johnson Vision Care, division of Johnson & Johnson, Inc.
In USA: Johnson & Johnson Vision Care, Inc.

Revision date: 03/16

Revision number: AO-03-16-12

ACUVUE OASYS® and HydraLuxe™ are Trademarks of the Johnson & Johnson Vision Care Companies

# APPENDIX C: PACKAGE INSERT (APPROVED PRODUCT)



IMPORTANT: Please read carefully and keep this information for future use.

This Package Insert and Fitting Guide is intended for the Eye Care Professional, but should be made available to patients upon request.

The Eye Care Professional should provide the patient with the appropriate instructions that pertain to the patient's prescribed lenses. Copies are available for download at www.acuvue.com.



ACUVUE OASYS® Brand Contact Lenses 1-Day with HydraLuxe™ Technology

**ACUVUE OASYS® Brand Contact Lenses 1-Day** with HydraLuxe™ Technology for ASTIGMATISM

senofilcon A Soft (hydrophilic) Contact Lenses Visibility Tinted with UV Blocker for Daily Disposable Wear



CAUTION: U.S. Federal law restricts this device to sale by or on the order of a licensed practitioner.

JJV/R-GOTTHEFF.NGIAL


# SYMBOLS KEY

The following symbols may appear on the label or carton:

| SYMBOL | DEFINITION |
|---|---|
| (i | Consult Instructions for Use |
| اس | Manufactured by or in |
| س | Date of Manufacture |
| $\mathbf{\Sigma}_{\mathbf{I}}$ | Use By Date (expiration date) |
| LOT | Batch Code |
| STERILE | Sterile Using Steam or Dry Heat |
| 2 | Single-Use |
| DIA | Diameter |
| BC | Base Curve |
| D | Diopter (lens power) |
| CYL | Cylinder |
| AXIS | Axis |
| <b>C€</b><br>0086 | Quality System Certification Symbol |
| W<br>UV Blocking | UV-Blocking |
| 0 | Fee Paid for Waste Management |
| <b>R</b> Only | CAUTION: U.S. Federal law restricts this device to sale by or on the order of a licensed practitioner |
| <b>□ ♥</b> | Lens Orientation Correct |
| W X | Lens Orientation Incorrect (Lens Inside Out) |

## **DESCRIPTION**

ACUVUE OASYS® Brand Contact Lenses 1-Day and ACUVUE OASYS® Brand Contact Lenses 1-Day for ASTIGMATISM are soft (hydrophilic) contact lenses made with HydraLuxe™ Technology. They are available as spherical or toric lenses respectively.

These lenses are made of a silicone hydrogel material containing an internal wetting agent, visibility tint, and UV absorbing monomer and are tinted blue using Reactive Blue Dye #4 to make the lenses more visible for handling.

A benzotriazole UV absorbing monomer is used to block UV radiation. The transmittance characteristics for these lenses are less than 1% in the UVB range of 280 nm to 315 nm and less than 10% in the UVA range of 316 nm to 380 nm for the entire power range.

#### **Lens Properties:**

#### The physical/optical properties of the lens are:

Specific Gravity (calculated): 0.98 - 1.12

1.42 Refractive Index:

85% minimum Light Transmission:

Surface Character: Hydrophilic

Water Content: 38%

Oxygen Permeability:

#### **VALUE METHOD**

122 x 10<sup>-11</sup> (cm<sup>2</sup>/sec) Fatt (boundary corrected, non-(ml O<sub>2</sub>/ml x mm Hg) at 35°C edge corrected) 103 x 10<sup>-11</sup> (cm<sup>2</sup>/sec) Fatt (boundary corrected, edge (ml O<sub>2</sub>/ml x mm Hg) at 35°C corrected)

#### **Lens Parameters:**

12.0 mm to 15.0 mm Diameter Range:

Center Thickness: varies with power

7.85 mm to 10.00 mm Base Curve Range:

Spherical Power Range: -20.00D to +20.00D

-0.25D to -10.00D Cylinder Power Range:

Axis Range: CR-5969 v3 0

5° to 180° JJVC CONFIDENTIAL


# **AVAILABLE LENS PARAMETERS**

ACUVUE OASYS® Brand 1-Day with HydraLuxe™ Technology are hemispherical shells of the following dimensions:

**Diameter:** 14.3 mm

**Center Thickness:** 0.085 mm to 0.221 mm (varies with power)

Base Curve: 8.5 mm, 9.0 mm

**Powers:** -0.50D to -6.00D (in 0.25D increments)

-6.50D to -12.00D (in 0.50D increments) +0.50D to +6.00D (in 0.25D increments) +6.50D to +8.00D (in 0.50D increments)

ACUVUE OASYS® Brand 1-Day with HydraLuxe™ Technology for ASTIGMATISM are hemitoric shells of the following dimensions:

**Diameter:** 14.3 mm

**Center Thickness:** 0.075 mm to 0.172 mm (varies with power)

**Base Curve:** 8.5 mm

**Powers:** +0.00D to -6.00D (in 0.25D increments)

Cylinders: -0.75D, -1.25D, -1.75D, -2.25D\*

Axis: 10° to 180° in 10° increments

\*-2.25D cylinder is availble in 10°, 20°, 70°, 80°, 90°, 100°, 110°,

160°, 170°, 180° axes only.

+0.25D to +4.00D (in 0.25D increments)

-6.50D to -9.00D (in 0.50D increments)

Cylinders: -0.75D, -1.25D, -1.75D

Axis: 10°, 20°, 70°, 80°, 90°, 100°, 110°, 160°,

170°, 180°

# TRANSMITTANCE CURVES

ACUVUE OASYS® 1-Day with HydraLuxe™ Technology (senofilcon A) Visibility Tinted with UV Blocker vs. 24 yr. old human cornea and 25 yr. old human crystalline lens.



<sup>\*</sup> The data was obtained from measurements taken through the central 3-5 mm portion for the thinnest marketed lens (-9.00D lens, 0.075 mm center thickness).

<sup>1</sup>Lerman, S., Radiant Energy and the Eye, MacMillan, New York, 1980, p. 58, figure 2-21

<sup>2</sup>Waxler, M., Hitchins, V.M., Optical Radiation and Visual Health, CRC Press, Boca Raton, Florida, 1986, p. 19, figure 5

WARNING: UV absorbing contact lenses are NOT substitutes for protective UV absorbing eyewear, such as UV absorbing goggles or sunglasses because they do not completely cover the eye and surrounding area. The patient should continue to use UV absorbing eyewear as directed.

### **ACTIONS**

In its hydrated state, the contact lens, when placed on the cornea, acts as a refracting medium to focus light rays onto the retina.

The transmittance characteristics for these lenses are less than 1% in the UVB range of 280 nm to 315 nm and less than 10% in the UVA range of 316 nm to 35,000 for the ge. JJVC CONFIDENTIAL

NOTE: Long-term exposure to UV radiation is one of the risk factors associated with cataracts. Exposure is based on a number of factors such as environmental conditions (altitude, geography, cloud cover) and personal factors (extent and nature of outdoor activities). UV-Blocking contact lenses help provide protection against harmful UV radiation. However, clinical studies have not been done to demonstrate that wearing UV-Blocking contact lenses reduces the risk of developing cataracts or other eye disorders. The Eye Care Professional should be consulted for more information.

# **INDICATIONS (USES)**

ACUVUE OASYS® Brand Contact Lenses 1-Day with HydraLuxe™ Technology are indicated for daily disposable wear for the optical correction of refractive ametropia (myopia and hyperopia) in phakic or aphakic persons with non-diseased eyes who may have 1.00D or less of astigmatism.

ACUVUE OASYS® Brand Contact Lenses 1-Day with HydraLuxe™ Technology for ASTIGMATISM are indicated for daily disposable wear for the optical correction of refractive ametropia (myopia and hyperopia) in phakic or aphakic persons with non-diseased eyes who may have 0.50D to 3.00D of astigmatism.

These lenses contain a UV Blocker to help protect against transmission of harmful UV radiation to the cornea and into the eye.

# **CONTRAINDICATIONS (REASONS NOT TO USE)**

# DO NOT USE these contact lenses when any of the following conditions exist:

- Acute or subacute inflammation or infection of the anterior chamber of the eye.
- Any eye disease, injury or abnormality that affects the cornea, conjunctiva, or eyelids.
- Severe insufficiency of lacrimal secretion (dry eye).


- Corneal hypoesthesia (reduced corneal sensitivity).
- Any systemic disease that may affect the eye or be exaggerated by wearing contact lenses.
- Allergic reactions of ocular surfaces or adnexa that may be induced or exaggerated by wearing contact lenses or use of contact lens solutions.
- Ocular irritation due to allergic reactions which may be caused by use of contact lens solutions (i.e., rewetting drops) that contain chemicals or preservatives (such as mercury, Thimerosal, etc.) to which some people may develop an allergic response.
- Any active corneal infection (bacterial, fungal, protozoal, or viral).
- If eyes become red or irritated.

### **WARNINGS**

Patients should be advised of the following warnings pertaining to contact lens wear:

EYE PROBLEMS, INCLUDING CORNEAL ULCERS, CAN DEVELOP RAPIDLY AND LEAD TO LOSS OF VISION; IF THE PATIENT EXPERIENCES:

- Eye Discomfort,
- Excessive Tearing,
- Vision Changes,
- Loss of Vision.
- Eye Redness,
- Or Other Eye Problems,

THE PATIENT SHOULD BE INSTRUCTED TO IMMEDIATELY REMOVE THE LENSES AND PROMPTLY CONTACT THE EYE CARE PROFESSIONAL.

 When prescribed for daily wear, patients should be instructed not to wear lenses while sleeping. Clinical studies have shown that the risk of serious adverse reactions is increased when lenses are worn swerpight, and that pulcerative were its is greater for


- extended wear contact lens users than for daily wear users.3
- Studies have shown that contact lens wearers who are smokers have a higher incidence of adverse reactions than nonsmokers.
- Problems with contact lenses or lens care products could result in serious injury to the eye. Patients should be cautioned that proper use and care of contact lenses and lens care products are essential for the safe use of these products.
- The overall risk of ulcerative keratitis may be reduced by carefully following directions for lens care.

#### **Specific Instructions for Use and Warnings:**

Water Activity

#### Instructions for Use

Do not expose contact lenses to water while wearing them.

#### **WARNING:**

Water can harbor microorganisms that can lead to severe infection, vision loss or blindness. If lenses have been submersed in water when participating in water sports or swimming in pools, hot tubs, lakes, or oceans, the patient should be instructed to discard them and replace them with a new pair. The Eye Care Professional should be consulted for recommendations regarding wearing lenses during any activity involving water.

# **PRECAUTIONS**

# **Special Precautions for Eye Care Professionals:**

Due to the small number of patients enrolled in clinical investigation of lenses, all refractive powers, design configurations, or lens parameters available in the lens material are not evaluated in significant numbers. Consequently, when selecting an appropriate lens design and parameters, the Eye Care Professional should consider all characteristics of the lens that can affect lens performance and ocular health, including oxygen permeability, wettability, central and peripheral thickness, and optic zone diameter.


<sup>&</sup>lt;sup>3</sup> New England Journal of Medicine, September 21, 1989; 321 (12), pp. 773-783

- The potential impact of these factors on the patient's ocular health should be carefully weighed against the patient's need for refractive correction; therefore, the continuing ocular health of the patient and lens performance on the eye should be carefully monitored by the prescribing Eye Care Professional.
- Patients who wear these lenses to correct presbyopia using monovision may not achieve the best corrected visual acuity for either far or near vision. Visual requirements vary with the individual and should be considered when selecting the most appropriate type of lens for each patient.
- Fluorescein, a yellow dye, should not be used while the lenses are on the eyes. The lenses absorb this dye and become discolored.
   Whenever fluorescein is used in eyes, the eyes should be flushed with a sterile saline solution that is recommended for in-eye use.
- Eye Care Professionals should instruct the patient to remove the lenses immediately if the eyes become red or irritated.

# Eye Care Professionals should carefully instruct patients about the following care regimen and safety precautions.

## **Handling Precautions:**

- Before leaving the Eye Care Professional's office, the patient should be able to promptly remove the lenses or should have someone else available who can remove the lenses for him or her.
- DO NOT use if the sterile blister package is opened or damaged.
- Always wash and rinse hands before handling lenses. Do not get cosmetics, lotions, soaps, creams, deodorants, or sprays in the eyes or on the lenses. It is best to put on lenses before putting on makeup. Water-based cosmetics are less likely to damage lenses than oil-based products.
- DO NOT touch contact lenses with the fingers or hands if the hands are not free of foreign materials, as microscopic scratches of the lenses may occur, causing distorted vision and/or injury to the eye.
- Carefully follow the handling, insertion, removal, and wearing instructions in the "Patien Guide" for the prescribed
   

wearing schedule and those prescribed by the Eye Care Professional.

- Always handle lenses carefully and avoid dropping them.
- Never use tweezers or other tools to remove lenses from the lens container unless specifically indicated for that use. Slide the lens up the side of the bowl until it is free of the container.
- Do not touch the lens with fingernails.

#### **Lens Wearing Precautions:**

- If the lens sticks (stops moving) on the eye, follow the recommended directions in "Care for a Sticking (Non-Moving) Lens." The lens should move freely on the eye for the continued health of the eye. If non-movement of the lens continues, the patient should be instructed to immediately consult his or her Eye Care Professional.
- Never wear lenses beyond the period recommended by the Eye Care Professional.
- The patient should be advised to never allow anyone else to wear their lenses. They have been prescribed to fit their eyes and to correct their vision to the degree necessary. Sharing lenses greatly increases the chance of eye infections.
- If aerosol products, such as hair spray, are used while wearing lenses, exercise caution and keep eyes closed until the spray has settled.
- Avoid all harmful or irritating vapors and fumes while wearing lenses.
- Always discard lenses worn as prescribed by the Eye Care Professional.

#### **Lens Care Precautions:**

 The patient should be informed that no cleaning or disinfection is needed when lenses are worn for daily disposable wear. Patients should always dispose of lenses when removed and have spare lenses or spectacles available.

CR-5969 v3 0



#### Other Topics to Discuss with Patients:

- Always contact the Eye Care Professional before using any medicine in the eyes.
- Certain medications, such as antihistamines, decongestants, diuretics, muscle relaxants, tranquilizers, and those for motion sickness may cause dryness of the eye, increased lens awareness, or blurred vision. Should such conditions exist, proper remedial measures should be prescribed. Depending on the severity, this could include the use of lubricating drops that are indicated for use with soft contact lenses or the temporary discontinuance of contact lens wear while such medication is being used.
- Oral contraceptive users could develop visual changes or changes in lens tolerance when using contact lenses. Patients should be cautioned accordingly.
- As with any contact lens, follow-up visits are necessary to assure the continuing health of the patient's eyes. The patient should be instructed as to a recommended follow-up schedule.

#### Who Should Know That the Patient is Wearing Contact Lenses?

- Patients should inform all doctors (Health Care Professionals) about being a contact lens wearer.
- Patients should always inform their employer of being a contact lens wearer. Some jobs may require use of eye protection equipment or may require that the patient not wear contact lenses.

# **ADVERSE REACTIONS**

# The patient should be informed that the following problems may occur when wearing contact lenses:

- The eye may burn, sting, and/or itch.
- There may be less comfort than when the lens was first placed on the eye.
- There may be a feeling of something in the eye (foreign body, scratched area).
- There snay to the 

peripheral infiltrates, peripheral corneal ulcers, or corneal erosion. There may be the potential for other physiological observations, such as local or generalized edema, corneal neovascularization, corneal staining, injection, tarsal abnormalities, iritis, and conjunctivitis; some of which are clinically acceptable in low amounts.

- There may be excessive watering, unusual eye secretions, or redness of the eye.
- Poor visual acuity, blurred vision, rainbows, or halos around objects, photophobia, or dry eyes may also occur if the lenses are worn continuously or for too long a time.

The patient should be instructed to conduct a simple 3-part self-examination at least once a day. They should ask themselves:

- How do the lenses feel on my eyes?
- How do my eyes look?
- Have I noticed a change in my vision?

If the patient reports any problems, he or she should be instructed to IMMEDIATELY REMOVE THE LENS. If the problem or discomfort stops, the patient should discard the lens and place a new fresh lens on the eye.

If after inserting the new lens, the problem continues, the patient should be directed to IMMEDIATELY REMOVE THE LENS AND CONTACT HIS OR HER EYE CARE PROFESSIONAL.

The patient should be instructed NOT to use a new lens as self-treatment for the problem.

The patient should be advised that when any of the above symptoms occur, a serious condition such as infection, corneal ulcer, neovascularization, or iritis may be present. He or she should be instructed to seek immediate professional identification of the problem and prompt treatment to avoid serious eye damage.



#### GENERAL FITTING GUIDELINES

#### A. Patient Selection

Patients selected to wear these lenses should be chosen based on:

- · Motivation to wear lenses
- · Ability to follow instructions regarding lens wear care
- · General health
- Ability to adequately handle and care for the lenses
- · Ability to understand the risk and benefits of lens wear

Patients who do not meet the above criteria should not be provided with contact lenses.

#### B. Pre-fitting Examination

Initial evaluation of the patient should begin with a thorough case history to determine if there are any contraindications to contact lens wear. During the case history, the patient's visual needs and expectations should be determined as well as an assessment of their overall ocular, physical, and mental health.

Preceding the initial selection of trial contact lenses, a comprehensive ocular evaluation should be performed that includes, but is not limited to, the measurement of distance and near visual acuity, distance and near refractive prescription (including determining the preferred reading distance for presbyopes), keratometry, and biomicroscopic evaluation.

Based on this evaluation, if it is determined that the patient is eligible to wear these lenses, the Eye Care Professional should proceed to the lens fitting instructions as outlined below.

#### C. Initial Power Determination

A spectacle refraction should be performed to establish the patient's baseline refractive status and to guide in the selection of the appropriate lens power. Remember to compensate for vertex distance if the refraction is greater than ±4.00D.

#### D. Base Curve Selection (Trial Lens Fitting)

The following trial lenses should be selected for patients regardless of keratometry readings. However, corneal curvature measurements should be performed to establish the patient's baseline ocular status.


- ACUVUE OASYS® 1-Day: 8.5 mm/14.3 mm
- ACUVUE OASYS® 1-Day for ASTIGMATISM: 8.5 mm/14.3 mm

The trial lens should be placed on each of the patient's eyes and evaluated after the patient has adjusted to the lenses.

# 1. Criteria of a Properly Fit Lens

A properly fit lens will center and completely cover the cornea (i.e., no limbal exposure), have sufficient movement to provide tear exchange under the contact lens with the blink, and be comfortable. The lens should move freely when manipulated digitally with the lower lid, and then return to its properly centered position when released.

# 2. Criteria of a Flat Fitting Lens

A flat fitting lens may exhibit one or more of the following characteristics: decentration, incomplete corneal coverage (i.e., limbal exposure), excessive movement with the blink, and/or edge standoff. If the lens is judged to be flat fitting, it should not be dispensed to the patient.

# 3. Criteria of a Steep Fitting Lens

A steep fitting lens may exhibit one or more of the following characteristics: insufficient movement with the blink, conjunctival indentation, and resistance when pushing the lens up digitally with the lower lid. If the lens is judged to be steep fitting, it should not be dispensed to the patient.

If the initial trial base curve is judged to be flat or steep fitting, the alternate base curve, if available, should be trial fit and evaluated after the patient has adjusted to the lens. The lens should move freely when manipulated digitally with the lower lid, and then return to a properly centered position when released. If resistance is encountered when pushing the lens up, the lens is fitting tightly and should not be dispensed to the patient.

# E. Final Lens Power (Spherical)

A spherical over-refraction should be performed to determine the final lens power after the lens fit is judged acceptable. The spherical over-refraction should be combined with the trial lens power to determine the final lens prescription. The patient should experience good visual acuity with the correct leas-prover unless there


| Example 1 | |
|----------------------------|--------|
| Diagnostic lens: | -2.00D |
| Spherical over-refraction: | -0.25D |
| Final lens power: | -2.25D |

| Example 2 | |
|----------------------------|--------|
| Diagnostic lens: | -2.00D |
| Spherical over-refraction: | +0.25D |
| Final lens power: | -1.75D |

If vision is acceptable, perform a slit lamp examination to assess adequate fit (centration and movement). If the fit is acceptable, dispense the lenses and instruct the patient to return in one week for reassessment (see dispensing and follow up information in **PATIENT MANAGEMENT**).

All patients should be supplied with a copy of the PATIENT INSTRUCTION GUIDE for these lenses. Copies are available for download at www.acuvue.com.

# TORIC FITTING GUIDELINES

Although most aspects of the fitting procedure are identical for all types of soft contact lenses, including toric lenses, there are some additional steps and/or rules to follow to assure the proper fit of toric lenses.

The only new steps you must follow in prescribing ACUVUE OASYS® 1-Day for ASTIGMATISM are that you must determine the stability, repeatability, and drift angle of the lens axis so that you can prescribe the correct lens axis for the patient.

# A. How to Determine Lens Cylinder and Axis Orientation

#### 1. Locate the Orientation Marks

To help determine the proper orientation of the toric lens, you'll find two primary marks approximately 1 mm from the lens edge representing the vertical position on opposite ends of the lens at 6 and 12 o'clock (Fig. 1). Because of the lens' ballasting system, either mark can represent the vertical position — there is no "top" and "bottom" as in a prism-ballasted lens. You don't need to view both marks to assess orientation; simply look for the 6 o'clock mark as you would with a prism-ballasted lens.


CR-5969 v3 0




You'll need a slit lamp biomicroscope with a 1 to 2 mm parallelepiped beam to highlight the marks when the lens is fitted to the eye. There are a number of techniques you can use to improve the visibility of the 6 o'clock mark. Using a parallelepiped beam and medium magnification (10x or 15x), slowly pan down the lens, looking just below the direct illumination at the retroilluminated area. Backlighting the mark this way should make it more visible. Sometimes manipulating the lower lid may be necessary to uncover the mark.

#### 2. Observe Lens Rotation and Stability

Observe the position and stability of the "bottom" mark. It usually stabilizes at the 6 o'clock position. If it does, calculation of the lens power will be straightforward. The 6 o'clock position is not a "must"; however, the absolute requirement is that the axis position be stable and repeatable.

The mark may stabilize somewhat left or right (drift) of the vertical meridian and still enable you to fit a toric lens for that eye, as long as the lens always returns to the same "drift axis" position after settling. The deviation can be compensated for in the final prescription. Your objective is to ensure that whatever position the initial lens assumes near 6 o'clock, this position must be stable and repeatable. With full eye movement or heavy blink, you may see the marks swing away, but they must return quickly to the original stable position. If the lens does not return quickly, you may need to select a different lens.

# 3. Assessing Rotation

Imagine the eye as a clock dial and every hour represents a 30° interval. If the orientation mark of the initial lens stabilizes somewhat left or right of the vertical position, the final lens will orient on the eye with the same deviation. You can use an axis reticule in the slit lamp or use a line-scribed lens in a spectacle trial frame to measure or estimate the "drift angle" of the cylinder axis.

To compensate for this "drift", measure or estimate the "drift", then add or subtract it from the refractive axis to determine the correct cylinder axis. Use the LARS (Left Add, Right Subtract) method to determine which direction to compensate.


#### **B. Final Lens Power**

When the diagnostic lens has its axis aligned in the same meridian as the patient's refractive axis, a spherocylindrical over-refraction may be performed and visual acuity determined. However, in the case of crossed axes, such as when the diagnostic lens axis is different from the spectacle cylinder axis, it is not advisable to perform a full spherocylindrical over-refraction because of the difficulty in computing the resultant power. A spherical over-refraction without cylinder refraction may be performed.

If the required cylinder correction falls between two available cylinder powers, it is recommended to prescribe the lower cylinder power lens. See below for instructions on how to determine the final lens power.

#### 1. For the Sphere

If sphere alone or combined sphere and cylinder Rx  $> \pm 4.00$ D, compensate for vertex distance. If sphere alone or combined sphere and cylinder Rx  $\leq \pm 4.00$ D, vertex compensation is not necessary.

#### 2. For the Cylinder

Adjust the axis by the drift angle using the LARS method. Choose a cylinder that is  $\leq 0.50D$  from the refractive cylinder.

#### 3. Case Examples

#### **Example 1**

Manifest (spectacle) refraction:

O.D. -2.50D / -1.25D x 180° 20/20

O.S. -2.00D / -1.00D x 180° 20/20

Choose a diagnostic lens for each eye with axis 180°. Place the lens on each eye and allow a minimum of 3 minutes for it to equilibrate, based on the patient's initial response to the lens. If the lens has not yet stabilized, recheck until stable.

Check the orientation of the axis mark. If the bottom axis mark is in the 6 o'clock position on both eyes, choose the appropriate cylinder as listed previously. If the lens has not yet stabilized, recheck until stable.

Here is the Rx Prescribed:

O.D. -2.50D / -1.25D x 180°

O.S. -2.00D / -0.75D x 180°

CR-5969 v3 0



#### **Example 2**

Manifest (spectacle) refraction: O.D. -3.00D / -1.00D x 90° 20/20 O.S. -4.75D / -2.00D x 90° 20/20

Choose diagnostic lenses of -3.00D / -0.75D x 90° for the right eye and -4.50D / -1.75D x 90° for the left eye, the nearest lenses available to the spherical power, cylinder power, and axis needed. For the left eye, since the manifest refraction called for -4.75D, compensating for vertex distance the sphere is reduced by 0.25D to -4.50D. The cylinder power will be -1.75D. Place the lens on each eye and allow a minimum of 3 minutes for it to equilibrate, based on the patient's initial response to the lens. If the lens has not yet stabilized, recheck until stable.

#### Right Eve

The orientation mark on the right lens rotates left from the 6 o'clock position by 10° and remains stable in this position. Compensation for this rotation should be done as follows:

Compensate the 10° axis drift by adding it to the manifest refraction axis.

Here is the Rx Prescribed: O.D. -3.00D / -0.75D x 100°

#### Left Eye

The orientation mark on the left lens rotates right from the 6 o'clock position by 10° and remains stable in this position.

Compensate for the 10° axis drift by subtracting it from the manifest refraction axis.

Here is the Rx Prescribed: O.S. -4.50D / -1.75D x 80°

If vision is acceptable, perform a slit lamp examination to assess adequate fit (centration and movement). If fit is acceptable, dispense the lenses instructing the patient to return in one week for reassessment (see dispensing and follow-up information in PATIENT MANAGEMENT).

All patients should be supplied with a copy of the PATIENT INSTRUCTION GUIDE for these lenses. Copies are available for download at www.acuvue.com.

CR-5969 v3 0


# MONOVISION FITTING GUIDELINES

#### A. Patient Selection

#### 1. Monovision Needs Assessment

For a good prognosis, the patient should have adequately corrected distance and near visual acuity in each eye. The amblyopic patient or the patient with significant astigmatism (greater than 1.00D) in one eye may not be a good candidate for monovision correction with these lenses.

Occupational and environmental visual demands should be considered. If the patient requires critical vision (visual acuity and stereopsis), it should be determined by trial whether this patient can function adequately with monovision correction. Monovision contact lens wear may not be optimal for activities such as:

- visually demanding situations such as operating potentially dangerous machinery or performing other potentially hazardous activities; and
- driving automobiles (e.g., driving at night). Patients who cannot meet state driver's licensing requirements with monovision correction should be advised to not drive with this correction, OR may require that additional over-correction be prescribed.

#### 2. Patient Education

All patients do not function equally well with monovision correction. Patients may not perform as well for certain tasks with this correction as they have with spectacles (multifocal, bifocal, trifocal, readers, progressives). Each patient should understand that monovision, as well as other presbyopic alternatives, can create a vision compromise that may reduce visual acuity and depth perception for distance and near tasks. Therefore, caution should be exercised when the patient is wearing the correction for the first time until they are familiar with the vision provided in visually challenging environments (e.g., reading a menu in a dim restaurant, driving at night in rainy/foggy conditions, etc.). During the fitting process, it is necessary for the patient to realize the disadvantages as well as the advantages of clear near vision and straight ahead and upward gaze that monovision contact lenses provide.


#### **B. Eye Selection**

#### 1. Ocular Preference Determination Methods

Generally, the non-dominant eye is corrected for near vision. The following two methods for eye dominance can be used.

Method 1: Determine which eye is the "sighting eye." Have the patient point to an object at the far end of the room. Cover one eye. If the patient is still pointing directly at the object, the eye being used is the dominant (sighting) eye.

Method 2: Determine which eye will accept the added power with the least reduction in vision. Place a hand-held trial lens equal to the spectacle near ADD in front of one eye and then the other while the distance refractive error correction is in place for both eyes. Determine whether the patient functions best with the near ADD lens over the right or left eye.

#### 2. Other Eye Selection Methods

Other methods include the "Refractive Error Method" and the "Visual Demands Method."

#### Refractive Error Method

For anisometropic correction, it is generally best to fit the more hyperopic (less myopic) eye for distance and the more myopic (less hyperopic) eye for near.

#### Visual Demands Method

Consider the patient's occupation during the eye selection process to determine the critical vision requirements. If a patient's gaze for near tasks is usually in one direction, correct the eye on that side for near.

Example: A secretary who places copy to the left side of the desk will function best with the near lens on the left eye.

# C. Special Fitting Characteristics

#### 1. Unilateral Vision Correction

There are circumstances where only one contact lens is required. As an example, an emmetropic patient would only require a near lens, whereas a bilateral uld require corrective lenses on CR-5969 v3 0


both eyes.

#### Examples:

A presbyopic emmetropic patient who requires a +1.75D ADD would have a +1.75D lens on the near eye and the other eye left without correction.

A presbyopic patient requiring a +1.50D ADD who is -2.50D myopic in the right eye and -1.50D myopic in the left eye may have the right eye corrected for distance and the left uncorrected for near.

#### 2. Near ADD Determination

Always prescribe the lens power for the near eye that provides optimal near acuity at the midpoint of the patient's habitual reading distance. However, when more than one power provides optimal reading performance, prescribe the least plus (most minus) of the powers.

#### 3. Trial Lens Fitting

A trial fitting is performed in the office to allow the patient to experience monovision correction. Lenses are fit according to the GENERAL FITTING GUIDELINES for base curve selection described in this Package Insert.

Case history and standard clinical evaluation procedure should be used to determine the prognosis. Determine the distance correction and the near correction. Next determine the near ADD. With trial lenses of the proper power in place, observe the reaction to this mode of correction.

Allow the lenses to settle for about 20 minutes with the correct power lenses in place. Walk across the room and have the patient look at you. Assess the patient's reaction to distance vision under these circumstances. Then have the patient look at familiar near objects such as a watch face or fingernails. Again assess the reaction. As the patient continues to look around the room at both near and distance objects, observe the reactions. Only after these vision tests are completed should the patient be asked to read print. Evaluate the patient's reaction to large print (e.g., typewritten copy) at first and then graduate to newsprint and finally smaller type sizes.

After the patient's performance under the above conditions is completed, tests of visual acuity and reading ability under CR-5969 v3 0


conditions of moderately dim illumination should be attempted.

An initial unfavorable response in the office, while indicative of a guarded prognosis, should not immediately rule out a more extensive trial under the usual conditions in which a patient functions.

#### 4. Adaptation

Visually demanding situations should be avoided during the initial wearing period. A patient may at first experience some mild blurred vision, dizziness, headaches, and a feeling of slight imbalance. You should explain the adaptational symptoms to the patient. These symptoms may last for a brief minute or for several weeks. The longer these symptoms persist, the poorer the prognosis for successful adaptation.

To help in the adaptation process, the patient can be advised to first use the lenses in a comfortable familiar environment such as in the home.

Some patients feel that automobile driving performance may not be optimal during the adaptation process. This is particularly true when driving at night. Before driving a motor vehicle, it may be recommended that the patient be a passenger first to make sure that their vision is satisfactory for operating an automobile. During the first several weeks of wear (when adaptation is occurring), it may be advisable for the patient to only drive during optimal driving conditions. After adaptation and success with these activities, the patient should be able to drive under other conditions with caution.

#### **D. Other Suggestions**

The success of the monovision technique may be further improved by having the patient follow the suggestions below:

- Have a third contact lens (distance power) to use when critical distance viewing is needed.
- Have a third contact lens (near power) to use when critical near viewing is needed.
- Having supplemental spectacles to wear over the monovision contact lenses for specific visual tasks may improve the success of monovision correction. This is particularly applicable for those patients who cannot meet state driver's licensing requirements with monovision correction.
- Make use of proper illumination when carrying out visual tasks.
   CR-5969 v3 0


Monovision fitting success can be improved by the following suggestions:

- Reverse the distance and near eyes if a patient is having trouble adapting.
- Refine the lens powers if there is trouble with adaptation. Accurate lens power is critical for presbyopic patients.
- Emphasize the benefits of clear near vision and straight ahead and upward gaze with monovision.

The decision to fit a patient with monovision correction is most appropriately left to the Eye Care Professional in conjunction with the patient after carefully considering the patient's needs.

All patients should be supplied with a copy of the PATIENT INSTRUCTION GUIDE for these lenses. Copies are available for download at www.acuvue.com.

#### PATIENT MANAGEMENT

#### Dispensing Visit

Each sterile lens is supplied in a foil-sealed plastic package containing buffered saline solution with methyl ether cellulose. To remove the lens from the container, peel back the foil seal, place a finger on the lens, and slide the lens up the side of the bowl of the lens package until it is free of the container.

- Evaluate the physical fit and visual acuity of the lens on each eye.
- Teach the patient how to apply and remove his or her lenses.
- Explain daily disposable lens wear and schedule a follow-up examination.
- Provide the patient with a copy of the PATIENT INSTRUCTION GUIDE for these lenses. Copies are available for download at www.acuvue.com.

REVIEW THESE INSTRUCTIONS WITH THE PATIENT SO THAT HE OR SHE CLEARLY UNDERSTANDS THE PRESCRIBED WEARING AND REPLACEMENT SCHEDULES.

#### **Follow-Up Examinations**

Follow-up care (necessary to ensure continued successful contact lens wear) should include routine periodic progress examinations, management of specific problems, if any, and a review with the patient of the wear schedule, daily disposable


Recommended Follow-up Examination Schedule (complications and specific problems should be managed on an individual patient basis):

- One week from the initial lens dispensing to patient
- 2. One month post-dispensing
- 3. Every three to six months thereafter

 $\ensuremath{\text{NOTE:}}$  Preferably, at the follow-up visits, lenses should be worn for at least six hours.

#### Recommended Procedures for Follow-up Visits:

- 1. Solicit and record patient's symptoms, if any.
- Measure visual acuity monocularly and binocularly at distance and near with the contact lenses.
- Perform an over-refraction at distance and near to check for residual refractive error.
- With the biomicroscope, judge the lens fitting characteristics (as described in the GENERAL FITTING GUIDELINES) and evaluate the lens surface for deposits and damage.
- 5. Following lens removal, examine the comea and conjunctiva with the biomicroscope and fluorescein (unless contraindicated).
  - The presence of vertical corneal striae in the posterior central cornea and/or corneal neovascularization is indicative of excessive corneal edema.
  - The presence of corneal staining and/or limbal-conjunctival hyperemia can be indicative of an unclean lens, a reaction to solution preservatives, excessive lens wear and/or a poorly fitting lens.
  - Papillary conjunctival changes may be indicative of an unclean and/or damaged lens.
- Periodically perform keratometry and spectacle refractions. The values should be recorded and compared to the baseline measurements.

If any observations are abnormal, use professional judgment to alleviate the problem and restore the eye to optimal conditions. If


the criteria for successful fit are not satisfied during any follow-up examinations, repeat the patient's trial fitting procedure and refit the patient.

# WEARING SCHEDULE

The wearing schedule should be determined by the Eye Care Professional. Regular checkups, as determined by the Eye Care Professional, are also extremely important.

Patients tend to overwear the lenses initially. The Eye Care Professional should emphasize the importance of adhering to the initial maximum wearing schedule. Maximum wearing time should be determined by the Eye Care Professional based upon the patient's physiological eye condition, because individual response to contact lenses varies.

The maximum suggested wearing time for these lenses is:

| Day | Hours |
|-------------|------------------|
| 1 | 6-8 |
| 2 | 8-10 |
| 3 | 10-12 |
| 4 | 12-14 |
| 5 and after | all waking hours |

# REPLACEMENT SCHEDULE

These lenses are indicated for daily disposable wear and should be discarded upon removal.

# LENS CARE DIRECTIONS

When lenses are prescribed for daily disposable wear, the Eye Care Professional should provide the patient with appropriate and adequate warnings and instructions for daily disposable lens wear at the time they are dispensed.

CR-5969 v3 0



The Eye Care Professional should review with patients that no cleaning or disinfection is needed with daily disposable lenses. Patients should always dispose of lenses when they are removed and have spare lenses or spectacles available.

#### **Basic Instructions**

- Always wash, rinse, and dry hands before handling contact lenses.
- Do not use saliva or anything other than the recommended solutions for lubricating or rewetting lenses. Do not put lenses in the mouth.
- Eye Care Professionals may recommend a lubricating/rewetting solution which can be used to wet (lubricate) lenses while they are being worn to make them more comfortable.

# Care for a Sticking (Non-Moving) Lens

If the lens sticks (stops moving), the patient should be instructed to apply a few drops of the recommended lubricating or rewetting solution directly to the eye and wait until the lens begins to move freely on the eye before removing it. If non-movement of the lens continues after a few minutes, the patient should immediately consult the Eye Care Professional.

# **EMERGENCIES**

The patient should be informed that if chemicals of any kind (household products, gardening solutions, laboratory chemicals, etc.) are splashed into the eyes, the patient should: FLUSH EYES IMMEDIATELY WITH TAP WATER AND IMMEDIATELY CONTACT THE EYE CARE PROFESSIONAL OR VISIT A HOSPITAL EMERGENCY ROOM WITHOUT DELAY.

# **HOW SUPPLIED**

Each UV-blocking sterile lens is supplied in a foil-sealed plastic package containing buffered saline solution with methyl ether cellulose. The plastic package is marked with the following:

- ACUVUE OASYS® 1-Day: base curve, power, diameter, lot number, and expiration date
- ACUVUE OASYS® 1-Day for ASTIGMATISM: base curve, power, diameter, cylinder, axis, lot number, and expiration date
   CR-5969 v3 0


# REPORTING OF ADVERSE REACTIONS

All serious adverse experiences and adverse reactions observed in patients wearing these lenses or experienced with these lenses should be reported to:

Johnson & Johnson Vision Care, Inc. 7500 Centurion Parkway Jacksonville, FL 32256 USA Tel: 1-800-843-2020 www.acuvue.com Johnson & Johnson Vision Care, Inc. 7500 Centurion Parkway Jacksonville, FL 32256 USA

Tel: 1-800-843-2020 **www.acuvue.com** 



©Johnson & Johnson Vision Care Companies 2016 In Canada: Johnson & Johnson Vision Care, division of Johnson & Johnson, Inc. In USA: Johnson & Johnson Vision Care, Inc. Printed in USA.

Revision date: 09/16

Revision number: AO-03-16-13

ACUVUE OASYS® and HydraLuxe™ are Trademarks of CR-5969 v30hnson & Johnson & Trademarks of Care Companies 

# APPENDIX D: LIPVIEW II MANUFACTURER INSTRUCTIONS


# \*TearScience®

# **OLIPIVIEW®**

Ocular Surface Interferometer

# Instructions for Use

Model LVI-2000 running Software Version 3.X

# Manufactured by:

TearScience, Inc.
5151 McCrimmon Parkway Suite 250
Morrisville, NC 27560
Phone: (919) 467-4007

Fax: (919) 467-3300



Donawa Lifescience Consulting Piazza Albania, 10 00153 Rome, Italy









"TearScience" and "LipiView" are registered trademarks of TearScience, Inc. in the United States and other jurisdictions. All other product or company names that may be mentioned in this publication are trade names, trademarks or registered trademarks of their respective owners.

| | Revision History | | |
|---|---|---|---|
| Revision | Date | Description of Changes | ECR # or PCR # |
| A | 19 Nov 2014 | Initial release of Instructions for Use for LipiView II/3.x software. | P1407211 |
| В | 31 July 2015 | Made updates for software version 3.11. Replaced Figure 6. Fixed minor typographical and formatting errors. | P1502121 |
| С | 1 February 2016 | Previous revisions of this document were numbered 012051-ENG. To accommodate the release of varied English versions, this document is now numbered as 012051-US with the following applicable changes: | P1601281 |
| | | Removed phrase "All of these image types can be photographically documented and visually monitored" from Indications for Use. | |
| | | Removed information pertaining to Model LVI-1001. | |
| | | Updated phototoxicity warning with ISO 15004-2 required information. | |
| | | Clarified patient contact components and added disinfection of Lid Everter to Device Description and Warning sections (already described in Cleaning and Instructions sections of the manual). | |
| | | Added inspection of Lid Everter to Device Description and Instructions. | |
| | | Added USB mouse and keyboard to Accessory Support. | |
| | | Updated recording time from 10 to 5 seconds in Capture Ocular Images procedure. | |
| | | Updated document copyright date to 2016. | |

# **Contents**

| 1 INTR | ODUCTION | 5 |
|-----------|------------------------------------------------|------|
| 2 Імро | RTANT DEVICE INFORMATION | 6 |
| 2.1 | Indications for Use | 6 |
| 2.2 | Contraindications | 6 |
| 2.3 | Precautions | 6 |
| 2.4 | Warnings | 6 |
| 2.5 | Potential Adverse Effects | 9 |
| 2.6 | Labeling | 9 |
| 2.7 | Device Description and Overview | .10 |
| 2.7.1 | Base with Computer System and Electronics | .13 |
| 2.7.2 | Forehead and Chin Rest with Fluted Roller | .14 |
| 2.7.3 | Motion Stage | .14 |
| 2.7.4 | Camera and Attached Lens | .14 |
| 2.7.5 | | |
| 2.7.6 | Pushbutton Controls | .14 |
| 2.7.7 | Touchscreen Display with Pivoting Arm | .14 |
| 2.7.8 | | |
| 2.7.9 | Handheld Near Infrared (IR) Lid Everter | .15 |
| 2.7.1 | | |
| 2.7.1 | | .15 |
| 2.8 | Storage and Transport | . 16 |
| 2.9 | Installation, Maintenance and Servicing | .16 |
| 2.10 | Cleaning | |
| 2.11 | Disposal | .17 |
| 2.12 | Warranty | .17 |
| 3 Inste | RUCTIONS FOR USE | .18 |
| 3.1 | Startup and Login | 18 |
| 3.2 | First Time Device Setup | 19 |
| 3.3 | Menu Bar | |
| 3.4 | Enter and Select a Patient and Imaging Mode | 21 |
| 3.5 | Capture Tear Film Images (Lipid Imaging Mode) | 22 |
| 3.6 | Review Tear Film Images (Lipid Imaging Mode) | |
| 3.7 | Capture Gland Images (Gland Imaging Mode) | 27 |
| 3.8 | Review Gland Images (Gland Imaging Mode) | |
| 3.9 | Capture Ocular Images (Ocular Imaging Mode) | 34 |
| 3.10 | Review Ocular Images (Ocular Imaging Mode) | 36 |
| 3.11 | Log Out and Power Off | |
| | BLESHOOTING GUIDE | |
| A DDENING | V. FI ECTROMACNETIC COMPATIBILITY DECLIREMENTS | 44 |

# **Figures**

| Figure 1. Front (Patient) View of LipiView II | |
|---|---|
| Figure 2. Rear (User) View of LipiView II | 12 |
| Figure 3. Handheld Near Infrared (IR) Lid Everter | 13 |
| Figure 4. External Connectors on Underside of Base | 13 |
| Figure 5. Warning Screen | 18 |
| Figure 6. Initialization Screen | 18 |
| Figure 7. Login Screen | 18 |
| Figure 8. Patient Records Screen | 19 |
| Figure 9. Main Admin Screen | |
| Figure 10. Menu Bar | 20 |
| Figure 11. Patient Records Screen | 21 |
| Figure 12. Patient Entry Screen. | 21 |
| Figure 13. Capture/View Screen | |
| Figure 14. Lipid Image Capture Screen with Labeled Controls | 23 |
| Figure 15. Export Dialog | 24 |
| Figure 16. Interferometric Colors | 24 |
| Figure 17. Review Lipid Images Screen with Labeled Controls | 25 |
| Figure 18. Example OD Image - Average Lipid Layer Thickness 39 nm | 26 |
| Figure 19. Example OS Image – Average Lipid Layer Thickness 100+ nm | 26 |
| Figure 20. Everting Lower Eyelid using Handheld Near IR Lid Everter | 28 |
| Figure 21. Everting Upper Eyelid using Cotton Swab | 28 |
| Figure 22. Gland Image Capture Screen with Labeled Controls | 29 |
| Figure 23. Pushbutton Controls (on top of unit) | 30 |
| Figure 24. Properly Focused Lower Lid Images: Reflected IR and Trans IR | 31 |
| Figure 25. Gland Example Images: No Dropout, Medium Dropout, High Dropout | |
| Figure 26. Gland Dilation Example, Lower Lid | 32 |
| Figure 27. Review Gland Images Screen with Labeled Controls | 33 |
| Figure 28. Ocular Image Capture Screen with Labeled Controls | 35 |
| Figure 29. Review Ocular Images with Labeled Controls | 36 |
| Tables | |
| Table 1: General and Operation Warnings | 7 |
| Table 2. Symbols Used on LipiView II Labeling | |
| Table 3. System and Environmental Specifications | |
| Table 4: LipiView II Cleaning Information | |
| Table 5. Main Admin Functions | |
| Table 6: Troubleshooting Unexpected Events | |
| Table 7. Operational System Messages and Descriptions | |
| Table 8: Guidance and Manufacturers Declaration-Electromagnetic Emissions | 44 |
| Table 9: Guidance and Manufacturers Declaration-Electromagnetic Immunity (part 1) | |
| Table 10: Guidance and Manufacturers Declaration-Electromagnetic Immunity (part 2) | |
| Table 11: Recommended Separation Distances Between Portable and Mobile RF | = • |
| Communications Equipment and LipiView II | 47 |
| | , |
| 012051-US Rev C | |

© 2016 TearScience, Inc.

CR-5969 v3 0

#### 1 Introduction

This manual provides the indications, contraindications, warnings, precautions, potential adverse effects and instructions for use for the *TearScience* LipiView II Ocular Surface Interferometer. Carefully read this manual in its entirety before using LipiView II. Failure to follow these instructions may result in improper use of the device.

This manual provides essential information for safe and proper use of LipiView II.

- Section 2 (Important Device Information: indications, contraindications, warnings, precautions, potential adverse effects, device description, storage and transport, service and maintenance, cleaning, disposal and warranty)
- Section 3 (Instructions for Use for Start-up, First Time Setup, Lipid Imaging, Gland Imaging and Ocular Imaging)
- Section 4 (Troubleshooting Guide)

The *LipiView II Administrator's Guide* contains information about the setup and administration of LipiView II.

 Prior to initial use of LipiView II, refer to Section 3.2 of this manual and/or the Administrator's Guide to ensure proper setup (including requirements for operator (user) names, passwords, network connections and file storage.)

NOTE: LipiView II has a firewall and disabled remote access to protect the device and ensure privacy of patient records over a network. However, if LipiView II is connected to a non-secure wireless network, exported patient data will not be protected from unauthorized access. TearScience recommends the LipiView II be connected to a password-protected wireless router utilizing the WPA or WPA2 security protocols to ensure protection of the device and patient records.

Strong passwords do not contain words that appear in a dictionary, are at least six characters long, and consist of a mixture of letters and numbers. TearScience recommends that you choose a strong password and change it regularly (for example, every 90 days.)

Contact TearScience (in North America, at +1 919 459 4891 or by email at customerservice@tearscience.com) with any questions about the information contained in this manual or for additional information on the safe and proper operation of LipiView II.

# 2 Important Device Information

# 2.1 Indications for Use

The LipiView II Ocular Surface Interferometer is an ophthalmic imaging device intended for use by a physician in adult patients to capture, archive, manipulate and store digital images of:

- Specular (interferometric) observations of the tear film. Using these images, LipiView
   II measures the absolute thickness of the tear film lipid layer.
- Meibomian glands under near-infrared (NIR) illumination
- The ocular surface and eyelids under white illumination

# 2.2 Contraindications

Contraindications are conditions in which the device should not be used because the risk of use clearly outweighs any benefit. No contraindications have been identified for LipiView II.

# 2.3 Precautions

The following patient conditions may affect the interferometry assessment of a patient's tear film using LipiView II:

- Use of ophthalmic drops such as artificial tear lubricants, ointments, and medications. Advise patients not to instill oil-based ophthalmic drops (e.g., Soothe®, Restasis®, Systane Balance®) for at least 12 hours prior to device use and not to instill ointments for at least 24 hours prior to device use. Wait at least 4 hours after instillation of all other ophthalmic drops prior to device use.
- **Soft or rigid contact lens wear.** Advise patients to remove contact lenses at least 4 hours prior to device use.
- Use of oil-based facial cosmetics around the eye.
- Eye rubbing.
- Recent swimming in a chlorinated pool. Advise patients not to swim for at least 12 hours prior to device use.
- Any ocular surface condition that affects the stability of the tear film. These conditions
  include disease, dystrophy, trauma, scarring, surgery, or abnormality.

# 2.4 Warnings

Review the warnings in Table 1 prior to using LipiView II.

#### **Table 1: General and Operation Warnings**



#### GENERAL WARNINGS

WARNING: No modification of this equipment is allowed.

*Caution:* Power Requirements. The LipiView II is a continuous operation device which requires a power source of 100-240 Volts AC  $\pm$  10%, 50/60 Hz single phase, 4 Amps. Connection to a power supply other than a supply mains with protective earth may result in electric shock.



Caution: The LipiView II has protection against electric shock of applied part classified as Type B. This device is classified as an IEC Class 1 product.

Caution: Voltage Protection and Fuse Selection. Contact TearScience to replace a blown fuse. TearScience personnel must replace only with a 5 x 20 mm, 4 A, 300 ms, 40 A breaking capacity fuse to avoid risk of fire. TearScience personnel must disconnect from power before servicing to avoid risk of electrical shock.

Caution: Backup Battery Replacement. Backup battery cannot be replaced.

*Caution:* Keep the LipiView II away from strong magnetic fields as it could damage the device's hard drive, but is not a safety hazard to the user or patient.

Caution: This equipment is intended for use by healthcare professionals only. This equipment may cause radio interference or may disrupt the operation of nearby equipment. It may be necessary to take mitigation measures, such as re-orienting or relocating the LipiView II or shielding the location.

*Caution:* Portable and mobile RF communications equipment can affect MEDICAL ELECTRICAL EQUIPMENT.

Caution: The use of ACCESSORIES, transducers and cables other than those specified, with the exception of transducers and cables sold by the manufacturer of the EQUIPMENT or DEVICE as replacement parts for internal components, may result in increased EMISSIONS or decreased IMMUNITY of the EQUIPMENT or DEVICE.

*Caution:* The EQUIPMENT or DEVICE should not be used adjacent to or stacked with other equipment and if adjacent or stacked use is necessary, the EQUIPMENT or DEVICE should be observed to verify normal operation in the configuration in which it will be used.

*Caution*: Degree of protection against harmful ingress of liquid: IPX0. This equipment has no protection against ingress of liquids.

Caution: This device is not suitable for use in the presence of flammable mixtures.

Caution: This device is not suitable for use in oxygen rich environments.

*Caution:* The device monitor and base unit may exceed 41°C. Device will remain within safe momentary contact temperature, below 51°C.

012051-US Rev C © 2016 TearScience, Inc.






Caution: Federal law restricts this device to sale by or on the order of a physician.

*Caution:* The chin and forehead rest surfaces and Handheld Near IR Lid Everter must be disinfected with alcohol immediately prior to use and prior to storage.

Caution: Photo-toxicity hazard. No acute optical radiation hazards have been identified for LipiView II under intended use conditions. Since prolonged intense light exposure can damage the retina, the use of the device for ocular examination should not be unnecessarily prolonged. The retinal exposure dose for a photochemical hazard is a product of the radiance and the exposure time. Aphakes and persons with diseased eyes will be at greater risk. The risk may also be increased if the person being examined has had any exposure with the same instrument or any other ophthalmic instrument using a visible or near-infrared light source during the previous 24 hours.

**Caution:** The light emitted from this instrument is potentially hazardous. The longer the duration of exposure, the greater the risk of ocular damage. Exposure to light from the instrument when operated at maximum intensity will exceed the safety guideline after 8 hours.

*Caution:* To prevent pinching, do not put fingers near illuminator, lens or chin rest during focusing. Instruct patient not to place hands on LipiView II during operation, and not to put fingers near illuminator, lens or chin rest.

*Caution:* If a problem occurs with LipiView II, identify the symptom then attempt to resolve the problem as indicated in Section 4, *Troubleshooting Guide*. If the problem cannot be resolved, stop using the device and contact TearScience.

*Caution:* To prevent electric shock or performance alteration, do not attempt to service the device or remove the cover. No maintenance is required for LipiView II, and the device and all of its associated parts are not serviceable by the user.

*Caution:* In order to isolate this equipment from supply mains the equipment must be unplugged from the wall. Do not position the equipment in a location which would prevent the unit from being unplugged in an emergency.

*Caution:* Do not store this instrument in conditions where the temperature may rise above 55°C or fall below -10°C.

*Caution:* When lifting or handling LipiView II, caution should be taken to prevent injury or damage to the device. Prior to moving the device, put the monitor arm into a locked position and unplug the power cord from the wall. If an external monitor is attached, disconnect the external monitor prior to moving the device.

Caution: Shock hazard. Do not touch patient and device under top cover simultaneously.

# 2.5 Potential Adverse Effects

There are no known or anticipated adverse effects associated with use of this device.

# 2.6 Labeling

Table 2 provides a description of the symbols used on LipiView II labeling.

Table 2. Symbols Used on LipiView II Labeling

| Label Symbol | Symbol Description |
|---|---|
| <b>*</b> | Type B applied part |
| (i | Consult operating instructions |
| <b>((1)</b> | Device transmits radiofrequency (RF) energy |
| | Text consists of a warning or precaution relating to safety. Read the text carefully and use the equipment as instructed to ensure safety. |
| REF | Reference Number |
| SN | Serial Number |
| Rx only | CAUTION: Federal law restricts this device to sale by or on the order of a physician. |
| 0086 | Mandatory conformity mark for medical device products in the European Economic Area (EEA). The CE marking certifies that a product has met consumer safety, health or environmental requirements. "0086" is the Notified Body Number. |
| C (TIME TEXT US | This model/product is Listed in Intertek's Directory of Listed Products. |



| Label Symbol | Symbol Description |
|---|---|
| | Date of Manufacture |
| | Manufacturer |
| | Temperature Limitation, defining upper and lower temperature limits; used for storage or shipping temperatures. |
| EC REP | Authorized Representative in the European Community |
| P/N | Part Number |
| Rev | Revision Level |

# 2.7 Device Description and Overview

The LipiView II is a bench-top device used as an ophthalmic camera for imaging the lipid layer of the tear film, meibomian glands, ocular surface and eyelids. There are three imaging modes: Lipid, Gland and Ocular.

In Lipid Imaging Mode, LipiView II operates on the principle of white light interferometry and provides an interferometry color assessment of the tear film by specular reflection. The patient's eye is positioned in front of an illumination source directed toward the tear film on the corneal surface. Light from the illumination source passes through the tear film and is specularly reflected into a camera. The light reflecting back through the lens in the camera forms an interference pattern, called an "interferogram." A video image file is recorded over time since the interference pattern changes as the tear film is distributed across the cornea during blinking.

The computer system captures and enhances the interference pattern and displays a profile corresponding to an interferometry color scale. This color scale has been validated to a known standard for measurement of thin film thickness, demonstrating that LipiView II has the ability to make absolute thickness measurements of the tear film lipid layer by the imaging interferometric colors. The measured lipid layer thickness may range from 10 to 240 nanometers (nm), with a precision of 1 nm and an accuracy of  $\pm 10$  nm. The conformance factor of the measured interference pattern is displayed as a "C-factor," which is equal to the proportion of measured colors that match the predicted interferometric color scale. The video image of the ocular surface may be viewed on the computer screen display and in a printed report.



In Gland Imaging Mode, LipiView II uses near infrared (NIR) illumination and an NIR-sensitive camera mounted on a motion control system to image the meibomian glands. The tissue between the meibomian glands and the surface of the eyelid are transparent to NIR light; the glands reflect NIR wavelengths, allowing them to be imaged.

In Ocular Imaging mode, LipiView II captures high-resolution still images or video to record relevant findings on the ocular surface and/or eyelids. The images can be taken using room light only or the device's built-in white light.

LipiView II contains the following components, which are identified in Figure 1 (Front/Patient View) and Figure 2 (Rear/User View):

- Base with Computer System and Electronics
- 2-position Forehead and Chin Rest with Fluted Roller (for height adjustment)
- Motion Stage
- Camera and Attached Lens
- Illuminator
- Pushbutton Controls
- Touchscreen Display with Pivoting Arm
- USB Ports
- Handheld Near Infrared (IR) Lid Everter, shown in Figure 3
- Connections for an External Monitor, the Near Infrared (IR) Lid Everter, and the power cord, shown in Figure 4.



Figure 1. Front (Patient) View of LipiView II

| | Key |
|---|---------------|
| 1 | Forehead Rest |

| 2 | Camera and Attached Lens | - 1 |
|----|------------------------------------------------------------|-----|
| 3 | Illuminator | |
| 4 | Chin Rest | |
| 5 | Fluted Roller (adjusts chinrest height) | |
| 6 | Chin Rest Base 2-position (toward/away from device) adjust | |
| 7 | Motion Stage | |
| 8 | Back of Touchscreen Display | |
| 9 | Pushbutton Controls (on top of unit) | |
| 10 | Base (contains Computer System and Electronics) | |



Figure 2. Rear (User) View of LipiView II

| | Key |
|---|---|
| 1 | Touchscreen Display |
| 2 | USB Port (another is on the other side, and a third is above the power switch) |
| 3 | Power Switch |
| 4 | Motion Stage |
| 5 | Chinrest2-position (toward/away from device) adjust |
| 6 | Base (contains Computer System and Electronics) |
| 7 | Pivoting Arm |




Figure 3. Handheld Near Infrared (IR) Lid Everter



Figure 4. External Connectors on Underside of Base

| Key | |
|-----|------------------------------------------------|
| 1 | Hardwired HDMI connection for external monitor |
| 2 | Connector for Handheld Near IR Lid Everter |
| 3 | Connector for Power Cord |

# 2.7.1 Base with Computer System and Electronics

The base houses the power connection and computer hardware. The base connects with the forehead and chin rest, motion stage and touchscreen display. The on/off power switch (Figure

012051-US Rev C © 2016 TearScience, Inc.


2) is located on the base opposite the chin rest. An external monitor connection is hardwired into the base, as is a connection point for the Near IR lid everter.

#### 2.7.2 Forehead and Chin Rest with Fluted Roller

The adjustable forehead and chin rest is designed to allow proper positioning of the patient's head to capture images. To ensure a properly focused image, the patient must place his/her forehead and chin firmly against the forehead and chin rests. The chin rest may be raised or lowered to accommodate different facial dimensions by spinning the fluted roller. The chin rest has a 2-position adjust (toward the device for Lipid imaging and away from the device for Gland and Ocular Imaging.)

Two canthus alignment marks are located on the left and right sides of the forehead rest. Adjusting the chin rest to position the lateral canthus of the patient's eye at these marks will optimize the range of camera motion.

The forehead and chin rest come in contact with the patient. Disinfect the forehead and chin rest surfaces with alcohol immediately prior to use and prior to storage.

#### 2.7.3 Motion Stage

The motion stage contains the camera, illuminator and motor controls used to adjust the camera and illuminator. The height of the motion stage is adjusted as part of the image capture process, to position the camera correctly.

#### 2.7.4 Camera and Attached Lens

The camera is located inside the motion stage and is not visible externally. The height of the camera is adjusted as part of the motion stage. The camera can also be adjusted left and right and backwards and forwards with separate controls.

#### 2.7.5 Illuminator

The grid-like fixture attached to the motion stage is the illuminator. The height of the illuminator is adjusted as part of the motion stage. There are no separate controls for the illuminator.

#### 2.7.6 Pushbutton Controls

LipiView II includes a pushbutton control keypad on top of the unit that may be used in all modes, to make it easier for the operator to capture images.

# 2.7.7 Touchscreen Display with Pivoting Arm

The touchscreen display is on a pivoting arm, which allows it to be positioned  $\pm$  45 degrees or  $\pm$  90 degrees from its location shown in Figure 1. To reposition the screen, press the button under the pivoting arm while moving the arm left or right to the approximate 45 or 90 degree location. Release the button and continue moving the arm until it locks into place.

012051-US Rev C © 2016 TearScience, Inc.


In addition to displaying images and information to the operator, the screen functions as a touchscreen user interface to the LipiView II. The operator touches the screen to operate the motion stage and camera controls and capture images.

#### 2.7.8 USB Ports

The lower base of the touchscreen display contains three USB ports, located as shown in Figure 2. These ports may be used to connect a printer or storage device.

## 2.7.9 Handheld Near Infrared (IR) Lid Everter

The Handheld Near Infrared (IR) Lid Everter is both a near-infrared light source and a shaped instrument that aids in the proper eversion of the lower eyelid. The Near IR Lid Everter contacts the patient's lower eyelid. Inspect the Near IR Lid Everter to ensure it is intact prior to use. Disinfect the Near IR Lid Everter with alcohol immediately prior to use and prior to storage. Place the Near IR Lid Everter slightly below the lash line and move the instrument slightly inward and upward to evert the entire length of the lower eyelid.

## 2.7.10 Operating Environment and Specifications

System and environmental specifications are displayed in Table 3.

**Table 3. System and Environmental Specifications** 

| Input Voltage | 100 – 240 VAC, 50 – 60 Hz |
|---|---|
| Product Safety Classification | Type B Applied Part |
| IEC 60601-1 — Medical electrical equipment — Part 1: | |
| General requirements for safety | |
| IEC 60601-1-2 — Medical electrical equipment—Part 1: | CISPR 11 (Class A, Group 1) |
| General requirements for safety—Section 2: Collateral | |
| standard—Electromagnetic compatibility—Requirements | |
| and tests; | |
| Accuracy of lipid layer thickness measurement | ±10 nm |
| Operating Temperature | 10°C to 35°C |
| Operating Relative Humidity | Up to 90% non-condensing |
| Atmospheric Pressure | 700 hPa to 1060 hPa |
| Storage Temperature | -10°C to 55°C |
| Transport Temperature | 5°C to 60°C |

## 2.7.11 Accessory Support

LipiView II may be used with the following USB accessories that are compatible with Windows 7 and USB 2.0:

- USB printer (Printer Support)
- USB external hard drive (External Backup Support)

012051-US Rev C © 2016 TearScience, Inc.


- USB flash drive (USB / Thumb Drive Support)
- USB mouse and keyboard (support for optional alternative to touchscreen controls)

LipiView II is designed to operate wirelessly with other network devices, such as a printer. Placement of LipiView II should be within range of the network, if a network system is used.

LipiView II may be used with an external monitor. The hardwired connection in the base will support HDMI or DVI inputs for an off-the-shelf external monitor, which has at least 1280 x 1024 resolution and supports 60Hz frame rates.

# 2.8 Storage and Transport

Before storage, ensure the power switch is off, and the chin and forehead rest surfaces, as well as the Near IR Lid Everter, are cleaned according to the instructions in Section 2.10, *Cleaning*. Store LipiView II in a way that prevents contamination and damage between uses.

For transport, ensure power cord is unplugged and secured off the ground. Grip onto metal portion of the device in two locations: 1) under the base or under the head containing the motion stage; and 2) monitor arm behind the screen. Carefully lift and move the device in an upright position.

# 2.9 Installation, Maintenance and Servicing

There are no specific installation requirements for LipiView II, other than unpacking the device from its carton and connecting power and accessories (the external monitor and Near IR Lid Everter.) The device is installed and ready to use safely and correctly if it passes its Power-On Self Test with no system errors.

LipiView II performs a calibration process at startup. LipiView II does not require preventive maintenance or scheduled calibration. If the touchscreen gets out of calibration, refer to the LipiView II Administrator's Guide for instructions on how to recalibrate the touchscreen using the built-in utility.

Expected life of LipiView II is 5 years. Note that no user serviceable components are inside the unit. For Field Service, contact TearScience in North America at +1 919 459 4891 or by email at customerservice@tearscience.com.

## 2.10 Cleaning

Table 4 identifies the components of LipiView II that require cleaning. For each component, the frequency and method of cleaning is provided.

Table 4: LipiView II Cleaning Information

| Component | Frequency | Method |
|---------------|--------------------------|---------|
| Chin rest and | Immediately prior to | Alcohol |
| forehead rest | use and prior to storage | |

012051-US Rev C

© 2016 TearScience, Inc.


| surfaces | | |
|---|---|---|
| Handheld Near IR | Immediately prior to | Alcohol |
| Lid Everter | use and prior to storage | |
| Camera lens and | Monthly | Wipe with a lint-free photographic quality |
| Illuminator | | lens cloth |
| Touchscreen | When soiled or as | Power off the device. |
| Display Monitor | needed | Apply window or glass cleaner to a |
| | | cloth rag and wipe the screen |
| | | Do not apply cleaner directly to the |
| | | screen |
| | | Do not clean the monitor with |
| | | alcohol, paint thinner, benzene or |
| | | compressed air |
| LipiView II | When soiled or as | Wipe down exterior of the device with |
| exterior, including | needed | a mild soapy cloth |
| keypad | | Do not use bleach, chlorine or |
| | | acetone-based solutions to clean any |
| | | part of the chin rest or the system |
| | | enclosure |
| External monitor | Follow manufacturer's | Follow manufacturer's cleaning |
| | cleaning instructions | instructions |

# 2.11 Disposal

LipiView II consists of an ABS plastic enclosure, aluminum chassis, circuit boards, and electrical components. In the unlikely event that the device is damaged and cannot be repaired, never dispose of the device. Return LipiView II to TearScience using the contact information on the first page of this manual.

# 2.12 Warranty

TearScience, Inc. warrants that each LipiView II: 1) is free from defects in materials and workmanship; and 2) conforms to TearScience Inc.'s official specifications. The warranty period for each LipiView II is one year commencing on the date of purchase. Any tampering or modifications to the device by the user will void the warranty.

## 3 Instructions for Use

# 3.1 Startup and Login

At startup, LipiView II performs a self-test, confirms camera connection, verifies system voltages, checks remaining hard drive space, and calibrates camera motors.



Figure 5. Warning Screen



Figure 6. Initialization Screen



Figure 7. Login Screen

- 1. Ensure the power cord is plugged into an electrical outlet. The power cord connection is located underneath the base of the device.
- Power on LipiView II by pressing the rocker switch on the device base (refer to Figure 2).
   The touchscreen display is initially blank and then displays a "Welcome" message and other messages related to self-test and initialization.
- 3. Press the OK button to acknowledge the warning (Figure 5) after ensuring the patient and operator are clear of the chinrest area. The motion stage moves during system hardware self-test, which takes about 20 seconds.
- 4. Touch the screen to continue when Figure 6 is displayed indicating that the device is ready for use. (Note that the software version displayed may differ from Figure 6.)
- 5. When the Login screen (Figure 7) is displayed, enter the operator name and password using the onscreen keyboard. (Operator name and password are provided by the Administrator or TearScience trainer.) Press *Log In*.

# 3.2 First Time Device Setup

Prior to initial use, ensure that the following instructions are completed by an Administrator. Other administrative functions, detailed in *LipiView II Administrator's Guide*, can be completed at the discretion of the Administrator. LipiView II has been set up with a default Operator Name (LIPIVIEW) and Password (LIPIVIEW) that has administrator privileges. After initial login, it is recommended but not required that the Administrator reset the password.



Figure 8. Patient Records Screen



Figure 9. Main Admin Screen

- 1. Power on the system.
- When the Login screen (Figure 7) is displayed, enter LIPIVIEW for both the Username and Password. (The onscreen keyboard only supports uppercase characters.) Press Log In. The Patient Records screen (Figure 8) is displayed.
- 3. Press the Gear icon [ on Menu bar (Figure 10) located in the upper right corner of the screen. The Main Admin screen (Figure 9) is displayed.
- Press Operator Setup. Add additional operator usernames and set or change passwords as needed.

Before capturing images, it is also recommended that the following items be set up using the functions on the Main Admin screen (Table 5).

## From Main Admin screen (Figure 9):

- 5. Press *Practice Info* to enter Practice Information.
- 6. Press System Info, then Press Set Date and Time to set System Date and Time.
- 7. Press *Network* to set up network connections.
- 8. Press *Close* to return to the Patient Records screen (Figure 8).

**Table 5. Main Admin Functions** 

| System Info | System information, including software versions and important utilities |
|---|---|
| | (Calibrate Touchscreen, Set Date and Time, Set Up System for Packaging, |
| · | |
| | Launch Remote Support, Software Update, Save Changes and Shut Down, Save |
| | as PDF) |
| Practice Info | Enter the name and business information for the medical practice |
| System Log | View the system log, which collects information about key system events and |
| | errors (useful for troubleshooting and technical support) |
| Operator Setup | Add or delete Operators (users) and/or Administrator |
| Export Setup | Select file formats for records export |
| Network | View network information |
| Hardware Status | See comprehensive status information for the hardware and software |
| Traceability Log | View records of all traceable events to ensure data integrity (e.g., users |
| | added/deleted, treatment records moved from one patient to another) |
| System Options | Set the automatic logout timer, choose display options |
| Modality | Set options for Lipid Imaging or Gland Imaging modes |
| Configuration | |
| Usage Summary | View statistics about use, selected by configurable criteria |
| Data Management | Delete or move patient records (creates a permanent record in the Traceability |
| _ | Log) |
| Backup/Restore | Backs up or restores LipiView II patient and treatment data to networked drive |
| | or other media |

#### 3.3 Menu Bar

The menu bar (Figure 10), shown at the top of the screen, has the following icons.



Figure 10. Menu Bar

| | Key |
|---|---|
| 1 | Patients Button – Touch to return to Patient Records screen (Figure 11) |
| 2 | Drawer Dropdown - Contains information on current patient and active imaging session |
| | (if any). Pull down to access patient history. |
| | When on Image Capture screens or Review Image screens, press <i>Capture/View Button</i> on |
| i | menu bar to return to Capture/View screen (Figure 13). |
| 3 | Admin - Touch to access Administrator screens (requires access privileges) |
| 4 | Log Out |

012051-US Rev C © 2016 TearScience, Inc.


# 3.4 Enter and Select a Patient and Imaging Mode

After Login, enter a new patient or search for an existing patient. Select the patient to capture new images or view prior images. Then, select an imaging mode.



Figure 11. Patient Records Screen



Figure 12. Patient Entry Screen



Figure 13. Capture/View Screen

1. For a *New Patient*, select *Add Patient* on Patients Records screen (Figure 11) to display Patient Entry screen (Figure 12).

- 2. Using onscreen keyboard, enter patient information, then press *Save*. Patient records must include at a minimum:
  - 1) Patient ID or
  - 2) Last Name, First Name and Date of Birth (enter the month and date as two-digit numbers, and the year as a four-digit number: MM/DD/YYYY).
- For an *Existing Patient*, enter patient data (patient ID or name) in Search field on Patient Records screen (Figure 11) to locate the record. To edit patient data, press Pencil icon to the right of the list.
- 4. Select the desired patient record from the patient listing table.

NOTE: The step keys can be used to move backwards or forwards through the table. When the list spans multiple pages, sort the table by pressing the header field by the desired column. Press the same header a second time to sort the table in the reverse order. A small triangle in the column header indicates the table is being displayed by this column. The triangle points down or up to specify the sorting direction.

5. When Capture/View screen (Figure 13) displays, select an imaging mode (Lipid Imaging, Gland Imaging or Ocular Imaging) to capture new images or view prior images for that patient. Select *All Exams* to view all images in the patient's history.

012051-US Rev C © 2016 TearScience, Inc.


#### 3.5 Capture Tear Film Images (Lipid Imaging Mode)

- 1. To image the tear film lipid layer by specular reflection of light, select Lipid Imaging from the Capture/View screen (Figure 13) and press New.
- 2. Disinfect the forehead and chin rest with alcohol prior to use.
- 3. Ensure the chin rest is in closest position toward the device.
- 4. Place the patient's chin fully forward into chin rest and forehead firmly against forehead rest. Adjust the height of the chin rest by spinning the fluted roller until the temporal canthus is aligned with the marks on the left and right sides of the forehead rest. Instruct the patient to look at the orange fixation light.

CAUTION: To prevent pinching, do not put fingers near illuminator, lens or chin rest during focusing. Instruct patient not to place hands on LipiView II during operation, and not to put fingers near illuminator, lens or chin rest.

- 5. Select OD (right eye) or OS (left eye) to image by touching the right or left side of the Lipid Image Capture screen (Figure 14).
- 6. Position the camera using one or a combination of methods: 1) If the pupil is visible on screen, press autoposition reticle to automatically center the camera on the pupil. 2) Touch the desired location (toward pupil) on screen, which will automatically move the camera and center on the location. 3) Press the manual position buttons, as needed, until the pupil appears in the center of the screen. (You may also use the keypad to position the camera.)

#### NOTE: Ensure the lower lid margin is visible to evaluate partial blinking

7. Focus the camera using one or a combination of methods: 1) Press autofocus reticle to focus (not necessary if reticle was already pressed to position camera); 2) press fine focus buttons to adjust the focus until the tear film image is clear. (You may also use the keypad to focus the camera.)

### NOTE: If the tear film image is not in focus, invalid video data may be saved.

- 8. Press Capture button to begin recording approximately 20 seconds of video. The blinking red light indicates LipiView II is recording. Press Capture button again to stop recording prior to 20 seconds, if desired.
- 9. Instruct the patient to blink naturally or to perform a squeezed blink, as desired.
- 10. When recording is complete, the illuminator turns off. Press *Notes* to add any notes to images, if desired.
- 11. Review video using onscreen playback button. If image quality is suboptimal, delete video using Trashcan icon and recapture another image.
- 12. Repeat steps 5 to 11 to capture an image of the other eye, if desired.
- 13. Press *Analyze* to save and process the image(s).

012051-US Rev C © 2016 TearScience, Inc.




Figure 14. Lipid Image Capture Screen with Labeled Controls

| | Key |
|---|---|
| 1 | Magnify View Icon - OD (right eye) is currently in view. OS (left eye) side is currently |
| | greyed out. Touch icon to capture images for OS (left eye). |
| 2 | Capture Video Button - Press to begin recording. Appears as a rectangle during recording; |
| | press rectangle to stop recording before 20 seconds. |
| 3 | Select Position/Focus Button - Press to toggle display of manual focusing and positioning |
| | button controls on or off. |
| 4 | Autoposition/Autofocus Reticle - Once the pupil is visible on screen, press the reticle to |
| | automatically center and focus the image. |
| 5 | Manual Fine Focus Buttons - Press plus or minus to focus image |
| 6 | Manual Positioning Buttons - Press to move camera left, right, up or down |
| 7 | Eye Position Indicator - Indicates the eye being imaged (OD in figure) |
| 8 | Analyze Button - Press to save, process and analyze captured imagery |
| 9 | Notes Button - Press to open notes field for text entry |

012051-US Rev C © 2016 TearScience, Inc.


# 3.6 Review Tear Film Images (Lipid Imaging Mode)

- 1. After pressing *Analyze* on the Lipid Image Capture screen (Figure 14), the Review Lipid Images screen (Figure 17) appears with the tear film lipid layer images.
- 2. To review prior tear film lipid images for an existing patient:
  - a. Select the patient from the Patient Records screen (Figure 11).
  - b. On the Capture/View screen (Figure 13), select Lipid Imaging to view prior lipid images or select All Exams to view all prior images.
  - c. A list of prior images is displayed on the Capture/View screen (Figure 13). Drag and drop the desired images from the list to the sides of the screen marked "Drop Here". Touch the image again to display the Review Lipid Images screen (Figure 17).



Figure 15. Export Dialog

- 3. Playback the video using onscreen controls.
- 4. If desired, press Export icon on the Review Lipid Images screen (Labeled 8 in Figure 17) to export or print images or report.
- From the Export dialog (Figure 15), press the button to save images, video or report to an external medium or network, or print a report. Exported images can be displayed with or without patient demographics.

The Review Lipid Images screen (Figure 17) displays numerical and graphical analysis of the measured lipid layer thickness in nanometers (nm) from 10 (thinnest) to 240 (thickest), with a precision of 1 nm and an accuracy of 10 nm. The interferometric color scale (Figure 16) has been validated to a known standard for measurement of thin film thickness. By comparison to this known standard, the lipid layer thickness values are absolute thickness measurements of the tear film lipid layer.



Figure 16. Interferometric Colors

NOTE: If analysis cannot be performed, a message NO VALID ANALYSIS DATA FOR VIDEO replaces the graph, and the numerical information shows as dashes (- - -).

012051-US Rev C © 2016 TearScience, Inc.


CR-5969 v3 0





Figure 17. Review Lipid Images Screen with Labeled Controls

| | Key |
|---|---|
| 1 | Interferometric Color Scale - Corresponds to lipid layer thickness value in nm |
| 2 | Video Playback Controls - Press to play, pause, forward step, reverse step |
| 3 | Full Screen Mode – Press to view screen in full screen mode |
| 4 | Numerical Analysis: |
| | <ul> <li>Avg LLT: Average lipid layer thickness in nm displayed in colored font corresponding to thickest (yellow),<br/>medium thickness (orange) and thinnest (red).<sup>1</sup></li> </ul> |
| | Max: Maximum lipid layer thickness in nm recorded for a given video frame. |
| | Min: Minimum lipid layer thickness in nm recorded for a given video frame. |
| | C-Factor: Conformance factor is the ratio of image pixels that fall on the interferometric color spectrum. C- |
| | factor of 1.0 indicates every tear film pixel throughout the entire video has found a close match to an interferometric color. |
| | St Dev: Standard deviation of the frame averages for lipid layer thickness. |
| | NOTE: Since most tear film images have an average thickness well below 100, the maximum thickness values |
| | displayed are 100 with values above 100 represented as "100+". |
| 5 | Partial Blinks Count - Presented as a fraction with the number of partial blinks (numerator) over the number of |
| | total blinks (denominator). In this OD example, 1 partial blink/9 total blinks. |
| 6 | Graphical Analysis: |
| | <ul> <li>Blue line shows average lipid layer thickness values over video sampling time.</li> </ul> |
| | <ul> <li>Partial Blink Eye icon represents video frame where partial blink occurred.</li> </ul> |
| 7 | Select View Mode: Press to toggle between Full Eye View (Eyeball icon), Isolated Tear Film View (Tiled icon), |
| | Blinking Frames Only View (Closed Eye icon) or Notes (Notepad icon). |
| 8 | Export Icon – Export saved images, video or report to external medium or print report |

012051-US Rev C © 2016 TearScience, Inc.


<sup>1</sup> Finis D, Pischel N, Schrader S, Geerling G. Evaluation of lipid layer thickness measurement of the tear film as a diagnostic tool for Meibomian gland dysfunction. Cornea. 2013; 32(12):1549-53.

The first images, labeled as "Example" on the Capture/View screen (Figure 13), are standard reference video images of eyes with different lipid layer thickness values, provided for purposes of comparison. These videos allow the physician to observe differences in interference colors for a variety of tear films. As shown in Figure 18, the thin lipid example image is an example of an average tear film lipid layer thickness of 39 nm, which is relatively thinner lipid layer with very little color appearing mostly gray. Conversely, the thick lipid example image (Figure 19) is an example of an average tear film lipid layer thickness above 100, where brown and blue colors are visible indicating a relatively thicker lipid layer.



Figure 18. Example OD Image - Average Lipid Layer Thickness 39 nm



Figure 19. Example OS Image – Average Lipid Layer Thickness 100+ nm

012051-US Rev C © 2016 TearScience, Inc.


# 3.7 Capture Gland Images (Gland Imaging Mode)

**NOTE:** One person can both evert the lids and operate the device, using the pushbutton controls on the top panel with an external monitor positioned behind the patient where the operator can easily see it. Alternatively, imaging the meibomian glands can be easier to perform as a two-person procedure: one person everting the eyelids, and one person operating and focusing LipiView II.

- 1. To image the meibomian glands, select Gland Imaging from the Capture/View screen (Figure 13) and press *New*.
- 2. **Turn the room lights off** (or down sharply) prior to imaging to ensure good contrast in the image quality.
- 3. Disinfect the forehead and chin rest and Handheld Near IR Lid Everter with alcohol prior to use. Inspect Handheld Near IR Lid Everter to ensure it is intact prior to use.
- 4. Ensure the chin rest is in the extended position away from the device (closer to the patient).
- 5. Place the patient's chin fully forward into chin rest and forehead firmly against forehead rest. Adjust the height of the chin rest by spinning the fluted roller until the temporal canthus is aligned with the marks on the left and right sides of the forehead rest.
- 6. Select the upper or lower eyelid of the OD (right eye) or OS (left eye) to image by touching the magnify view icon in the applicable quadrant on Gland Image Capture screen (Figure 22). (You may also use the buttons on the keypad.)
- 7. Carefully evert the eyelid and ensure that the full extent of the meibomian glands is visible over the entire nasal to temporal length of the eyelid.
  - a. Evert entire length of lower eyelid: place Handheld Near IR Lid Everter (Figure 20) slightly below lash line; while maintaining contact, pull the lid down and then roll instrument slightly inward and upward.
  - b. Evert upper lid at the top of the tarsal plate: use a cotton swab, finger or other handheld instrument (Figure 21). Ensure the fingertip or cotton swab is not blocking the inner surface of the eyelid before capturing the image.

012051-US Rev C © 2016 TearScience, Inc.








Figure 21. Everting Upper Eyelid using Cotton Swab

Figure 20. Everting Lower Eyelid using Handheld Near IR Lid Everter

- 8. Position the camera using onscreen or pushbutton controls (Figure 23) on top of the unit to center the image of the everted eyelid on the screen. Alternatively, when using the touchscreen, touch the desired location to center the image on the screen and the device will automatically center the image in that location.
- 9. Press the autofocus reticle to focus the image using onscreen or pushbutton controls. If needed, press fine focus onscreen controls until the image is clear. (The F3 and F4 buttons on the keypad can also be used for fine focus.)

NOTE: Ensure full extent of the glands is visible over entire nasal to temporal length of the eyelid. When imaging lower eyelid, toggle between **Reflected IR** and **Trans IR** views (Figure 24) to ensure both views are of good image quality.

- 10. Press Capture button using onscreen or pushbutton controls to capture image.
- 11. Review gland image to ensure good image quality, including in both Reflected IR and Trans IR views for lower lid images (as shown in Figure 24). If the image is suboptimal (e.g., blurred focus, poor centration, only a partial lid eversion, finger obscuring view, washed out), delete image by selecting the Trashcan icon and recapture the image. Press *Notes* to add any notes to images, if desired.
- 12. Repeat steps 6 to 11 to capture the remaining images of other eyelid locations until all four eyelid images (i.e., upper and lower eyelid of the right and left eyes) are captured for the patient, if desired.
- 13. Press Analyze to save the image(s).

NOTE: PRESSING ANALYZE IS REQUIRED TO SAVE ALL IMAGES.

If *Analyze* is not pressed before exiting the imaging screen, a message will appear as a reminder to save the images.

012051-US Rev C © 2016 TearScience, Inc.




Figure 22. Gland Image Capture Screen with Labeled Controls

| | Key |
|---|---|
| 1 | Autofocus Reticle - Press the reticle to automatically focus the image |
| 2 | Select Position/Focus Button - Press to toggle display of manual focusing and positioning |
| | button controls on or off |
| 3 | Camera Button – Press to capture still image |
| 4 | Magnify View Icon - OD (right eye) lower lid is currently in view |
| | Touch to image OD (right eye) upper lid. |
| 5 | Magnify View Icon - Touch to image OS (left eye) upper lid |
| 6 | Magnify View Icon - Touch to image OS (left eye) lower lid |
| 7 | Light Source - Toggle between Reflected IR and Trans IR illumination views to image |
| | lower lid. Only Reflected IR illumination is used for upper lid. |
| 8 | Review Image Mode - Preview Captured Reflected IR, Trans IR and Merged images (after |
| | image capture, these small windows are populated with thumbnails of the different images) |
| 9 | Analyze Button – Press to save captured imagery |
| 10 | Notes Button - Press to open notes field for text entry |
| 11 | Manual Fine Focus Buttons - Press plus or minus to focus image |
| 12 | Manual Positioning Buttons - Press to move camera left, right, up or down |

012051-US Rev C © 2016 TearScience, Inc.


## Gland Image Modes:

- Reflected IR view is shown for both upper and lower eyelid gland images.
- Trans (Transillumination) IR view is shown only for lower eyelid gland images, if images were captured using Handheld Near IR Lid Everter.
- Merged view is the combination of the Reflected IR and Trans IR views and is shown only for the lower eyelid gland images.



Figure 23. Pushbutton Controls (on top of unit)

| | Key |
|---|---|
| 1 | Function Keys |
| | F1: In pre-capture view, toggles between Reflected IR and Trans IR mode |
| | F2: In post-capture review, changes view mode to captured Reflected IR image |
| | F3: In pre-capture mode, focuses in; post-capture review, changes view mode to captured |
| | Trans IR image |
| | F4: In pre-capture mode, focuses out; In post-capture review, changes view mode to |
| | captured Merged image |
| 2 | Select Eye/Lid - OD for right eye or OS for left eye and upper or lower lid |
| 3 | Position/Autofocus Buttons - Press up, down, right and left buttons to center on the |
| | desired lid. Tap to move in small increments or hold button down to move until released. |
| | Once lid is positioned, press reticle to autofocus. |
| 4 | Camera Button – Press to capture an image |





**OD Lower, Reflected IR View** 

OS Lower, Reflected IR View







**OS Lower, Trans IR View** 

Figure 24. Properly Focused Lower Lid Images: Reflected IR and Trans IR

# 3.8 Review Gland Images (Gland Imaging Mode)

- 1. To review prior gland images for an existing patient:
  - a. Select the patient from the Patient Records screen (Figure 11).
  - b. On the Capture/View screen (Figure 13), select Gland Imaging to view prior gland images or select All Exams to view all prior images.
  - c. A list of prior images is shown on the Capture/View screen (Figure 13). Drag and drop the desired images from the list to the sides of the screen marked "Drop Here". Touch the image again to display the Review Gland Images screen (Figure 27).
- 2. If desired, press the Export icon at the bottom of the Review Gland Images screen (Labeled 4 in Figure 27) to export or print images or report.
- 3. From the Export dialog (Figure 15), press the button to save images or report to an external medium or network, or print a report. Exported images can be displayed with or without patient demographics.

The first images, labeled as "Example" on the Capture/View screen (Figure 13), are standard reference images of upper and lower eyelids with different gland findings, provided for purposes of comparison. As shown in Figure 25, the image set labeled high dropout is an example of an eye with severely truncated meibomian glands. The image set labeled as medium dropout is an example of an eye with some evidence of gland loss. The image set labeled as no dropout is an

012051-US Rev C © 2016 TearScience, Inc.


example of an eye with no signs of gland loss. In Figure 26, the lower lid image labeled as dilation is an example of glands that appear dilated (enlarged), indicating a possible structural change or blockage.



**No Dropout** 

**Medium Dropout** 

**High Dropout** 

Figure 25. Gland Example Images: No Dropout, Medium Dropout, High Dropout



Figure 26. Gland Dilation Example, Lower Lid



Figure 27. Review Gland Images Screen with Labeled Controls

| | Key |
|---|---|
| 1 | Full Screen Mode - Press to view screen in full screen mode |
| 2 | Image Details - Timestamp date of image collection and Operator name |
| 3 | Select View Mode: Press to toggle between views; |
| | Reflected IR view (Light from above icon) |
| | Trans IR view (Light from below icon) – only displayed for lower lid images |
| | captured using Handheld Near IR Lid Everter |
| | Merged view (Lower Eyelid icon) – only displayed for lower lid images captured |
| | using Handheld Near IR Lid Everter |
| | Notes (Notepad icon) |
| 4 | Export Icon – Export saved images or report to external medium or print report |

# 3.9 Capture Ocular Images (Ocular Imaging Mode)

In Ocular Imaging mode, high-resolution images of the surface of the eye or the eyelids can be taken. White-light illumination may be switched on or off.

- 1. To image the ocular surface or eyelids, select Ocular Imaging from the Capture/View screen (Figure 13) and press *New*.
- 2. Disinfect the forehead and chin rest with alcohol prior to use.
- 3. Ensure the chin rest is in the extended position away from the device.
- 4. Place the patient's chin fully forward into chin rest and forehead firmly against forehead rest. Adjust the height of the chin rest by spinning the fluted roller until the temporal canthus is aligned with the marks on the left and right sides of the forehead rest. Instruct the patient to look at the orange fixation light.

CAUTION: To prevent pinching, do not put fingers near illuminator, lens or chin rest during focusing. Instruct patient not to place hands on LipiView II during operation, and not to put fingers near illuminator, lens or chin rest.

- 5. Select OD (right eye) or OS (left eye) to image by touching the right or left side of the Ocular Image Capture screen (Figure 28).
- 6. Select to turn white light illumination on, or turn off to capture images using room illumination only.
- 7. Position the camera by touching the desired location to be imaged on screen, which will automatically move the camera and center on the location. Press the position keys, as needed, until the location appears in the center of the screen.
- 8. Press the reticle to autofocus, or press the fine focus buttons to adjust the focus until the image is clear.
- 9. Press *Camera* icon to capture a still image. Press *Capture Video* button to begin recording approximately 5 seconds of video. The blinking red light indicates LipiView II is recording video. Press *Capture Video* button again to stop recording prior to 5 seconds, if desired. You can capture up to 10 still images and one video per eye.
- 10. When recording is complete, the illuminator turns off (if white illumination was turned on during imaging). Press *Notes* to add any notes to images, if desired.
- 11. Review still image or video using onscreen playback button. If image quality is suboptimal, delete image using Trashcan icon and recapture another image.
- 12. Repeat steps 5 to 11 to capture an image of the other eye, if desired.
- 13. Press *Save* to save the video or image(s).

012051-US Rev C © 2016 TearScience, Inc.




Figure 28. Ocular Image Capture Screen with Labeled Controls

| | Key |
|---|---|
| 1 | Eye Position Indicator - Indicates the eye being imaged (OD in figure) |
| 2 | Magnify View Icon - OD (right eye) is currently in view. OS (left eye) side is currently |
| | greyed out. Touch icon to capture images for OS (left eye). |
| 3 | Capture Video Button - Press to begin recording. Appears as a rectangle during |
| | recording; press rectangle to stop recording before 10 seconds. |
| 4 | Camera Button – Press to capture still image |
| 5 | Full Screen Mode – Press to view screen in full screen mode |
| 6 | Manual Positioning Buttons - Press to move camera left, right, up or down |
| 7 | Manual Fine Focus Buttons - Press plus or minus to focus image |
| 8 | Autofocus Reticle - Press the reticle to automatically focus the image |
| 9 | Save Button – Press to save captured imagery |
| 10 | Notes Button - Press to open notes field for text entry |
| 11 | White Light Illumination – Press to toggle illuminator on or off |

# 3.10 Review Ocular Images (Ocular Imaging Mode)

- 1. To review prior ocular images or video for an existing patient:
  - a. Select the patient from the Patient Records screen (Figure 11).
  - b. On the Capture/View screen (Figure 13), select Ocular Imaging to view prior ocular images or select All Exams to view all prior images.
  - c. A list of prior images is shown on the Capture/View screen (Figure 13). Drag and drop the desired images from the list to the sides of the screen marked "Drop Here". Touch the image again to display the Review Ocular Images screen (Figure 29).
- 2. If desired, press the Export icon on the Review Ocular Images screen (Labeled 6 in Figure 29) to export or print images or report.
- 3. From the Export dialog save, (Figure 15), press the icon to save images, video or report to an external medium or network, or print a report. Exported images can be displayed with or without patient demographics.





Figure 29. Review Ocular Images with Labeled Controls

| Key | |
|---|---|
| 1 | Video Playback Controls - Press to play, pause, forward step, reverse step (for captured video only) |
| 2 | Full Screen Mode – Press to view screen in full screen mode |
| 3 | Video Preview |
| 4 | Image Preview |
| 5 | Notes Button - Press to open and view notes field for text entry |
| 6 | Export Icon – Export saved images, video or report to external medium or print report |

012051-US Rev C © 2016 TearScience, Inc.


# 3.11 Log Out and Power Off

Press the Log Out tab (Labeled 4 in Figure 10) on the menu bar to log out when the device is not is use.

Power off LipiView II overnight to allow the device to cool down. The device does not need to be powered off between patient examinations during the day.

#### **Troubleshooting Guide** 4

Table 6 lists the troubleshooting actions for Unexpected Events. For technical support, contact TearScience in North America at +1 919 459 4891 or by email at customerservice@tearscience.com.

**Table 6: Troubleshooting Unexpected Events** 

| Event | Action to Take |
|---|---|
| Device will not power up | Ensure device is connected to a power outlet and the |
| (after pressing the power | connection into the device is secure, then press the power |
| switch, the screen remains | switch again. |
| dark) | If the problem persists, contact TearScience. |
| Problem reported during Power | Turn the device off then on again. |
| On Self Test (POST) | If the problem persists, contact TearScience. |
| Touch Screen does not | Turn the device off then on again. |
| respond | If the problem persists, contact TearScience. |
| Illuminator does not light | Turn the device off then on again. |
| during lipid image capture | If the problem persists, contact TearScience. |
| Camera stops working | Turn the device off then on again. |
| <u> </u> | If the problem persists contact TearScience |
| Disk Space Indicator shows | Contact the Administrator to archive data. |
| internal disk drive is full | If the problem persists, contact TearScience. |
| The system works except the | An error was detected during power on self-test, which affects |
| Capture screen will not | image acquisition. Turn the device off then on again. |
| respond (for Lipid, Gland, or | If the error persists, contact TearScience. |
| Ocular Imaging) | |
| Device will not process images | The internal hard drive is full. Contact the site Administrator |
| after acquisition | to archive data. |
| | If the problem persists, contact TearScience. |
| Device no longer allows image | A power on self-test problem has been found. |
| acquisition | If the problem persists, contact TearScience. |
| The Review Lipid Images | The patient's head may not have been pushed forward, the |
| screen does not display a | patient's forehead may not have been firmly pressed against |
| numerical lipid layer thickness | the forehead rest, or the tear film image may have been out of |
| value | focus. Collect another video of the patient after ensuring that |
| | the patient's head is positioned properly and that the image is |
| | clearly focused. |
| Network is not connected | Contact the Administrator. |
| | If the problem persists, call TearScience. |

CR-5969 v3 0

| Event | Action to Take |
|---|---|
| External monitor does not | Ensure the monitor is powered on before LipiView II. Ensure |
| work | connections to the DVI or HDMI are made, and proper video |
| | input is selected. Ensure the Administrator has activated and |
| | properly configured the monitor on the Computer Info screen |
| | in the Admin interface. |
| Administrator forgets | Contact TearScience. |
| password after resetting it | |
| When accessing options on the | Selected options on the System Information Administration |
| System Information | screen cannot be accessed after more than 10 minutes has |
| Administration screen, this | elapsed since the system was started. Turn the device off then |
| message displays: "Too much | on again. |
| time has elapsed since system | Then, attempt to access the option again on the System |
| startup to access this function" | Information Administration screen. |
| When accessing the | The system's disk drive usage is beyond the level specified in |
| Capture/View screen, a message | the Networking/Backup Administration screen. Contact the |
| displays stating disk space usage | Administrator to perform a system backup. |
| has surpassed the warning level | |
| When accessing the | The system's disk drive usage is beyond the maximum level |
| Capture/View screen, a | specified by TearScience. Contact the Administrator to |
| message displays stating disk | perform a system backup. Video capture is disabled until |
| space usage has surpassed the | system backup is performed. |
| critical level | |

Table 7 describes the Operational System Messages categorized by type as: "E" for Error Message; "C" for User Confirmation Message; and "I" for Information Message Requiring User Attention. For a list of system messages related to System Administrative functions, refer to LipiView II Administrator's Guide.

System messages are generated when something unexpected occurs, when the user attempts to perform an invalid operation, or to confirm completion of an event. These messages may instruct the user on a particular action to take (e.g., enter a missing field, or correct the format of a date field). When a system message is displayed, it requires a response from the user by pressing a button (e.g., Close or OK) on the message before any other input from the screen is accepted. System messages related to Windows error codes will also be listed in the System Log.

Table 7. Operational System Messages and Descriptions

| ID | Type | Displayed Text | Description |
|---|---|---|---|
| 1 | E | You must enter a user name and password. | Displayed on Login screen if operator touches Login button without entering a username or a password |
| 2 | E | Invalid user name or password. | Displayed on Login screen if operator enters and invalid username and/or password and attempts to login to the system. |
| 3 | E | An internal system error was | Displayed on Login screen if the system database is corrupt |

012051-US Rev C © 2016 TearScience, Inc.


| m | Type | Displayed Text | Description |
|---|---|---|---|
| | | encountered when attempting to log | and the system is unable to log an operator into the system. |
| | | operator into system. Consult the | Service call or remote support is required to fix. |
| | | system log for details. | 11 1 |
| 4 | E | An internal system error was | Displayed on Patient Records screen if the system database is |
| | | encountered when attempting to access | corrupt and the system is unable to obtain a list of patients. |
| | | the patient list. Consult the system log | Service call or remote support is required to fix. |
| | | for details. | |
| 5 | Ι | Ensure patient and operator are clear of | Displayed on Warning Screen during the system power-on |
| | | the chinrest area. The unit will now | self-test before the system performs initialization. |
| | | automatically home the motor system. | |
| | | Press the OK button to begin. | |
| 6 | E | An error was encountered obtaining the | Displayed on Networking Administrator screen if the system |
| | | list of network adapters. Consult the | is unable to obtain a list of network adapters from the |
| | | system log for details. | operating system. Service call or remote support is required to |
| | | | fix. |
| 7 | E | An error was encountered obtaining the | Displayed on Networking Administrator screen if the system |
| | | status of a network adapter. Consult the | is unable to obtain the status of the network adapters from the |
| | | system log for details. | operating system. Service call or remote support is required to fix. |
| 8 | E | Image capture functionality has been | Displayed on Capture Screen if a system error has prevented |
| ľI | L | disabled due to a system error. Consult | new images from being captured. Reboot the system to see if |
| | | the system log for details. | the error clears. If the error does not clear, service call or report |
| | | the system log for details. | support is required. |
| 9 | E | The Capture screen is not configured | Displayed on Capture screen if the system database is corrupt |
| | ~ | correctly. Contact TearScience for | and the Capture screen cannot reads its configuration. Service |
| | | technical support. | call or remote support is required to fix. |
| 10 | E | Unable to set up the system for image | Displayed on Capture screen if an error was encountered from |
| | | capture. Consult the system log for | the system hardware while attempting to configure the system |
| | | details. | to capture images. Try to enter the Capture screen again to see |
| | | | if the error clears. If the error does not clear, a service call or |
| | | | remote support is required to fix. |
| 11 | E | The live video stream from the camera | Displayed on Capture screen if an error was encountered from |
| | | has been interrupted. Please exit the | the camera during live video streaming. Try to enter the |
| | | Capture screen and try again. Consult | Capture screen again to see if the error clears. If the error does |
| | | the system log for details. | not clear, a service call or remote support is required to fix. |
| 12 | E | A motion control error was | Displayed on Capture screen if an error was encountered |
| | | encountered. Consult the system log for | trying to move a motion control axis. Try to enter the Capture |
| | | details. | screen again to see if the error clears. If the error does not clear, |
| | | | a service call or remote support is required to fix. |
| 13 | E | An error was encountered during video | Displayed on Capture screen if an error was encountered |
| | | capture. Consult the system log for | during video capture. Try to enter the Capture screen again to |
| | | details. | see if the error clears. If the error does not clear, a service call or |
| 1.4 | E | The perions of data of the territory | remote support is required to fix. |
| 14 | E | The patient's date of birth is invalid.<br>Please enter a valid date of birth. | Displayed on Patient Records screen if a patient is added or |
| 15 | E | A first name must be entered for the | edited and an invalid date of birth in entered for the patient. |
| 13 | E | _ | Displayed on Patient Records screen if a patient is added or |
| | | patient. | edited and the first name is omitted without a patient ID having been entered. |
| 16 | E | A last name must be entered for the | Displayed on Patient Records screen if a patient is added or |
| 10 | ند | patient. | edited and the last name is omitted without a patient ID |
| | | parient | having been entered. |
| | | | Having Occil circicu. |

012051-US Rev C © 2016 TearScience, Inc.


| 110 | Type | Displayed Text | Description |
|---|---|---|---|
| 17 | E | A first and last name plus a date of | Displayed on Patient Records screen if a patient is added or |
| | | birth, OR a Patient ID, must be entered | edited and the patient ID is omitted. |
| | | for the patient. | · |
| 18 | E | The entered Patient ID already exists | Displayed on Patient Records screen if a patient ID is entered |
| | | for another patient. | for a patient and the patient ID is already used by another |
| | | •. | patient in the system. |
| 19 | E | An internal system error was | Displayed on Patient Records screen if a system database error |
| | | encountered when attempting to add | prevented system from adding a new patient. Service call or |
| | | the patient to the system. Consult the | remote support is required to fix. |
| | | system log for details. | |
| 20 | E | An internal system error was | Displayed on Patient Records screen if a system database error |
| | | encountered when attempting to | prevented the system from editing an existing patient. Service |
| | | update the patient demographics. | call or remote support is required to fix. |
| | | Consult the system log for details. | |
| 21 | E | An internal system error was | Displayed on Capture screen if the system is unable to perform |
| | | encountered when attempting to | an analysis when the Analyze button is pressed on the Capture |
| | | perform the analysis. Consult the | screen. Service call or remote support is required to fix. |
| | | system log for details. | |
| 22 | С | No data has been collected for either | Displayed on Capture screen if the operator pressed the |
| | | eye. Are you sure you wish to exit the | Analyze/Save button without having collected any data on the |
| | | Capture screen?" | capture screen. |
| 23 | С | Data has been collected for only one | Displayed on Capture screen if the operator pressed the |
| | | eye. Are you sure you wish to exit and | Analyze/Save button and has only collected data for one eye. |
| | | analyze? | |
| 24 | С | Are you sure you wish to discard the | Displayed on Capture screen if the operator clicked the Trash |
| | | collected video? | button in an attempt to discard the collected video. |
| 25 | С | Are you sure you wish to discard the | Displayed on Capture screen if the operator clicked the Trash |
| | | collected image? | button in an attempt to discard a collected still frame image. |
| 26 | E | The View Analysis screen is not | Displayed on View Analysis screen if it is unable to display the |
| | | configured correctly. Contact | View Analysis sub-screen for a modality. Service call or remote |
| | | TearScience for technical support. | support is required to fix. |
| 27 | E | An internal system error was | An internal system error was encountered during the |
| | | encountered processing the data | processing of an analysis. Service call or remote support is |
| | | analysis. Consult the system log for | required to fix. |
| | - | details. | |
| 28 | E | An internal system error was | An internal system error was encountered attempting to load |
| | | encountered loading the analysis data. | analysis data from disk into memory for display. Service call or |
| | T | Consult the system log for details. | remote support is required to fix. |
| 29 | E | The data storage disk space used has | Displayed on Capture screen when the data disk used space is |
| | | reached a critical level. Please perform a | greater than 95%. Further image capture has been disabled. |
| | | data archival operation. Image capture | Site administrator must either perform a system backup or |
| | | has been disabled until this problem is | delete some imaging sessions to gain free space. |
| 20 | T | resolved. | Dial de Control de la |
| 30 | I | The data storage disk space usage is | Displayed on Capture screen when the data disk used space is |
| | | above the warning threshold. Please | above the warning threshold specified in the Backup/Restore |
| | | perform a data archival operation when | Administration screen (default 75%). This message is to |
| | | convenient. | remind the operator to perform a backup in the near future. |

| ID. | Туре | Displayed Text | Description |
|---|---|---|---|
| 37 | С | There is unsaved data collected on the | Displayed on Capture Screen if the operator attempts to exit |
| | | Capture Screen and the requested | the Capture screen with unsaved/unanalyzed data present. |
| | | operation will discard this data. Are you | |
| | | sure you wish to proceed? | |
| 38 | E | The operating system encountered an | Displayed when the Destination Drive list dialog is displayed |
| | | error obtaining a list of drives on the | but the system in unable to get a list of removable/networked |
| | | system. Consult the system log for | drives from the operating system. Service call or remote |
| | | details. | support is required. |
| 39 | С | Please select one or more destinations | Displayed on the Destination Drive list dialog is displayed |
| | | for the output: | informing the operator of the intent of the drive list. |
| 40 | E | The output file '%1' is unable to be | The system attempted to output a file of some type (e.g. video |
| ll | | opened. The operating system error | or still image) to an external USB or network drive and was |
| | | code is '%2'. | unable to write the file. Check health and status of the storage |
| | | | location and try again. |
| 44 | I | No available drives are detected on the | Displayed by the Destination Drive dialog to inform the |
| | | system. | operator the system did not detect any external storage |
| | | | locations (either USB or networked). |
| 54 | E | An internal error was encountered | The operator attempted to access the Notes Editor screen but |
| | | accessing the notes database. Please | a system internal error prevented the notes data from being |
| | | contact TearScience for technical | accessed. Service call or remote is support required to fix. |
| | | support. | |
| 55 | С | Are you sure you wish to delete the | The operator has clicked the Delete Note icon and this |
| | | selected note? | message asks the operator to confirm the deletion. |
| 56 | С | Note information exists that has not | The operator has entered text into a new note but has not |
| | | been saved. Are you sure you wish to | clicked the Save Note button and is attempting to exit the |
| | | exit without saving the information? | Notes screen. |
| 60 | С | Please select the destination drive(s) for | The operator clicked the Export Images button on the Export |
| | | the exported images: | Screen and this message appears on the Destination Drive |
| | | | selection dialog to inform the operator of the function of the |
| - | | | drive selection dialog. |
| 62 | E | An error was encountered producing | An internal system error occurred while producing export |
| | | the requested output. Please check the | images or videos. Check the system log for more details. |
| | | system log for details. | Service call or remote support is likely required. |
| 63 | E | An error was encountered producing | An error occurred with an external storage location in |
| | | the requested output. The error | attempting to export images or videos to the storage location. |
| | | information from the operating system | Evaluate the error information given and resolve the problem. |
| | | is '%1' (%2). | Examples of problems would be insufficient disk space to store |
| - | | | the output, etc. |
| 64 | E | An error was encountered attempting | An error occurred attempting to load a web page in the |
| | | to load the web page. The error | internal web browser (e.g. the Remote Support login screen). |
| | | information is '%2' (Code: %3). | Attempt to access the page and ensure connectivity to the |
| 7/ | | Discoulated at the 12 (12 C | Internet. |
| 76 | С | Please select the destination drive(s) for | Displayed on Destination Drive selection dialog to prompt |
| 02 | -c | the exported videos: | user to select destination for exported videos. |
| 96 | ١ | Data has not been collected for all eye | Displayed on the Gland Image Capture screen if the operator |
| | | and lid combinations. Are you sure you | has not collected image for both lids on both eyes. |
| 100 | | wish to exit the Capture screen? | Did I d Die Gleich field |
| 109 | С | Please select the destination printer for | Displayed on the Printer Selection list when the operator |
| 110 | | the report: | chooses the Print Report feature from the Export screen. |
| 110 | Е | The operating system encountered an | The system was unable to get a list of printers from the |
| | | error obtaining a list of printers. | operating system. Turn the device off then on again, and try to |

012051-US Rev C © 2016 TearScience, Inc.


| 10 | Туре | Displayed Text | Description |
|---|---|---|---|
| | | Consult the system log for details. | print the report again. |
| 111 | I | Video Data File Not Found On System | Displayed in the video pane of an analysis view screen if the source video file could not be located on the system or attached external storage. |
| 112 | Ī | Image Data File Not Found On System | Displayed in the still frame pane of an analysis view screen if the source image file could not be located on the system or attached storage. |
| 113 | С | Please select the destination drive for the PDF: | Displayed on the Drive Select list dialog after the operator has chosen to Save a PDF file of the report by touching the Save PDF button from the Export screen. |
| 114 | I | No printers are installed on the system | Displayed on the Printer Selection list dialog when no printers are installed on the system. Install a printer before attempting to print. |
| 125 | I | The entered password is not correct. | Displayed where an operator is required to enter a password and enters an incorrect password. |
| 127 | I | Please check the position of the chinrest and ensure it is in the rear position. | Displayed when the chinrest is not in the correct position for imaging. |
| 128 | I | The maximum number of images has been captured. To capture additional images, delete one or more of the existing images. | Displayed on the Ocular Image Capture screen when the operator has captured the maximum number of still images and then attempts to capture another. |

# **Appendix: Electromagnetic Compatibility** Requirements

Table 8: Guidance and Manufacturers Declaration-Electromagnetic Emissions

| LipiView II is intended for use in the electromagnetic environment specified below. The customer | | |
|---|---|---|
| or the user of LipiView II should assure that it is used in such an environment. | | |
| Emissions Test Compliance Electromagnetic Environment-Guidance | | |
| RF emissions CISPR 11 | Group 1 | LipiView II uses RF energy only for its internal function. Therefore, its RF emissions are very low and are not likely to cause any interference in nearby electronic equipment. |
| RF emissions<br>CISPR 11 | Class A | NA |
| Harmonic emissions IEC 61000-3-2 | Class A | NA |
| Voltage fluctuations Flicker emissions IEC 61000-3-3 | Complies | LipiView II is suitable for use in all establishments other than domestic and those directly connected to the public low-voltage power supply network that supplies buildings for domestic purposes. |

CR-5969 v3 0

Table 9: Guidance and Manufacturers Declaration-Electromagnetic Immunity (part 1)

LipiView II is intended for use in the electromagnetic environment specified below. The customer or the user of LipiView II should assure that it is used in such an environment. Immunity Test IEC 60601 **Compliance Level Electromagnetic Environment-**Test Level Guidance Electrostatic +6 kV contact ±6 kV contact Floors should be wood, concrete or discharge (ESD) ±8 kV air ±8 kV air ceramic tile. If floors are covered with IEC 61000-4-2 synthetic material, the relative humidity should be at least 30% Electrical fast ±2 kV for power ±2 kV for power Mains power quality should be that of a supply lines supply lines transient/burst typical commercial or hospital IEC 61000-4-4 ±1 kV for ±1 kV for environment input/output input/output lines lines ±1 kV +1 kV differential Surge Mains power quality should be that of a IEC 61000-4-5 differential mode typical commercial or hospital mode ±2 kV common environment. ±2 kV common mode mode Voltage dips, short <5 % U<sub>T</sub> <5 % U<sub>T</sub> Mains power quality should be that of a (>95 % dip in interruptions and (>95 % dip in U<sub>T</sub> for typical commercial or hospital voltage variations U<sub>T</sub> for 0,5 cycle 0,5 cycle environment. If the user of the on power supply 40 % U<sub>T</sub> 40 % U<sub>T</sub> equipment requires continued operation (60 % dip in U<sub>T</sub>) input lines  $(60 \% \text{ dip in } U_T)$ during power mains interruptions, it is IEC 61000-4-11 recommended that the equipment be for 5 cycles for 5 cycles powered from an uninterruptible power 70% U<sub>T</sub> 70% U<sub>T</sub> supply or a battery.  $(30\% \text{ dip in } U_T)$  $(30\% \text{ dip in } U_T)$ for 25 cycles for 25 cycles <5% U<sub>T</sub> <5% U<sub>T</sub> (>95 % dip in (>95 % dip in U<sub>T</sub>)  $U_{\rm T}$ ) for 5 sec for 5 sec Power frequency 3 A/m 3 A/m Power frequency magnetic fields should (50/60 Hz)be at levels characteristic of a typical magnetic field location in a typical commercial or IEC 61000-4-8 hospital environment. \*NOTE:  $U_T$  is the a.c. mains voltage prior to application of the test level.

Table 10: Guidance and Manufacturers Declaration-Electromagnetic Immunity (part 2)

LipiView II is intended for use in the electromagnetic environment specified below. The customer or the user of LipiView II should assure that it is used in such an environment.

| Immunity Test | IEC 60601 Test | Compliance | Electromagnetic Environment-Guidance |
|---|---|---|---|
| | Level | Level | |
| | | | Portable and mobile RF communications equipment should be used no closer to any part of the LipiView II, including cables, than the recommended separation distance calculated from the equation applicable to the frequency of the transmitter. |
| | | | Recommended Separation Distance |
| Conducted RF<br>IEC 61000-4-6 | 3 Vrms<br>150 kHz to 80<br>MHz | 10 V | $d = [3.5/V1]\sqrt{P}$ $d = [3.5/E1]\sqrt{P} 80MHz to 800MHz$ $d = [7.0/E1]\sqrt{P} 800MHz to 2.5GHz$ |
| Conducted RF<br>IEC 61000-4-3 | 3 Vrms<br>80 MHz to 2,5<br>GHz | 3 V/m | Where P is the maximum output power rating of the transmitter in watts (W) according to the transmitter manufacturer and d is the recommended separation distance in meters (m). Field strengths from fixed RF transmitters, are determined by an electromagnetic site survey, a should be less than the compliance level in each frequency range. Interference may occur in the vicinity of equipment marked with the following symbol: |
| | | | (( <u>(</u> )) |

NOTE 1 At 80 MHz and 800 MHz, the higher frequency range applies.

NOTE 2 These guidelines may not apply in all situations. Electromagnetic propagation is affected by absorption and reflection from structures, objects and people.

<sup>&</sup>lt;sup>a</sup> Field strengths from fixed transmitters, such as base stations for radio (cellular/cordless) telephones and land mobile radios, amateur radio, AM and FM radio broadcast and TV broadcast cannot be predicted theoretically with accuracy. To assess the electromagnetic environment due to fixed RF transmitters, an electromagnetic site survey should be considered. If the measured field strength in the location in which the LipiView II is used exceeds the applicable RF compliance level above, the LipiView II should be observed to verify normal operation. If abnormal performance is observed, additional measures may be necessary, such as re-orienting or relocating the LipiView II.

<sup>&</sup>lt;sup>b</sup> Over the frequency range 150 kHz to 80 MHz, field strengths should be less than 3 V/m.

## Table 11: Recommended Separation Distances Between Portable and Mobile RF Communications Equipment and LipiView II

LipiView II is intended for use in an electromagnetic environment in which radiated RF disturbances are controlled. The customer or the user of LipiView II can help prevent electromagnetic interference by maintaining a minimum distance between portable and mobile RF communications equipment (transmitters) and LipiView II as recommended below, according to the maximum output power of the communications equipment.

| | Separation distance according to frequency of transmitter | | |
|---|---|---|---|
| Rated maximum<br>output power of<br>transmitter<br>W | 150 kHz to 80 MHz<br>d=[3.5/V₁]√P | 80 MHz to 800 MHz $d=[3.5/E_1]\sqrt{P}$ | 800 MHz to 2,5<br>GHz<br>d=[7/E <sub>1</sub> ]√P |
| 0,01 | 0.12 | 0.12 | 0.23 |
| 0,1 | 0.37 | 0.37 | 0.74 |
| 1 | 1.2 | 1.2 | 2.3 |
| 10 | 3.7 | 3.7 | 7.4 |
| 100 | 12 | 12 | 23 |

For transmitters rated at a maximum output power not listed above, the recommended separation distance d in meters (m) can be estimated using the equation applicable to the frequency of the transmitter, where P is the maximum output power rating of the transmitter in watts (W) according to the transmitter manufacturer.

NOTE 1 At 80 MHz and 800 MHz, the separation distance for the higher frequency range applies.

NOTE 2 These guidelines may not apply in all situations. Electromagnetic propagation is affected by absorption and reflection from structures, objects and people.



2012© Dr. Heiko Pult – Optometry & Vision Research, Germany www.heiko-pult.de Fig. 1.
Five-grade meiboscale [14].

## APPENDIX F: EVALUATION OF LID WIPER EPITHELIOPATHY (LWE)

#### **Procedure for Evaluation of LWE**

#### Materials:

Fluorescein sodium ophthalmic strips USP; each strip contains 1mg Fluorescein sodium USP.

#### Procedure:

- 1. Wet a fluorescein strip strip with sterile saline (2 drops).
- Wait for 3 seconds to ensure that fluorescein particles dissolve before applying the strip.
- 3. Ask subject to look down and apply strip onto the superior bulbar conjunctiva.
- 4. Sixty seconds later, apply a second strip of fluorescein by repeating steps 1, 2 and 3.
- 5. Wait 3 minutes before lid eversion and assessment of LWE.
- 6. While everting the lid be careful to avoid any trauma to the lid margin region.
- 7. Evaluate the upper lid margin with the slit-lamp
  - a) Blue Cobalt filter (light source)
  - b) Wratten No.12 yellow barrier filter
  - c) View at 12X magnification ensuring that almost the whole width (or as much as possible) is visible.
  - d) Grade horizontal length and sagittal width of staining using the scale below:
- 8. Evaluate the lower lid margin with the slit-lamp following the same procedure (7a-d)

| Grading: | | | |
|---|---|---|---|
| Horizontal length of staining | Grade | Sagittal width of staining | Grade |
| <2 mm | 0 | <25% of the width of wiper | 0 |
| 2-4 mm | 1 | 25% - <50% width of wiper | 1 |
| 5-9 mm | 2 | 50% - <75% width of wiper | 2 |
| >10 mm | 3 | ≥ 75% of the width of wiper | 3 |

#### Grading:

| Classification * | | | | |
|---|---|---|---|---|
| Final Grade [ (UL + LL)/2 ] | | | | |
| Average | | | | |
| Sagittal | _ | | _ | _ |
| Horizontal | _ | - | _ | _ |
| Area | Upper Lid (UL) | Lower Lid (LL) | Upper Lid (UL) | Lower Lid (LL) |
| | has a more a common money and a common management | | A CONSTRUCTION CONTRACTOR STOREST STOR | S |

\* Subjects will be classified according to their final LWE grade for each eye.

| Fin | al LWE Grade |
|-------------|--------------|
| 0 | None |
| 0.25 - 1.00 | Mild |
| 1.25 - 2.00 | Moderate |
| 2.25 3.00 | Severe |

#### APPENDIX G: LIPCOF GRADING SCALE

LIPCOF will be evaluated in the area perpendicular to the temporal and nasal limbus on the bulbar conjunctiva above the lower lid (temporal and nasal LIPCOF, respectively) with a slit-lamp microscope, and classified using the LIPCOF grading scale below.

A further combined LIPCOF score (LIPCOF Sum) will be calculated by adding together the nasal LIPCOF grade and temporal LIPCOF grade.

# EDUCATIONAL MOMENTS



**INSPIRING CARE** 

How to manage patients with Lid Parallel Conjunctival Folds (LIPCOF)

| | | 1 What You Need to Know | en e en | olen gyölken manna mann |
|---|---|---|---|---|
| lit Lamp Viewing: | | ) Medium magnification (16-27<br>perpendicular to temporal and | | |
| irading: | A combined score (LIPCO | OF Sum) can be calculated by a | dding nasal and temp | oral LIPCOF grades |
| t pp | | Grade 0: No conjunctival folds | | Grade 1: One permanent and |
| | | | | clear parallel fol |
| | 9. | Grade 2: Two | | Grade 3: More |
| | | permanent and clear parallel folds (normally | NA | than two<br>permanent and |
| | er egypte | <0.2mm) | | clear parallel<br>folds (normally<br>>0.2mm) |

| | LIPCOF |
|---------------------------------------------------|--------|
| | GRADE |
| NO CONJUNCTIVAL FOLDS | 0 |
| ONE PERMANENT AND CLEAR PARALLEL FOLD | 1 |
| TWO PERMANENT AND CLEAR PARALLEL FOLDS, | 2 |
| (NORMALLY LOWER THAN 0.2MM) | |
| More than two permanent and clear parallel folds, | 3 |
| (NORMALLY HIGHER THAN 0.2MM) | |
# APPENDIX H: MEIBOMIAN GLAND EVALUATOR MANUFACTURER INSTRUCTIONS

Procedure and directions for use of TearScience® Meibomian Gland Evaluator found in manufacture instruction in package insert (calculation of Total Meibomian Gland Secretion Score will be undertaken by Sponsor data management and need not be calculated by Clinical Study Site):

Melbomian Gland Evaluator Model MGE-1001 Package Insert - English

### Meibomian Gland Evaluator Device Description:

The Meibornian Gland Evaluator is a handheld instrument used by a physician to evaluate Meibornian gland secretions in adult patients during a routine eye examination. The instrument provides a standardized method to apply consistent, gentle pressure to the outer skin of the lower eyelid while visualizing the secretions from the Meibornian gland orifices through a sitt tamp biomicroscope. The pressure applied to the eyelid when using the device is between 0.8 g/mm² and 1.2 g/mm².

### Directions for Use:

Assess the Meibornian glands in the three regions under the eyelid: temporal, central and nasal. Approximately five glands are expressed per region with each use of the Meibornian Gland Evaluator.



Figure 1: Eyelid Gland Regions

### Melbomian Gland Evaluation - Step by Step:

- Prior to initial use of the Meibomlan Gland Evaluator, check for any rough surfaces that may come in contact with a patient's eyelid.
- Wash your hands and disinfect the Meibornian Gland Evaluator with alcohol prior to use on each patient.
- Under the slit lamp at 10x-16x magnification, locate the lower eyelid and gland regions. (Figure 1).

### Starting with the temporal region:

- Instruct the patient to look upwards. Avoid any contact of the instrument with the eye.
- Holding the Meibornian Gland Evaluator between your forefinger and the finumb, place the shaft to the skin immediately below the lash line of the lower eyelid so that the long dimension is paratlet to the eyelid margin.
- Once full contact is achieved between the contact surface and the outer surface of the lower eyelid, rotate the shaft of the instrument downward approximately 15 to 45 degrees so that the leading face is tangential to the eyeball.



Figure 2: Melbomian Gland Evaluator Placement

- Depress the shaft of the instrument mid-way (approximately 3mm) to exert a
  constant force on the meibornian glands. Adjust the position of the instrument to
  cause the flat surface of the lower eyelld margin to roll alightly outward for a clear
  view of the Meibornian gland orifices.
- To facilitate observation of the gland secretions, gently wipe clean the gland orifices along the eyelid margin with a cotton swab immediately after applying pressure and while holding the instrument in position and maintaining pressure.
- Hold the instrument in place over the Meibornian glands for approximately 10-15 seconds while evaluating the secretion characteristics from each Meibornian gland.
- 10. Assess 5 consecutive glands in the center of the Meibornian Gland Evaluator
- 11. Repeat steps 4-9 for the central and nasal regions. (Figure 1)
- 12. Refer to the Secretion grading scale below to grade secretions for each of the 5 glands selected within the three regions (temporal, central and nessif). Record the grades for a total of 15 glands on the patient's chart. Next, calculate the Total Meibornian Gland Secretion Score by adding the grades for the 15 glands assessed. Record this score on patient's chart.
- 13. Disinfect the instrument with alcohol after each use.

### Meibomian Gland Secretion Grading Scale:

| Grade | Secretion Quality |
|-------|-------------------------------------------------------|
| 3 | Clear Liquid Oil |
| 2 | Colored/Cloudy Liquid |
| 1 , | Inspissated (semi-solid, toothpaste-like consistency) |
| 0 | No Secretion (Includes capped orifices) |



Grade 3: Clear Llouid Oil



Grade 1: Inspissated



Grade 2: Colored/Cloudy Liquid Oil



Grade 0: No secretion

# Contraindications: No contraindications are known.

### **Precautions**

Do not depress the shaft to the endpoint of the spring. Do not apply any additional force after the shaft has been depressed approximately 6 mm. Applying additional force negates the benefit of using the instrument to apply a standard force. Familiarity with use of a six lamp biomicroscope is required to use Meibomian Gland Evaluator for assessment of the meibomian gland secretions.

### APPENDIX I: MEIBOMIAN GLAND SECRETION GRADING SCALE

### Melbomian Gland Secretion Grading Scale:

| Grade | Secretion Quality |
|-------|-------------------------------------------------------|
| 3 | Clear Liquid Oil |
| 2 | Colored/Cloudy Liquid |
| 1 . | Inspissated (semi-solid, toothpaste-like consistency) |
| 0 | No Secretion (Includes capped orifices) |

# Example

| | O.D. | O.D. | O.S. | |
|--------------------|------|------|------|---|
| Central Lower Lid | | | | |
| Temporal Lower Lid | | | | : |
| Nasal Lower Lid | | | | |

### APPENDIX J: CLINICAL TECHNICAL PROCEDURES (CTP)

Pre-Ocular and Pre-Lens Wettability

Limbal and Conjunctival (Bulbar) Redness

**Expanded Sodium Fluorescein Corneal Staining** 

**Lens Fitting Characteristics** 

Subject Reported Ocular Symptoms/Problems

Front and Back Surface Lens Deposit Grading Procedure

**Determination of Distance Spherocylindrical Refractions** 

**Biomicroscopy Scale** 

**Conjunctival Staining** 

**Keratometry Procedure** 

Distance and Near Visual Acuity Evaluation

Lens Insertion and Removal

White Light Lens Surface Wettability

# PRE-OCULAR AND PRE-LENS WETTABILITY

CR-5969 v3.0

# Pre-Ocular and Pre-Lens Wettability























# LIMBAL AND CONJUNCTIVAL (BULBAR) REDNESS



















CR-5969 v3.0



# **EXPANDED SODIUM FLUORESCEIN CORNEAL STAINING**













# LENS FITTING CHARACTERISTICS





| | | | | | | <br> | | |
|---|---|---|---|---|---|---|---|---|
| | | | Electronic Committee of the Committee of | | | | | |
| | | | | | | <br> | | and the second s |
| | | | | i | | | | |
| | | | - | | | <br> | | |
| | A 1 3 TO 80 TO 8 | | | | | | | |
| | | | | | <br> | <br> | | |
| | | , | | | | | | |
| | | | | | <br> | <br> | <b>-</b> | |
| _ | ······ | | | | | | | |










# SUBJECT REPORTED OCULAR SYMPTOMS/PROBLEMS



# **Subject Reported Ocular Symptoms/Problems**

# FRONT AND BACK SURFACE LENS DEPOSIT GRADING PROCEDURE














# **DETERMINATION OF DISTANCE SPHEROCYLINDRICAL REFRACTIONS**




















# BIOMICROSCOPY SCALE

















# CONJUNCTIVAL STAINING






ATTACHMENT A Visual representation of fluorescein grading.





# KERATOMETRY PROCEDURE




# DISTANCE AND NEAR VISUAL ACUITY EVALUATION












# LENS INSERTION AND REMOVAL





Page 1 of 2





## WHITE LIGHT LENS SURFACE WETTABILITY



# APPENDIX K: WORK AID: NON-INVASIVE TEAR BREAK-UP TIME (NIBUT) MEASUREMENT USING THE MEDMONT E300 CORNEAL TOPOGRAPHER

# WORK AID: NON-INVASIVE TEAR BREAK-UP TIME (NIBUT) MEASUREMENT USING THE MEDMONT E300 CORNEAL TOPOGRAPHER

#### 1.0 OBJECTIVES

Tear break-up time is a standard clinical measurement used to indicate the stability of the preocular tear film. An individual with an unstable tear film can experience symptoms of visual
disturbances or discomfort. The Medmont videokeratoscope is one type of instrument which may
be used to view the regularity of the tear film, since it displays a live video image of a set of
illuminated rings reflected by the eye surface. Disturbances to the tear film can be visualized as
disruptions to the reflected ring pattern. This measurement is a form of non-invasive tear breakup time (NIBUT), since the instrument does not touch the eye and there is no use of topical dyes.

### 2.0 MATERIALS

The Medmont E300 Corneal Topographer is a computerized videokeratometer which uses Placido rings to map the surface of the human cornea.

### **SOFTWARE VERSION**

The E300 Software is part of the Medmont Studio integrated software environment. The instructions in this Appendix apply to Medmont Studio 4 software *version 4.14.1*. Other versions of the software are unlikely to have substantial difference in basic function or data integrity.

## 3.0 DATA MANAGEMENT

The Medmont videokeratoscope consists of a light source made up of a series of concentric rings, and a video camera for recording the reflected image of these rings. For tear break-up time measurement, it is not necessary to save the series of images, but this may be done as an optional step for proof of performance or if needed for further analysis. Tear break-up time is measured with a stopwatch and the results are recorded on paper CRF forms or an eCRF data entry screen.

## 4.0 PROCEDURES

#### MEDMONT SOFTWARE SETUP

If videokeratoscope images are not being saved, it is not necessary to enter a new patient name or date of birth. Selecting video data collection mode will ensure that a continuous live video view of the participant's eye is shown on the computer monitor.


Work Aid: NIBUT Measurement using Medmont E300 Corneal Topographer



Figure 1. Selecting Normal (single frames) or Video capture control



#### PARTICIPANT SETUP

While instrument and participant alignment is being set up, the participant should be instructed to continue blinking normally.

The patient should sit comfortably in the chair. Ask the participant to put their chin onto the chinrest and put their forehead firmly against the forehead rest. Adjust the chinrest height until the eye is approximately level with the mark on the vertical bar of the headrest. The participant should push their chin forward slightly on the chinrest. Ask the participant to look into the centre of the green central illuminated ring and keep their gaze on this target during the measurement. The investigator will use the instrument joystick to move the instrument to the correct distance from the eye, and to align the instrument axis (shown as a green cross overlay) with the reflection of the central reflected ring. A red line indicates whether the instrument is too close or too far away from the participant's eye.

Figure 2: Focus examples showing Too Far, In Focus, and Too Near







If it is not possible to move the instrument in to best focus due to obstruction by the eyebrow, instruct the participant to move their chin slightly further forward on the chinrest, or their forehead slightly back from the headrest. If the instrument is obstructed by the side of the nose, ask the participant to turn their head so that their nose moves further away from the instrument.

### MEASURING TEAR BREAK-UP TIME

When the examiner is ready to commence the measurement, the participant is instructed to have a final blink (the blink should be natural, not forceful) and then to stop blinking for as long as possible and continue to look straight ahead at the central green ring. NIBUT is measured as the time interval in seconds after the final blink to the first appearance of distortion in the reflected rings; or to the time that the participant has to blink due to discomfort. The investigator must


Work Aid: NIBUT Measurement using Medmont E300 Corneal Topographer

watch for a change in the appearance of the ring pattern compared to the immediate post-blink appearance. Events that are considered distortions and thus endpoints include: debris that causes a break in the grid pattern, localized bending or blurring of a section of the ring pattern, or a distinct doubling of any lines.

The standard measurement of tear film break-up time involves three measurements on each eye. Between measurements, ask the participant to sit back from the chinrest for at least 30 seconds and to blink naturally. Taking measurements too rapidly without a sufficient rest period can result in a gradually worsening (ie. decreasing) tear film break-up time.



Figure 3: An example of the appearance of tear breakup


Work Aid: NIBUT Measurement using Medmont E300 Corneal Topographer

## **SAVING THE SERIES OF IMAGES (OPTIONAL)**

The raw images may be saved using "File/Save All Images".

In order to also save the series of topography maps, click on "File/Analyze All" before "File/Save All Images".

### 5.0 PHOTODOCUMENTATION

Not applicable

### 6.0 ADDITIONAL INFORMATION

Not applicable

## 7.0 TRAINING REQUIREMENTS

Read only

## 8.0 CASE REPORT FORM MODULE

The standard Bioclinica eCRF screen will record three measurements of NIBUT (in seconds) for each eye.

## **DOCUMENT CHANGE HISTORY**

| Originator | Change Description | Effective Date |
|-------------|--------------------|------------------|
| R. Franklin | New specification. | October 21, 2014 |


## PROTOCOL COMPLIANCE INVESTIGATOR(S) SIGNATURE PAGE

Protocol Number and Title: <u>CR-5969</u>: Clinical Characterization of Symptomatic Populations

Version and Date: v3.0 03-Oct-2017

I have read and understand the protocol specified above and agree on its content.

I agree to conduct this study according to GCP and ICH guidelines, the Declaration of Helsinki, ISO 14155<sup>2</sup>, United States (US) Code of Federal Regulations (CFR), and the pertinent individual country laws/regulations and to comply with its obligations, subject to ethical and safety considerations. The Principal Investigator is responsible for ensuring that all clinical site personnel, including Sub-Investigators adhere to all ICH regulations and GCP guidelines regarding clinical trials during and after study completion.

I will assure that no deviation from, or changes to the protocol will take place without prior agreement from the Sponsor and documented approval from the Institutional Review Board (IRB), except where necessary to eliminate an immediate hazard(s) to the trial participants.

I am responsible for ensuring that all clinical site personnel including Sub-Investigators adhere to all ICH regulations and GCP guidelines regarding clinical trials during and after study completion.

All clinical site personnel involved in the conduct of this study have completed Human Subjects Protection Training.

I agree to ensure that all clinical site personnel involved in the conduct of this study are informed about their obligations in meeting the above commitments.

I shall not disclose the information contained in this protocol or any results obtained from this study without written authorization.

| Principal Investigator: | | |
|---|---|---|
| - | Signature | Date |
| | Name and Professional Position (Printed) | - |
| Institution/Site: | | |
| | Institution/Site Name | |
| | Institution/Site Address | Processing the second s |